CLINICAL TRIAL: NCT02365649
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study of Upadacitinib (ABT-494) for the Induction of Symptomatic and Endoscopic Remission in Subjects With Moderately to Severely Active Crohn's Disease Who Have Inadequately Responded to or Are Intolerant to Immunomodulators or Anti-TNF Therapy
Brief Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study of ABT-494 for the Induction of Symptomatic and Endoscopic Remission in Subjects With Moderately to Severely Active Crohn's Disease Who Have Inadequately Responded to or Are Intolerant to Immunomodulators or Anti-TNF Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M13-740; 2014-003240-12 (EudraCT Number)
Record Dates: First submitted 2015-02-16; First posted 2015-02-19 (Estimated); Results first posted 2023-08-14 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Crohn's Disease
Keywords: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — upadacitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (9):
- Induction Period ABT-494 Twice Daily Medium/High Dose (Active Comparator): Induction Period ABT-494 Twice Daily Medium/High Dose orally dosed twice a day
  Interventions: Drug: ABT-494
- Extension Phase ABT-494 High Dose (Active Comparator): Extension Phase ABT-494 High Dose orally dosed twice a day
  Interventions: Drug: ABT-494
- Induction Period Placebo (Placebo Comparator): Induction Period Placebo orally dosed twice a day
  Interventions: Drug: Placebo
- Induction Period ABT-494 Low Dose (Active Comparator): Induction Period ABT-494 Low Dose orally dosed twice a day
  Interventions: Drug: ABT-494
- Induction Period ABT-494 Once Daily Medium/High Dose (Active Comparator): Induction Period ABT-494 Once Daily Medium/High Dose orally dosed once a day
  Interventions: Drug: ABT-494
- Extension Phase ABT-494 Low Dose (Active Comparator): Extension Phase ABT-494 Low Dose orally dosed twice a day
  Interventions: Drug: ABT-494
- Induction Period ABT-494 High Dose (Active Comparator): Induction Period ABT-494 High Dose orally dosed twice a day
  Interventions: Drug: ABT-494
- Induction Period ABT-494 Low/Medium Dose (Active Comparator): Induction Period ABT-494 Low/Medium Dose orally dosed twice a day
  Interventions: Drug: ABT-494
- Extension Phase ABT-494 Medium Dose (Active Comparator): Extension Phase ABT-494 Medium Dose orally dosed twice a day
  Interventions: Drug: ABT-494

INTERVENTIONS:
Drug: Placebo — Oral Dosing
  Arms: Induction Period Placebo
Drug: ABT-494 — Oral Dosing
  Other Names: Upadacitinib
  Arms: Extension Phase ABT-494 High Dose; Extension Phase ABT-494 Low Dose; Extension Phase ABT-494 Medium Dose; Induction Period ABT-494 High Dose; Induction Period ABT-494 Low Dose; Induction Period ABT-494 Low/Medium Dose; Induction Period ABT-494 Once Daily Medium/High Dose; Induction Period ABT-494 Twice Daily Medium/High Dose

SUMMARY:
To determine the efficacy and safety of multiple doses of ABT-494 in subjects with moderately to severely active Crohn's Disease with a history of inadequate response to or intolerance to Immunomodulators or anti-Tumor Necrosis Factor (TNF) therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Crohn's disease (CD) for at least 90 days.
2. Crohn's Disease Activity Index (CDAI) greater than or equal to 220 and less than or equal to 450.
3. Subject inadequately responded to or experienced intolerance to previous treatment with immunomodulators (e.g. azathioprine, 6-mercaptopurine, or methotrexate) and/or anti-TNF agent (e.g., infliximab, adalimumab, or certolizumab pegol).

Exclusion Criteria:

1. Subjects with ulcerative colitis (UC), collagenous colitis or indeterminate colitis.
2. Subject who has had surgical bowel resections in the past 6 months or is planning resection.
3. Subjects with an ostomy or ileoanal pouch.
4. Subject with symptomatic bowel stricture or abdominal or peri-anal abcess.
5. Subject who has short bowel syndrome.
6. Subject with recurring infections or active Tuberculosis (TB).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2015-03-17 (Actual); Primary Completion 2016-11-25 (Actual); Study Completion 2017-08-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sandborn WJ, Lewis JD, Panes J, Loftus EV, D'Haens G, Yu Z, Huang B, Lacerda AP, Pangan AL, Feagan BG. Association Between Proposed Definitions of Clinical Remission/Response and Well-Being in Patients With Crohn's Disease. J Crohns Colitis. 2022 Mar 14;16(3):444-451. doi: 10.1093/ecco-jcc/jjab161. PMID 34546360
- [Derived] Aguilar D, Revilla L, Garrido-Trigo A, Panes J, Lozano JJ, Planell N, Esteller M, Lacerda AP, Guay H, Butler J, Davis JW, Salas A. Randomized Controlled Trial Substudy of Cell-specific Mechanisms of Janus Kinase 1 Inhibition With Upadacitinib in the Crohn's Disease Intestinal Mucosa: Analysis From the CELEST Study. Inflamm Bowel Dis. 2021 Nov 15;27(12):1999-2009. doi: 10.1093/ibd/izab116. PMID 34042156
- [Derived] Peyrin-Biroulet L, Louis E, Loftus EV Jr, Lacerda A, Zhou Q, Sanchez Gonzalez Y, Ghosh S. Quality of Life and Work Productivity Improvements with Upadacitinib: Phase 2b Evidence from Patients with Moderate to Severe Crohn's Disease. Adv Ther. 2021 May;38(5):2339-2352. doi: 10.1007/s12325-021-01660-7. Epub 2021 Mar 23. PMID 33755884
- [Derived] Sandborn WJ, Feagan BG, Loftus EV Jr, Peyrin-Biroulet L, Van Assche G, D'Haens G, Schreiber S, Colombel JF, Lewis JD, Ghosh S, Armuzzi A, Scherl E, Herfarth H, Vitale L, Mohamed MF, Othman AA, Zhou Q, Huang B, Thakkar RB, Pangan AL, Lacerda AP, Panes J. Efficacy and Safety of Upadacitinib in a Randomized Trial of Patients With Crohn's Disease. Gastroenterology. 2020 Jun;158(8):2123-2138.e8. doi: 10.1053/j.gastro.2020.01.047. Epub 2020 Feb 8. PMID 32044319

RESULTS

PARTICIPANT FLOW:
Groups:
- Double-Blind Induction Phase: Placebo BID: Placebo BID during the 16-week double-blind Induction Phase.
- Double-Blind Induction Phase: Upadacitinib 3 mg BID: Upadacitinib 3 mg BID during the 16-week double-blind Induction Phase.
- Double-Blind Induction Phase: Upadacitinib 6 mg BID: Upadacitinib 6 mg BID during the 16-week double-blind Induction Phase.
- Double Blind Induction Phase: Upadacitinib 12 mg BID: Upadacitinib 12 mg BID during the 16-week double-blind Induction Phase.
- Double Blind Induction Phase: Upadacitinib 24 mg BID: Upadacitinib 24 mg BID during the 16-week double-blind Induction Phase.
- Double Blind Induction Phase: Upadacitinib 24 mg QD: Upadacitinib 24 mg once daily (consisting of two 12 mg immediate release [IR] doses) during the 16- week double-blind Induction Phase.
- Double Blind Extension Phase: Upadacitinib 3 mg BID: Upadacitinib 3 mg BID during the 36-week double-blind Extension Phase.
- Double Blind Extension Phase: Upadacitinib 6 mg BID: Upadacitinib 6 mg BID during the 36-week double-blind Extension Phase.
- Double Blind Extension Phase: Upadacitinib 12 mg BID: Upadacitinib 12 mg BID during the 36-week double-blind Extension Phase.
- Double Blind Extension Phase: Upadacitinib 24 mg QD: Upadacitinib 24 mg QD (consisting of two 12 mg IR doses) during the 36-week double-blind Extension Phase.
Period: Double-Blind Induction (Weeks 1-16)
Arm/Group | Double-Blind Induction Phase: Placebo BID | Double-Blind Induction Phase: Upadacitinib 3 mg BID | Double-Blind Induction Phase: Upadacitinib 6 mg BID | Double Blind Induction Phase: Upadacitinib 12 mg BID | Double Blind Induction Phase: Upadacitinib 24 mg BID | Double Blind Induction Phase: Upadacitinib 24 mg QD | Double Blind Extension Phase: Upadacitinib 3 mg BID | Double Blind Extension Phase: Upadacitinib 6 mg BID | Double Blind Extension Phase: Upadacitinib 12 mg BID | Double Blind Extension Phase: Upadacitinib 24 mg QD
Started | 37 | 39 | 37 | 36 | 36 | 35 | 0 | 0 | 0 | 0
Completed | 27 | 34 | 33 | 27 | 29 | 30 | 0 | 0 | 0 | 0
Not Completed | 10 | 5 | 4 | 9 | 7 | 5 | 0 | 0 | 0 | 0
Not completed — Requires alternative therapy | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 3 | 4 | 0 | 7 | 1 | 2 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 3 | 1 | 1 | 1 | 2 | 1 | 0 | 0 | 0 | 0
Not completed — Other | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Subject Non-Compliance | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Double-Blind Extension (Weeks 16-52)
Arm/Group | Double-Blind Induction Phase: Placebo BID | Double-Blind Induction Phase: Upadacitinib 3 mg BID | Double-Blind Induction Phase: Upadacitinib 6 mg BID | Double Blind Induction Phase: Upadacitinib 12 mg BID | Double Blind Induction Phase: Upadacitinib 24 mg BID | Double Blind Induction Phase: Upadacitinib 24 mg QD | Double Blind Extension Phase: Upadacitinib 3 mg BID | Double Blind Extension Phase: Upadacitinib 6 mg BID | Double Blind Extension Phase: Upadacitinib 12 mg BID | Double Blind Extension Phase: Upadacitinib 24 mg QD
Started | 0 | 0 | 0 | 0 | 0 | 0 | 61 | 23 | 59 | 37
Switched to OL 12 mg BID (Participants who met inadequate response criteria at or after Week 20 and switched to OL 12 mg BID.) | 0 | 0 | 0 | 0 | 0 | 0 | 21 | 5 | 17 | 17
Further Dose Escalated to OL 24 mg BID (Participants who were switched to OL 12 mg BID and then further dose escalated to OL 24 mg BID.) | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 2 | 10 | 10
Dose De-escalated to OL 12 mg BID (Participants who were dose escalated to OL 24 mg BID and then dose de-escalated to OL 12 mg BID.) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 43 | 21 | 43 | 22
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 18 | 2 | 16 | 15
Not completed — Requires Alternative Therapy | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 4 | 4
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 2 | 8 | 10
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1
Not completed — Subject Noncompliance | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Double-Blind Induction Phase: Placebo BID | Double-Blind Induction Phase: Upadacitinib 3 mg BID | Double-Blind Induction Phase: Upadacitinib 6 mg BID | Double Blind Induction Phase: Upadacitinib 12 mg BID | Double Blind Induction Phase: Upadacitinib 24 mg BID | Double Blind Induction Phase: Upadacitinib 24 mg QD | Total
Number analyzed (Participants) | 37 | 39 | 37 | 36 | 36 | 35 | 220
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.5 (12.14) | 39.7 (14.03) | 40.5 (13.41) | 40.8 (15.18) | 42.5 (10.02) | 40.2 (12.60) | 40.7 (12.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 19 | 21 | 17 | 25 | 19 | 125
  Male | 13 | 20 | 16 | 19 | 11 | 16 | 95
High-sensitivity C-reactive protein (hsCRP) [Mean (Standard Deviation); unit: mg/L] | 20.8 (34.29) | 23.6 (51.43) | 17.9 (17.92) | 26.9 (28.86) | 17.1 (26.49) | 17.1 (20.83) | 20.6 (32.11)
Fecal Calprotectin [Mean (Standard Deviation); unit: mcg/g] — Population: participants with an assessment at baseline
  mcg/g
    number analyzed (Participants) | 31 | 33 | 36 | 33 | 29 | 31 | 193
    (all) | 1734.7 (2444.07) | 1925.9 (2804.07) | 2128.5 (1978.73) | 2067.9 (2250.97) | 2074.8 (2324.15) | 1808.7 (2548.11) | 1960.8 (2371.86)
Inflammatory Bowel Disease Questionnaire (IBDQ) [Mean (Standard Deviation); unit: units on a scale] — The IBDQ is a disease-specific instrument composed of 32 Likert-scaled items. The total score ranges from 32 to 224 using the 7-point response options, with higher scores indicating better health-related quality of life. Population: participants with an assessment at baseline
  units on a scale
    number analyzed (Participants) | 37 | 38 | 36 | 35 | 36 | 34 | 216
    (all) | 118.0 (28.45) | 115.2 (27.48) | 113.7 (25.86) | 115.2 (36.05) | 113.8 (35.97) | 120.7 (36.25) | 116.1 (31.60)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieve Endoscopic Remission at Week 12/16
Description: Endoscopic remission was determined using Simplified Endoscopic Score for Crohn's Disease (SES-CD). SES-CD subscores assess the following: presence and size of ulcers in 5 visualized bowel segments; extent of ulcerated surface in 5 visualized bowel segments; extent of affected surface in 5 visualized bowel segments; presence and type of narrowings in 5 visualized bowel segments. Subscores range from 0 to 15, and are summed for a total SES-CD score ranging from 0 to 56; higher scores indicate greater severity of mucosal inflammation. Endoscopic remission: SES-CD ≤ 4 and at least 2-point reduction versus Baseline and no subscore > 1 in any individual variable.
Time Frame: Up to Week 16. (At Baseline, participants were allocated by randomization 1:1 to have their end of induction colonoscopy done at either Week 12 or Week 16; this endpoint combines the two time points.)
Population: Modified intention to Treat (mITT) Population: all randomized participants who took at least 1 dose of study drug in the Induction Period. Non-responder imputation.
Measure: Number; unit: percentage of participants
Arm/Group | Double-Blind Induction Phase: Placebo BID | Double-Blind Induction Phase: Upadacitinib 3 mg BID | Double-Blind Induction Phase: Upadacitinib 6 mg BID | Double Blind Induction Phase: Upadacitinib 12 mg BID | Double Blind Induction Phase: Upadacitinib 24 mg BID | Double Blind Induction Phase: Upadacitinib 24 mg QD
Number analyzed (Participants) | 37 | 39 | 37 | 36 | 36 | 35
percentage of participants | 0 | 10.3 | 8.1 | 8.3 | 22.2 | 14.3
Statistical Analysis 1: Comparison: Double-Blind Induction Phase: Placebo BID vs Double-Blind Induction Phase: Upadacitinib 3 mg BID; Test type: Superiority; p = 0.056, Cochran-Mantel-Haenszel — Statistical significance was prespecified at α = 0.1. Based on Cochran-Mantel-Haenszel (CMH) test stratified by baseline SES-CD (SES-CD <15 and SES-CD >=15); Adjusted risk difference from placebo = 9.9, 95% CI 2-sided [-0.3 to 20.1]
Statistical Analysis 2: Comparison: Double-Blind Induction Phase: Placebo BID vs Double-Blind Induction Phase: Upadacitinib 6 mg BID; Test type: Superiority; p = 0.108, Cochran-Mantel-Haenszel — Statistical significance was prespecified at α = 0.1. Based on CMH test stratified by baseline SES-CD (SES-CD <15 and SES-CD >=15); Adjusted risk difference from placebo = 7.4, 95% CI 2-sided [-1.6 to 16.4]
Statistical Analysis 3: Comparison: Double-Blind Induction Phase: Placebo BID vs Double Blind Induction Phase: Upadacitinib 12 mg BID; Test type: Superiority; p = 0.099, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Adjusted risk difference from placebo = 7.7, 95% CI 2-sided [-1.5 to 16.8]
Statistical Analysis 4: Comparison: Double-Blind Induction Phase: Placebo BID vs Double Blind Induction Phase: Upadacitinib 24 mg BID; Test type: Superiority; p = 0.004, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Adjusted risk difference from placebo = 21, 95% CI 2-sided [6.8 to 35.2]
Statistical Analysis 5: Comparison: Double-Blind Induction Phase: Placebo BID vs Double Blind Induction Phase: Upadacitinib 24 mg QD; Test type: Superiority; p = 0.025, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Adjusted risk difference from placebo = 13.6, 95% CI 2-sided [1.8 to 25.5]

2. Primary Outcome: Percentage of Participants Who Achieve Clinical Remission at Week 16
Description: Clinical remission: average daily stool frequency ≤ 1.5 and not worse than Baseline AND average daily abdominal pain ≤ 1.0 and not worse than Baseline. The very soft/liquid stool frequency and abdominal pain scores at a visit were the average of the daily values reported during the 7 usable days preceding the scheduled assessment visit. Abdominal Pain was rated on a 4-point scale from 0 (none) to 3 (severe).
Time Frame: Week 16
Population: mITT Population: all randomized participants who took at least 1 dose of study drug in the Induction Period. Non-responder imputation.
Measure: Number; unit: percentage of participants
Arm/Group | Double-Blind Induction Phase: Placebo BID | Double-Blind Induction Phase: Upadacitinib 3 mg BID | Double-Blind Induction Phase: Upadacitinib 6 mg BID | Double Blind Induction Phase: Upadacitinib 12 mg BID | Double Blind Induction Phase: Upadacitinib 24 mg BID | Double Blind Induction Phase: Upadacitinib 24 mg QD
Number analyzed (Participants) | 37 | 39 | 37 | 36 | 36 | 35
percentage of participants | 10.8 | 12.8 | 27.0 | 11.1 | 22.2 | 14.3
Statistical Analysis 1: Comparison: Double-Blind Induction Phase: Placebo BID vs Double-Blind Induction Phase: Upadacitinib 3 mg BID; Test type: Superiority; p = 0.74, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Adjusted risk difference from placebo = 2.5, 95% CI 2-sided [-12.3 to 17.3]
Statistical Analysis 2: Comparison: Double-Blind Induction Phase: Placebo BID vs Double-Blind Induction Phase: Upadacitinib 6 mg BID; Test type: Superiority; p = 0.082, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Adjusted risk difference from placebo = 16.2, 95% CI 2-sided [-2.0 to 34.3]
Statistical Analysis 3: Comparison: Double-Blind Induction Phase: Placebo BID vs Double Blind Induction Phase: Upadacitinib 12 mg BID; Test type: Superiority; p = 0.952, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Adjusted risk difference from placebo = 0.5, 95% CI 2-sided [-14.1 to 15.0]
Statistical Analysis 4: Comparison: Double-Blind Induction Phase: Placebo BID vs Double Blind Induction Phase: Upadacitinib 24 mg BID; Test type: Superiority; p = 0.205, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Adjusted risk difference from placebo = 11.2, 95% CI 2-sided [-6.1 to 28.5]
Statistical Analysis 5: Comparison: Double-Blind Induction Phase: Placebo BID vs Double Blind Induction Phase: Upadacitinib 24 mg QD; Test type: Superiority; p = 0.607, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Adjusted risk difference from placebo = 4.1, 95% CI 2-sided [-11.5 to 19.6]

3. Secondary Outcome: Percentage of Participants Who Achieve Crohn's Disease Activity Index (CDAI) < 150 at Week 16
Description: CDAI is used to quantify the signs and symptoms of subjects with Crohn's disease. The score includes the frequency of stools, abdominal pain and general well-being as well as the presence of complications, use of antidiarrheals, presence of abdominal mass, hematocrit and weight. CDAI generally ranges from 0 to 600 where higher scores indicate more severe disease. A score below 150 indicates remission.
Time Frame: Week 16
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Double-Blind Induction Phase: Placebo BID | Double-Blind Induction Phase: Upadacitinib 3 mg BID | Double-Blind Induction Phase: Upadacitinib 6 mg BID | Double Blind Induction Phase: Upadacitinib 12 mg BID | Double Blind Induction Phase: Upadacitinib 24 mg BID | Double Blind Induction Phase: Upadacitinib 24 mg QD
Number analyzed (Participants) | 37 | 39 | 37 | 36 | 36 | 35
percentage of participants | 16.2 | 20.5 | 29.7 | 38.9 | 30.6 | 20.0
Statistical Analysis 1: Comparison: Double-Blind Induction Phase: Placebo BID vs Double-Blind Induction Phase: Upadacitinib 3 mg BID; Test type: Superiority; p = 0.564, Cochran-Mantel-Haenszel — Based on CMH test stratified by baseline SES-CD (SES-CD <15 and SES-CD >=15); Adjusted risk difference from placebo = 5.2, 95% CI 2-sided [-12.5 to 22.9]
Statistical Analysis 2: Comparison: Double-Blind Induction Phase: Placebo BID vs Double-Blind Induction Phase: Upadacitinib 6 mg BID; Test type: Superiority; p = 0.221, Cochran-Mantel-Haenszel — Based on CMH test stratified by baseline SES-CD (SES-CD <15 and SES-CD >=15); Adjusted risk difference from placebo = 12, 95% CI 2-sided [-7.2 to 31.2]
Statistical Analysis 3: Comparison: Double-Blind Induction Phase: Placebo BID vs Double Blind Induction Phase: Upadacitinib 12 mg BID; Test type: Superiority; p = 0.036, Cochran-Mantel-Haenszel — Based on CMH test stratified by baseline SES-CD (SES-CD <15 and SES-CD >=15); Adjusted risk difference from placebo = 22.2, 95% CI 2-sided [1.4 to 43]
Statistical Analysis 4: Comparison: Double-Blind Induction Phase: Placebo BID vs Double Blind Induction Phase: Upadacitinib 24 mg BID; Test type: Superiority; p = 0.179, Cochran-Mantel-Haenszel — Based on CMH test stratified by baseline SES-CD (SES-CD <15 and SES-CD >=15); Adjusted risk difference from placebo = 13.4, 95% CI 2-sided [-6.2 to 33.1]
Statistical Analysis 5: Comparison: Double-Blind Induction Phase: Placebo BID vs Double Blind Induction Phase: Upadacitinib 24 mg QD; Test type: Superiority; p = 0.677, Cochran-Mantel-Haenszel — Based on CMH test stratified by baseline SES-CD (SES-CD <15 and SES-CD >=15); Adjusted risk difference from placebo = 3.9, 95% CI 2-sided [-14.3 to 22]

4. Secondary Outcome: Percentage of Participants With a Decrease in CDAI ≥ 70 Points From Baseline at Week 16
Description: CDAI is used to quantify the signs and symptoms of subjects with Crohn's disease. The score includes the frequency of stools, abdominal pain and general well-being as well as the presence of complications, use of antidiarrheals, presence of abdominal mass, hematocrit and weight. CDAI generally ranges from 0 to 600 where higher scores indicate more severe disease. A 70-point decrease in the CDAI index refers to improvement in the disease activity from Baseline.
Time Frame: Week 16
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Double-Blind Induction Phase: Placebo BID | Double-Blind Induction Phase: Upadacitinib 3 mg BID | Double-Blind Induction Phase: Upadacitinib 6 mg BID | Double Blind Induction Phase: Upadacitinib 12 mg BID | Double Blind Induction Phase: Upadacitinib 24 mg BID | Double Blind Induction Phase: Upadacitinib 24 mg QD
Number analyzed (Participants) | 37 | 39 | 37 | 36 | 36 | 35
percentage of participants | 35.1 | 46.2 | 54.1 | 44.4 | 61.1 | 48.6
Statistical Analysis 1: Comparison: Double-Blind Induction Phase: Placebo BID vs Double-Blind Induction Phase: Upadacitinib 3 mg BID; Test type: Superiority; p = 0.363, Cochran-Mantel-Haenszel — Based on CMH test stratified by baseline SES-CD (SES-CD <15 and SES-CD >=15); Adjusted risk difference from placebo = 10.4, 95% CI 2-sided [-12 to 32.9]
Statistical Analysis 2: Comparison: Double-Blind Induction Phase: Placebo BID vs Double-Blind Induction Phase: Upadacitinib 6 mg BID; Test type: Superiority; p = 0.137, Cochran-Mantel-Haenszel — Based on CMH test stratified by baseline SES-CD (SES-CD <15 and SES-CD >=15); Adjusted risk difference from placebo = 17.3, 95% CI 2-sided [-5.5 to 40]
Statistical Analysis 3: Comparison: Double-Blind Induction Phase: Placebo BID vs Double Blind Induction Phase: Upadacitinib 12 mg BID; Test type: Superiority; p = 0.512, Cochran-Mantel-Haenszel — Based on CMH test stratified by baseline SES-CD (SES-CD <15 and SES-CD >=15); Adjusted risk difference from placebo = 7.5, 95% CI 2-sided [-14.9 to 29.9]
Statistical Analysis 4: Comparison: Double-Blind Induction Phase: Placebo BID vs Double Blind Induction Phase: Upadacitinib 24 mg BID; Test type: Superiority; p = 0.035, Cochran-Mantel-Haenszel — Based on CMH test stratified by baseline SES-CD (SES-CD <15 and SES-CD >=15); Adjusted risk difference from placebo = 25, 95% CI 2-sided [-1.8 to 48.2]
Statistical Analysis 5: Comparison: Double-Blind Induction Phase: Placebo BID vs Double Blind Induction Phase: Upadacitinib 24 mg QD; Test type: Superiority; p = 0.29, Cochran-Mantel-Haenszel — Based on CMH test stratified by baseline SES-CD (SES-CD <15 and SES-CD >=15); Adjusted risk difference from placebo = 12.5, 95% CI 2-sided [-10.7 to 35.6]

5. Secondary Outcome: Percentage of Participants Who Achieve Clinical Remission at Week 12
Description: as for outcome 2
Time Frame: Week 12
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Double-Blind Induction Phase: Placebo BID | Double-Blind Induction Phase: Upadacitinib 3 mg BID | Double-Blind Induction Phase: Upadacitinib 6 mg BID | Double Blind Induction Phase: Upadacitinib 12 mg BID | Double Blind Induction Phase: Upadacitinib 24 mg BID | Double Blind Induction Phase: Upadacitinib 24 mg QD
Number analyzed (Participants) | 37 | 39 | 37 | 36 | 36 | 35
percentage of participants | 10.8 | 10.3 | 29.7 | 13.9 | 25.0 | 8.6
Statistical Analysis 1: Comparison: Double-Blind Induction Phase: Placebo BID vs Double-Blind Induction Phase: Upadacitinib 3 mg BID; Test type: Superiority; p = 0.896, Cochran-Mantel-Haenszel — Based on CMH test stratified by baseline SES-CD (SES-CD <15 and SES-CD >=15); Adjusted risk difference from placebo = -0.9, 95% CI 2-sided [-15.0 to 13.1]
Statistical Analysis 2: Comparison: Double-Blind Induction Phase: Placebo BID vs Double-Blind Induction Phase: Upadacitinib 6 mg BID; Test type: Superiority; p = 0.05, Cochran-Mantel-Haenszel — Based on CMH test stratified by baseline SES-CD (SES-CD <15 and SES-CD >=15); Adjusted risk difference from placebo = 18.6, 95% CI 2-sided [0.0 to 37.3]
Statistical Analysis 3: Comparison: Double-Blind Induction Phase: Placebo BID vs Double Blind Induction Phase: Upadacitinib 12 mg BID; Test type: Superiority; p = 0.702, Cochran-Mantel-Haenszel — Based on CMH test stratified by baseline SES-CD (SES-CD <15 and SES-CD >=15); Adjusted risk difference from placebo = 3.0, 95% CI 2-sided [-12.4 to 18.4]
Statistical Analysis 4: Comparison: Double-Blind Induction Phase: Placebo BID vs Double Blind Induction Phase: Upadacitinib 24 mg BID; Test type: Superiority; p = 0.117, Cochran-Mantel-Haenszel — Based on CMH test stratified by baseline SES-CD (SES-CD <15 and SES-CD >=15); Adjusted risk difference from placebo = 14.3, 95% CI 2-sided [-3.6 to 32.2]
Statistical Analysis 5: Comparison: Double-Blind Induction Phase: Placebo BID vs Double Blind Induction Phase: Upadacitinib 24 mg QD; Test type: Superiority; p = 0.736, Cochran-Mantel-Haenszel — Based on CMH test stratified by baseline SES-CD (SES-CD <15 and SES-CD >=15); Adjusted risk difference from placebo = -2.4, 95% CI 2-sided [-16.4 to 11.6]

6. Secondary Outcome: Percentage of Participants Who Achieve Remission at Week 16
Description: Remission is defined as endoscopic remission at Week 12/16 AND clinical remission at Week 16. Endoscopic remission: SES-CD ≤ 4 and at least 2-point reduction versus Baseline and no subscore > 1 in any individual variable. Clinical remission: average daily stool frequency ≤ 1.5 and not worse than Baseline AND average daily abdominal pain ≤ 1.0 and not worse than Baseline. The very soft/liquid stool frequency and abdominal pain scores at a visit were the average of the daily values reported during the 7 usable days preceding the scheduled assessment visit. Abdominal Pain was rated on a 4-point scale from 0 (none) to 3 (severe). Details of the SES-CD scale are provided in the description of the first primary endpoint.
Time Frame: Week 16
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Double-Blind Induction Phase: Placebo BID | Double-Blind Induction Phase: Upadacitinib 3 mg BID | Double-Blind Induction Phase: Upadacitinib 6 mg BID | Double Blind Induction Phase: Upadacitinib 12 mg BID | Double Blind Induction Phase: Upadacitinib 24 mg BID | Double Blind Induction Phase: Upadacitinib 24 mg QD
Number analyzed (Participants) | 37 | 39 | 37 | 36 | 36 | 35
percentage of participants | 0.0 | 2.6 | 5.4 | 2.8 | 8.3 | 5.7
Statistical Analysis 1: Comparison: Double-Blind Induction Phase: Placebo BID vs Double-Blind Induction Phase: Upadacitinib 3 mg BID; Test type: Superiority; p = 0.276, Cochran-Mantel-Haenszel — Based on CMH test stratified by baseline SES-CD (SES-CD <15 and SES-CD >=15); Adjusted risk difference from placebo = 2.9, 95% CI 2-sided [-2.3 to 8.1]
Statistical Analysis 2: Comparison: Double-Blind Induction Phase: Placebo BID vs Double-Blind Induction Phase: Upadacitinib 6 mg BID; Test type: Superiority; p = 0.195, Cochran-Mantel-Haenszel — Based on CMH test stratified by baseline SES-CD (SES-CD <15 and SES-CD >=15); Adjusted risk difference from placebo = 4.9, 95% CI 2-sided [-2.5 to 12.4]
Statistical Analysis 3: Comparison: Double-Blind Induction Phase: Placebo BID vs Double Blind Induction Phase: Upadacitinib 12 mg BID; Test type: Superiority; p = 0.355, Cochran-Mantel-Haenszel — Based on CMH test stratified by baseline SES-CD (SES-CD <15 and SES-CD >=15); Adjusted risk difference from placebo = 2.6, 95% CI 2-sided [-2.9 to 8.0]
Statistical Analysis 4: Comparison: Double-Blind Induction Phase: Placebo BID vs Double Blind Induction Phase: Upadacitinib 24 mg BID; Test type: Superiority; p = 0.099, Cochran-Mantel-Haenszel — Based on CMH test stratified by baseline SES-CD (SES-CD <15 and SES-CD >=15); Adjusted risk difference from placebo = 7.7, 95% CI 2-sided [-1.5 to 16.8]
Statistical Analysis 5: Comparison: Double-Blind Induction Phase: Placebo BID vs Double Blind Induction Phase: Upadacitinib 24 mg QD; Test type: Superiority; p = 0.185, Cochran-Mantel-Haenszel — Based on CMH test stratified by baseline SES-CD (SES-CD <15 and SES-CD >=15); Adjusted risk difference from placebo = 5.2, 95% CI 2-sided [-2.5 to 12.9]

7. Secondary Outcome: Percentage of Participants Who Achieve Response at Week 16
Description: Response is defined as endoscopic response at Week 12/16 AND clinical response at Week 16. Endoscopic response: SES-CD at least 25% reduction from Baseline. Clinical response: average daily stool frequency at least 30% reduction from Baseline and average daily abdominal pain not worse than Baseline OR average daily abdominal pain at least 30% reduction from Baseline and average daily stool frequency not worse than Baseline. The very soft/liquid stool frequency and abdominal pain scores at a visit were the average of the daily values reported during the 7 usable days preceding the scheduled assessment visit. Abdominal Pain was rated on a 4-point scale from 0 (none) to 3 (severe). Details of the SES-CD scale are provided in the description of the first primary endpoint.
Time Frame: Week 16
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Double-Blind Induction Phase: Placebo BID | Double-Blind Induction Phase: Upadacitinib 3 mg BID | Double-Blind Induction Phase: Upadacitinib 6 mg BID | Double Blind Induction Phase: Upadacitinib 12 mg BID | Double Blind Induction Phase: Upadacitinib 24 mg BID | Double Blind Induction Phase: Upadacitinib 24 mg QD
Number analyzed (Participants) | 37 | 39 | 37 | 36 | 36 | 35
percentage of participants | 2.7 | 15.4 | 32.4 | 27.8 | 38.9 | 34.3
Statistical Analysis 1: Comparison: Double-Blind Induction Phase: Placebo BID vs Double-Blind Induction Phase: Upadacitinib 3 mg BID; Test type: Superiority; p = 0.05, Cochran-Mantel-Haenszel — Based on CMH test stratified by baseline SES-CD (SES-CD <15 and SES-CD >=15); Adjusted risk difference from placebo = 13.2, 95% CI 2-sided [0.0 to 26.5]
Statistical Analysis 2: Comparison: Double-Blind Induction Phase: Placebo BID vs Double-Blind Induction Phase: Upadacitinib 6 mg BID; Test type: Superiority; p = 0.001, Cochran-Mantel-Haenszel — Based on CMH test stratified by baseline SES-CD (SES-CD <15 and SES-CD >=15); Adjusted risk difference from placebo = 29.5, 95% CI 2-sided [11.9 to 47.1]
Statistical Analysis 3: Comparison: Double-Blind Induction Phase: Placebo BID vs Double Blind Induction Phase: Upadacitinib 12 mg BID; Test type: Superiority; p = 0.003, Cochran-Mantel-Haenszel — Based on CMH test stratified by baseline SES-CD (SES-CD <15 and SES-CD >=15); Adjusted risk difference from placebo = 25.2, 95% CI 2-sided [8.5 to 42.0]
Statistical Analysis 4: Comparison: Double-Blind Induction Phase: Placebo BID vs Double Blind Induction Phase: Upadacitinib 24 mg BID; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — Based on CMH test stratified by baseline SES-CD (SES-CD <15 and SES-CD >=15); Adjusted risk difference from placebo = 36.5, 95% CI 2-sided [17.6 to 55.4]
Statistical Analysis 5: Comparison: Double-Blind Induction Phase: Placebo BID vs Double Blind Induction Phase: Upadacitinib 24 mg QD; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — Based on CMH test stratified by baseline SES-CD (SES-CD <15 and SES-CD >=15); Adjusted risk difference from placebo = 32.0, 95% CI 2-sided [13.9 to 50.2]

8. Secondary Outcome: Percentage of Participants With Endoscopic Response at Week 12/16
Description: Endoscopic response: SES-CD at least 25% reduction from Baseline. Details of the SES-CD scale are provided in the description of the first primary endpoint.
Time Frame: Up to Week 16 (At Baseline, participants were allocated by randomization 1:1 to have their end of induction colonoscopy done at either Week 12 or Week 16; this endpoint combines the two time points.)
Population: mITT Population: all randomized subjects who took at least 1 dose of study drug in the Induction Period. Non-responder imputation.
Measure: Number; unit: percentage of participants
Arm/Group | Double-Blind Induction Phase: Placebo BID | Double-Blind Induction Phase: Upadacitinib 3 mg BID | Double-Blind Induction Phase: Upadacitinib 6 mg BID | Double Blind Induction Phase: Upadacitinib 12 mg BID | Double Blind Induction Phase: Upadacitinib 24 mg BID | Double Blind Induction Phase: Upadacitinib 24 mg QD
Number analyzed (Participants) | 37 | 39 | 37 | 36 | 36 | 35
percentage of participants | 13.5 | 23.1 | 43.2 | 36.1 | 50.0 | 48.6
Statistical Analysis 1: Comparison: Double-Blind Induction Phase: Placebo BID vs Double-Blind Induction Phase: Upadacitinib 3 mg BID; Test type: Superiority; p = 0.243, Cochran-Mantel-Haenszel — Based on CMH test stratified by baseline SES-CD (SES-CD <15 and SES-CD >=15); Adjusted risk difference from placebo = 10.5, 95% CI 2-sided [-7.2 to 28.2]
Statistical Analysis 2: Comparison: Double-Blind Induction Phase: Placebo BID vs Double-Blind Induction Phase: Upadacitinib 6 mg BID; Test type: Superiority; p = 0.006, Cochran-Mantel-Haenszel — Based on CMH test stratified by baseline SES-CD (SES-CD <15 and SES-CD >=15); Adjusted risk difference from placebo = 29.1, 95% CI 2-sided [8.3 to 49.9]
Statistical Analysis 3: Comparison: Double-Blind Induction Phase: Placebo BID vs Double Blind Induction Phase: Upadacitinib 12 mg BID; Test type: Superiority; p = 0.017, Cochran-Mantel-Haenszel — Based on CMH test stratified by baseline SES-CD (SES-CD <15 and SES-CD >=15); Adjusted risk difference from placebo = 24.2, 95% CI 2-sided [4.4 to 44.1]
Statistical Analysis 4: Comparison: Double-Blind Induction Phase: Placebo BID vs Double Blind Induction Phase: Upadacitinib 24 mg BID; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — Based on CMH test stratified by baseline SES-CD (SES-CD <15 and SES-CD >=15); Adjusted risk difference from placebo = 36.5, 95% CI 2-sided [14.8 to 58.1]
Statistical Analysis 5: Comparison: Double-Blind Induction Phase: Placebo BID vs Double Blind Induction Phase: Upadacitinib 24 mg QD; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — Based on CMH test stratified by baseline SES-CD (SES-CD <15 and SES-CD >=15); Adjusted risk difference from placebo = 36.8, 95% CI 2-sided [15.2 to 58.3]

9. Secondary Outcome: Percentage of Participants Who Achieve Clinical Response at Week 16
Description: Clinical response: average daily stool frequency at least 30% reduction from Baseline and average daily abdominal pain not worse than Baseline OR average daily abdominal pain at least 30% reduction from Baseline and average daily stool frequency not worse than Baseline. The very soft/liquid stool frequency and abdominal pain scores at a visit were the average of the daily values reported during the 7 usable days preceding the scheduled assessment visit. Abdominal Pain was rated on a 4-point scale from 0 (none) to 3 (severe).
Time Frame: Week 16
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Double-Blind Induction Phase: Placebo BID | Double-Blind Induction Phase: Upadacitinib 3 mg BID | Double-Blind Induction Phase: Upadacitinib 6 mg BID | Double Blind Induction Phase: Upadacitinib 12 mg BID | Double Blind Induction Phase: Upadacitinib 24 mg BID | Double Blind Induction Phase: Upadacitinib 24 mg QD
Number analyzed (Participants) | 37 | 39 | 37 | 36 | 36 | 35
percentage of participants | 32.4 | 43.6 | 56.8 | 47.2 | 61.1 | 48.6
Statistical Analysis 1: Comparison: Double-Blind Induction Phase: Placebo BID vs Double-Blind Induction Phase: Upadacitinib 3 mg BID; Test type: Superiority; p = 0.353, Cochran-Mantel-Haenszel — Based on CMH test stratified by baseline SES-CD (SES-CD <15 and SES-CD >=15); Adjusted risk difference from placebo = 10.5, 95% CI 2-sided [-11.7 to 32.7]
Statistical Analysis 2: Comparison: Double-Blind Induction Phase: Placebo BID vs Double-Blind Induction Phase: Upadacitinib 6 mg BID; Test type: Superiority; p = 0.05, Cochran-Mantel-Haenszel — Based on CMH test stratified by baseline SES-CD (SES-CD <15 and SES-CD >=15); Adjusted risk difference from placebo = 22.7, 95% CI 2-sided [0.0 to 45.5]
Statistical Analysis 3: Comparison: Double-Blind Induction Phase: Placebo BID vs Double Blind Induction Phase: Upadacitinib 12 mg BID; Test type: Superiority; p = 0.268, Cochran-Mantel-Haenszel — Based on CMH test stratified by baseline SES-CD (SES-CD <15 and SES-CD >=15); Adjusted risk difference from placebo = 12.5, 95% CI 2-sided [-9.6 to 34.6]
Statistical Analysis 4: Comparison: Double-Blind Induction Phase: Placebo BID vs Double Blind Induction Phase: Upadacitinib 24 mg BID; Test type: Superiority; p = 0.018, Cochran-Mantel-Haenszel — Based on CMH test stratified by baseline SES-CD (SES-CD <15 and SES-CD >=15); Adjusted risk difference from placebo = 28.0, 95% CI 2-sided [4.8 to 51.2]
Statistical Analysis 5: Comparison: Double-Blind Induction Phase: Placebo BID vs Double Blind Induction Phase: Upadacitinib 24 mg QD; Test type: Superiority; p = 0.204, Cochran-Mantel-Haenszel — Based on CMH test stratified by baseline SES-CD (SES-CD <15 and SES-CD >=15); Adjusted risk difference from placebo = 14.9, 95% CI 2-sided [-8.1 to 37.8]

10. Secondary Outcome: Percentage of Participants With an Average Daily Stool Frequency ≥ 2.5 AND Average Daily Abdominal Pain ≥ 2.0 at Baseline Who Achieve Clinical Remission at Week 16
Description: as for outcome 2
Time Frame: Week 16
Population: mITT Population: all randomized participants who took at least 1 dose of study drug in the Induction Period. Includes only mITT participants with an average daily stool frequency ≥ 2.5 AND average daily abdominal pain ≥ 2.0 at Baseline. Non-responder imputation.
Measure: Number; unit: percentage of participants
Arm/Group | Double-Blind Induction Phase: Placebo BID | Double-Blind Induction Phase: Upadacitinib 3 mg BID | Double-Blind Induction Phase: Upadacitinib 6 mg BID | Double Blind Induction Phase: Upadacitinib 12 mg BID | Double Blind Induction Phase: Upadacitinib 24 mg BID | Double Blind Induction Phase: Upadacitinib 24 mg QD
Number analyzed (Participants) | 14 | 17 | 16 | 18 | 12 | 18
percentage of participants | 7.1 | 17.6 | 18.8 | 16.7 | 25.0 | 11.1
Statistical Analysis 1: Comparison: Double-Blind Induction Phase: Placebo BID vs Double-Blind Induction Phase: Upadacitinib 3 mg BID; Test type: Superiority; p = 0.421, Cochran-Mantel-Haenszel — Based on CMH test stratified by baseline SES-CD (SES-CD <15 and SES-CD >=15); Adjusted risk difference from placebo = 10.0, 95% CI 2-sided [-14.4 to 34.4]
Statistical Analysis 2: Comparison: Double-Blind Induction Phase: Placebo BID vs Double-Blind Induction Phase: Upadacitinib 6 mg BID; Test type: Superiority; p = 0.371, Cochran-Mantel-Haenszel — Based on CMH test stratified by baseline SES-CD (SES-CD <15 and SES-CD >=15); Adjusted risk difference from placebo = 11.5, 95% CI 2-sided [-13.8 to 36.8]
Statistical Analysis 3: Comparison: Double-Blind Induction Phase: Placebo BID vs Double Blind Induction Phase: Upadacitinib 12 mg BID; Test type: Superiority; p = 0.445, Cochran-Mantel-Haenszel — Based on CMH test stratified by baseline SES-CD (SES-CD <15 and SES-CD >=15); Adjusted risk difference from placebo = 9.2, 95% CI 2-sided [-14.4 to 32.8]
Statistical Analysis 4: Comparison: Double-Blind Induction Phase: Placebo BID vs Double Blind Induction Phase: Upadacitinib 24 mg BID; Test type: Superiority; p = 0.198, Cochran-Mantel-Haenszel — Based on CMH test stratified by baseline SES-CD (SES-CD <15 and SES-CD >=15); Adjusted risk difference from placebo = 19.5, 95% CI 2-sided [-10.2 to 49.3]
Statistical Analysis 5: Comparison: Double-Blind Induction Phase: Placebo BID vs Double Blind Induction Phase: Upadacitinib 24 mg QD; Test type: Superiority; p = 0.654, Cochran-Mantel-Haenszel — Based on CMH test stratified by baseline SES-CD (SES-CD <15 and SES-CD >=15); Adjusted risk difference from placebo = 5.0, 95% CI 2-sided [-17.0 to 27.0]

11. Secondary Outcome: Percentage of Participants Taking Corticosteroids at Baseline Who Discontinued Corticosteroid Use and Achieve CDAI < 150 at Week 16
Description: as for outcome 3
Time Frame: Week 16
Population: mITT Population: all randomized participants who took at least 1 dose of study drug in the Induction Period. Includes only participants taking corticosteroids at Baseline. Non-responder imputation.
Measure: Number; unit: percentage of participants
Arm/Group | Double-Blind Induction Phase: Placebo BID | Double-Blind Induction Phase: Upadacitinib 3 mg BID | Double-Blind Induction Phase: Upadacitinib 6 mg BID | Double Blind Induction Phase: Upadacitinib 12 mg BID | Double Blind Induction Phase: Upadacitinib 24 mg BID | Double Blind Induction Phase: Upadacitinib 24 mg QD
Number analyzed (Participants) | 15 | 21 | 18 | 17 | 15 | 10
percentage of participants | 0.0 | 19.0 | 22.2 | 41.2 | 33.3 | 10.0
Statistical Analysis 1: Comparison: Double-Blind Induction Phase: Placebo BID vs Double-Blind Induction Phase: Upadacitinib 3 mg BID; Test type: Superiority; p = 0.093, Cochran-Mantel-Haenszel — Based on CMH test stratified by baseline SES-CD (SES-CD <15 and SES-CD >=15); Adjusted risk difference from placebo = 18.7, 95% CI 2-sided [-3.1 to 40.5]
Statistical Analysis 2: Comparison: Double-Blind Induction Phase: Placebo BID vs Double-Blind Induction Phase: Upadacitinib 6 mg BID; Test type: Superiority; p = 0.176, Cochran-Mantel-Haenszel — Based on CMH test stratified by baseline SES-CD (SES-CD <15 and SES-CD >=15); Adjusted risk difference from placebo = 13.5, 95% CI 2-sided [-6.1 to 33.1]
Statistical Analysis 3: Comparison: Double-Blind Induction Phase: Placebo BID vs Double Blind Induction Phase: Upadacitinib 12 mg BID; Test type: Superiority; p = 0.017, Cochran-Mantel-Haenszel — Based on CMH test stratified by baseline SES-CD (SES-CD <15 and SES-CD >=15); Adjusted risk difference from placebo = 35.9, 95% CI 2-sided [6.3 to 65.5]
Statistical Analysis 4: Comparison: Double-Blind Induction Phase: Placebo BID vs Double Blind Induction Phase: Upadacitinib 24 mg BID; Test type: Superiority; p = 0.044, Cochran-Mantel-Haenszel; Adjusted risk difference from placebo = 26.1, 95% CI 2-sided [0.7 to 51.5]
Statistical Analysis 5: Comparison: Double-Blind Induction Phase: Placebo BID vs Double Blind Induction Phase: Upadacitinib 24 mg QD; Test type: Superiority; p = 0.121, Cochran-Mantel-Haenszel — Based on CMH test stratified by baseline SES-CD (SES-CD <15 and SES-CD >=15); Adjusted risk difference from placebo = 13.1, 95% CI 2-sided [-3.5 to 29.6]

12. Secondary Outcome: Percentage of Participants Taking Corticosteroids at Baseline Who Discontinued Corticosteroid Use and Achieve Remission at Week 12/16 and Clinical Remission at Week 16
Description: as for outcome 6
Time Frame: Up to Week 16. (At Baseline, subjects were allocated by randomization 1:1 to have their end of induction colonoscopy done at either Week 12 or Week 16; this endpoint combines the two time points.)
Population: as for outcome 11
Measure: Number; unit: percentage of participants
Arm/Group | Double-Blind Induction Phase: Placebo BID | Double-Blind Induction Phase: Upadacitinib 3 mg BID | Double-Blind Induction Phase: Upadacitinib 6 mg BID | Double Blind Induction Phase: Upadacitinib 12 mg BID | Double Blind Induction Phase: Upadacitinib 24 mg BID | Double Blind Induction Phase: Upadacitinib 24 mg QD
Number analyzed (Participants) | 15 | 21 | 18 | 17 | 15 | 10
percentage of participants | 0.0 | 0.0 | 5.6 | 5.9 | 13.3 | 0.0
Statistical Analysis 1: Comparison: Double-Blind Induction Phase: Placebo BID vs Double-Blind Induction Phase: Upadacitinib 6 mg BID; Test type: Superiority; p = 0.564, Cochran-Mantel-Haenszel — Based on CMH test stratified by baseline SES-CD (SES-CD <15 and SES-CD >=15); Adjusted risk difference from placebo = 3.4, 95% CI 2-sided [-8.1 to 14.9]
Statistical Analysis 2: Comparison: Double-Blind Induction Phase: Placebo BID vs Double Blind Induction Phase: Upadacitinib 12 mg BID; Test type: Superiority; p = 0.584, Cochran-Mantel-Haenszel — Based on CMH test stratified by baseline SES-CD (SES-CD <15 and SES-CD >=15); Adjusted risk difference from placebo = 3.4, 95% CI 2-sided [-8.8 to 15.7]
Statistical Analysis 3: Comparison: Double-Blind Induction Phase: Placebo BID vs Double Blind Induction Phase: Upadacitinib 24 mg BID; Test type: Superiority; p = 0.326, Cochran-Mantel-Haenszel — Based on CMH test stratified by baseline SES-CD (SES-CD <15 and SES-CD >=15); Adjusted risk difference from placebo = 8.7, 95% CI 2-sided [-8.7 to 26.1]

13. Secondary Outcome: Percentage of Participants Taking Corticosteroids at Baseline Who Discontinued Corticosteroid Use and Achieve Clinical Remission at Week 16
Description: as for outcome 2
Time Frame: Week 16
Population: as for outcome 11
Measure: Number; unit: percentage of participants
Arm/Group | Double-Blind Induction Phase: Placebo BID | Double-Blind Induction Phase: Upadacitinib 3 mg BID | Double-Blind Induction Phase: Upadacitinib 6 mg BID | Double Blind Induction Phase: Upadacitinib 12 mg BID | Double Blind Induction Phase: Upadacitinib 24 mg BID | Double Blind Induction Phase: Upadacitinib 24 mg QD
Number analyzed (Participants) | 15 | 21 | 18 | 17 | 15 | 10
percentage of participants | 0.0 | 14.3 | 22.2 | 11.8 | 33.3 | 10.0
Statistical Analysis 1: Comparison: Double-Blind Induction Phase: Placebo BID vs Double-Blind Induction Phase: Upadacitinib 3 mg BID; Test type: Superiority; p = 0.195, Cochran-Mantel-Haenszel — Based on CMH test stratified by baseline SES-CD (SES-CD <15 and SES-CD >=15); Adjusted risk difference from placebo = 12.2, 95% CI 2-sided [-6.2 to 30.7]
Statistical Analysis 2: Comparison: Double-Blind Induction Phase: Placebo BID vs Double-Blind Induction Phase: Upadacitinib 6 mg BID; Test type: Superiority; p = 0.116, Cochran-Mantel-Haenszel — Based on CMH test stratified by baseline SES-CD (SES-CD <15 and SES-CD >=15); Adjusted risk difference from placebo = 17.9, 95% CI 2-sided [-4.4 to 40.1]
Statistical Analysis 3: Comparison: Double-Blind Induction Phase: Placebo BID vs Double Blind Induction Phase: Upadacitinib 12 mg BID; Test type: Superiority; p = 0.178, Cochran-Mantel-Haenszel — Based on CMH test stratified by baseline SES-CD (SES-CD <15 and SES-CD >=15); Adjusted risk difference from placebo = 12.8, 95% CI 2-sided [-5.8 to 31.5]
Statistical Analysis 4: Comparison: Double-Blind Induction Phase: Placebo BID vs Double Blind Induction Phase: Upadacitinib 24 mg BID; Test type: Superiority; p = 0.031, Cochran-Mantel-Haenszel — Based on CMH test stratified by baseline SES-CD (SES-CD <15 and SES-CD >=15); Adjusted risk difference from placebo = 30.4, 95% CI 2-sided [2.8 to 58.0]
Statistical Analysis 5: Comparison: Double-Blind Induction Phase: Placebo BID vs Double Blind Induction Phase: Upadacitinib 24 mg QD; Test type: Superiority; p = 0.121, Cochran-Mantel-Haenszel — Based on CMH test stratified by baseline SES-CD (SES-CD <15 and SES-CD >=15); Adjusted risk difference from placebo = 13.1, 95% CI 2-sided [-3.5 to 29.6]

14. Secondary Outcome: Percentage of Participants Taking Corticosteroids at Baseline Who Discontinued Corticosteroid Use and Achieve Endoscopic Remission at Week 12/16
Description: Endoscopic remission: SES-CD ≤ 4 and at least 2-point reduction versus Baseline and no subscore > 1 in any individual variable. Details of the SES-CD scale are provided in the description of the first primary endpoint.
Time Frame: as for outcome 1
Population: as for outcome 11
Measure: Number; unit: percentage of participants
Arm/Group | Double-Blind Induction Phase: Placebo BID | Double-Blind Induction Phase: Upadacitinib 3 mg BID | Double-Blind Induction Phase: Upadacitinib 6 mg BID | Double Blind Induction Phase: Upadacitinib 12 mg BID | Double Blind Induction Phase: Upadacitinib 24 mg BID | Double Blind Induction Phase: Upadacitinib 24 mg QD
Number analyzed (Participants) | 15 | 21 | 18 | 17 | 15 | 10
percentage of participants | 0.0 | 0.0 | 11.1 | 5.9 | 20.0 | 10.0
Statistical Analysis 1: Comparison: Double-Blind Induction Phase: Placebo BID vs Double-Blind Induction Phase: Upadacitinib 6 mg BID; Test type: Superiority; p = 0.392, Cochran-Mantel-Haenszel — Based on CMH test stratified by baseline SES-CD (SES-CD <15 and SES-CD >=15); Adjusted risk difference from placebo = 6.8, 95% CI 2-sided [-8.7 to 22.2]
Statistical Analysis 2: Comparison: Double-Blind Induction Phase: Placebo BID vs Double Blind Induction Phase: Upadacitinib 12 mg BID; Test type: Superiority; p = 0.584, Cochran-Mantel-Haenszel — Based on CMH test stratified by baseline SES-CD (SES-CD <15 and SES-CD >=15); Adjusted risk difference from placebo = 3.4, 95% CI 2-sided [-8.8 to 15.7]
Statistical Analysis 3: Comparison: Double-Blind Induction Phase: Placebo BID vs Double Blind Induction Phase: Upadacitinib 24 mg BID; Test type: Superiority; p = 0.199, Cochran-Mantel-Haenszel — Based on CMH test stratified by baseline SES-CD (SES-CD <15 and SES-CD >=15); Adjusted risk difference from placebo = 13.0, 95% CI 2-sided [-6.8 to 32.9]
Statistical Analysis 4: Comparison: Double-Blind Induction Phase: Placebo BID vs Double Blind Induction Phase: Upadacitinib 24 mg QD; Test type: Superiority; p = 0.439, Cochran-Mantel-Haenszel — Based on CMH test stratified by baseline SES-CD (SES-CD <15 and SES-CD >=15); Adjusted risk difference from placebo = 6.9, 95% CI 2-sided [-10.6 to 24.5]

15. Secondary Outcome: Change From Baseline in Fecal Calprotectin Level Over Time During the Induction Phase
Time Frame: Baseline, Week 4, Week 16
Population: mITT Population: all randomized participants who took at least 1 dose of study drug in the Induction Period. Includes only participants with an assessment at Baseline and Week 16 and with an assessment at given time point.
Measure: Mean (Standard Deviation); unit: μg/g
Arm/Group | Double-Blind Induction Phase: Placebo BID | Double-Blind Induction Phase: Upadacitinib 3 mg BID | Double-Blind Induction Phase: Upadacitinib 6 mg BID | Double Blind Induction Phase: Upadacitinib 12 mg BID | Double Blind Induction Phase: Upadacitinib 24 mg BID | Double Blind Induction Phase: Upadacitinib 24 mg QD
Number analyzed (Participants) | 28 | 26 | 31 | 28 | 25 | 26
μg/g
  Week 4 | 83.7 (1024.11) | -310.3 (2415.43) | -436.9 (1505.75) | -915.7 (1600.31) | -876.2 (2240.93) | -255.8 (2407.47)
  Week 16: number analyzed (Participants) | 18 | 21 | 21 | 19 | 12 | 19
  Week 16 | -128.9 (373.53) | -534.5 (3279.19) | -429.4 (2505.21) | -475.1 (2668.93) | -828.7 (986.09) | -698.4 (2228.85)
Statistical Analysis 1: Comparison: Double-Blind Induction Phase: Placebo BID vs Double-Blind Induction Phase: Upadacitinib 3 mg BID; Week 4; Test type: Superiority; p = 0.788, mixed-effect model repeated measure — P value for test of difference using the repeated measure model including treatment, Baseline disease severity (SES-CD < 15 and ≥ 15), week, Baseline, interaction of treatment and week; LS Mean Difference = -103.9, 95% CI 2-sided [-865.69 to 657.87]
Statistical Analysis 2: Comparison: Double-Blind Induction Phase: Placebo BID vs Double-Blind Induction Phase: Upadacitinib 6 mg BID; Week 4; Test type: Superiority; p = 0.325, mixed-effect model repeated measure — [p-value comment as in outcome 15, analysis 1]; LS Mean Difference = -364.3, 95% CI 2-sided [-1092.83 to 364.29]
Statistical Analysis 3: Comparison: Double-Blind Induction Phase: Placebo BID vs Double Blind Induction Phase: Upadacitinib 12 mg BID; Test type: Superiority; p = 0.015, mixed-effect model repeated measure — [p-value comment as in outcome 15, analysis 1]; LS Mean Difference = -926.2, 95% CI 2-sided [-1672.78 to -179.63]
Statistical Analysis 4: Comparison: Double-Blind Induction Phase: Placebo BID vs Double Blind Induction Phase: Upadacitinib 24 mg BID; Week 4; Test type: Superiority; p = 0.053, mixed-effect model repeated measure — [p-value comment as in outcome 15, analysis 1]; LS Mean Difference = -763.1, 95% CI 2-sided [-1534.52 to 8.39]
Statistical Analysis 5: Comparison: Double-Blind Induction Phase: Placebo BID vs Double Blind Induction Phase: Upadacitinib 24 mg QD; Week 4; Test type: Superiority; p = 0.352, mixed-effect model repeated measure — [p-value comment as in outcome 15, analysis 1]; LS Mean Difference = -359.5, 95% CI 2-sided [-1119.52 to 400.56]
Statistical Analysis 6: Comparison: Double-Blind Induction Phase: Placebo BID vs Double-Blind Induction Phase: Upadacitinib 3 mg BID; Week 16; Test type: Superiority; p = 0.503, mixed-effect model repeated measure — [p-value comment as in outcome 15, analysis 1]; LS Mean Difference = -396.2, 95% CI 2-sided [-1565.39 to 772.90]
Statistical Analysis 7: Comparison: Double-Blind Induction Phase: Placebo BID vs Double-Blind Induction Phase: Upadacitinib 6 mg BID; Week 16; Test type: Superiority; p = 0.537, mixed-effect model repeated measure — [p-value comment as in outcome 15, analysis 1]; LS Mean Difference = -364.3, 95% CI 2-sided [-1531.04 to 802.44]
Statistical Analysis 8: Comparison: Double-Blind Induction Phase: Placebo BID vs Double Blind Induction Phase: Upadacitinib 12 mg BID; Week 16; Test type: Superiority; p = 0.425, mixed-effect model repeated measure — [p-value comment as in outcome 15, analysis 1]; LS Mean Difference = -483.2, 95% CI 2-sided [-1677.87 to 711.52]
Statistical Analysis 9: Comparison: Double-Blind Induction Phase: Placebo BID vs Double Blind Induction Phase: Upadacitinib 24 mg BID; Week 16; Test type: Superiority; p = 0.134, mixed-effect model repeated measure — [p-value comment as in outcome 15, analysis 1]; LS Mean Difference = -1025.6, 95% CI 2-sided [-2373.24 to 322.08]
Statistical Analysis 10: Comparison: Double-Blind Induction Phase: Placebo BID vs Double Blind Induction Phase: Upadacitinib 24 mg QD; Week 16; Test type: Superiority; p = 0.293, mixed-effect model repeated measure — [p-value comment as in outcome 15, analysis 1]; LS Mean Difference = -637.9, 95% CI 2-sided [-1833.82 to 557.96]

16. Secondary Outcome: Change From Baseline in High-Sensitivity C-Reactive Protein (Hs-CRP) at Week 16
Time Frame: Baseline, Week 16
Population: mITT Population: all randomized participants who took at least 1 dose of study drug in the Induction Period. Includes only participants with an assessment at Baseline and Week 16.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Double-Blind Induction Phase: Placebo BID | Double-Blind Induction Phase: Upadacitinib 3 mg BID | Double-Blind Induction Phase: Upadacitinib 6 mg BID | Double Blind Induction Phase: Upadacitinib 12 mg BID | Double Blind Induction Phase: Upadacitinib 24 mg BID | Double Blind Induction Phase: Upadacitinib 24 mg QD
Number analyzed (Participants) | 29 | 35 | 34 | 31 | 27 | 32
mg/L | -0.1 (11.96) | -3.0 (19.60) | -3.9 (19.47) | -6.1 (27.02) | -14.8 (26.38) | -2.7 (13.74)
Statistical Analysis 1: Comparison: Double-Blind Induction Phase: Placebo BID vs Double-Blind Induction Phase: Upadacitinib 3 mg BID; Test type: Superiority; p = 0.921, mixed-effect model repeated measure — [p-value comment as in outcome 15, analysis 1]; LS Mean Difference = 0.5, 95% CI 2-sided [-9.02 to 9.97]
Statistical Analysis 2: Comparison: Double-Blind Induction Phase: Placebo BID vs Double-Blind Induction Phase: Upadacitinib 6 mg BID; Test type: Superiority; p = 0.75, mixed-effect model repeated measure — [p-value comment as in outcome 15, analysis 1]; LS Mean Difference = -1.6, 95% CI 2-sided [-11.19 to 8.08]
Statistical Analysis 3: Comparison: Double-Blind Induction Phase: Placebo BID vs Double Blind Induction Phase: Upadacitinib 12 mg BID; Test type: Superiority; p = 0.7, mixed-effect model repeated measure — [p-value comment as in outcome 15, analysis 1]; LS Mean Difference = -1.9, 95% CI 2-sided [-11.7 to 7.87]
Statistical Analysis 4: Comparison: Double-Blind Induction Phase: Placebo BID vs Double Blind Induction Phase: Upadacitinib 24 mg BID; Test type: Superiority; p = 0.024, mixed-effect model repeated measure — [p-value comment as in outcome 15, analysis 1]; LS Mean Difference = -11.4, 95% CI 2-sided [-21.38 to -1.51]
Statistical Analysis 5: Comparison: Double-Blind Induction Phase: Placebo BID vs Double Blind Induction Phase: Upadacitinib 24 mg QD; Test type: Superiority; p = 0.845, mixed-effect model repeated measure — [p-value comment as in outcome 15, analysis 1]; LS Mean Difference = -1.0, 95% CI 2-sided [-10.72 to 8.79]

17. Secondary Outcome: Change From Baseline in Inflammatory Bowel Disease Questionnaire (IBDQ) Over Time During the Induction Phase
Description: The IBDQ is a disease-specific instrument composed of 32 Likert-scaled items. The total score ranges from 32 to 224 using the 7-point response options, with higher scores indicating better health-related quality of life.
Time Frame: Baseline, Week 8, Week 16
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Double-Blind Induction Phase: Placebo BID | Double-Blind Induction Phase: Upadacitinib 3 mg BID | Double-Blind Induction Phase: Upadacitinib 6 mg BID | Double Blind Induction Phase: Upadacitinib 12 mg BID | Double Blind Induction Phase: Upadacitinib 24 mg BID | Double Blind Induction Phase: Upadacitinib 24 mg QD
Number analyzed (Participants) | 33 | 36 | 35 | 34 | 31 | 33
units on a scale
  Week 8 | 16.6 (25.38) | 18.9 (40.35) | 34.6 (36.22) | 24.9 (30.95) | 39.7 (40.76) | 23.3 (30.34)
  Week 16: number analyzed (Participants) | 29 | 35 | 33 | 28 | 29 | 32
  Week 16 | 14.5 (29.15) | 24.6 (42.98) | 41.8 (47.02) | 32.1 (38.57) | 44.4 (40.05) | 22.5 (27.82)
Statistical Analysis 1: Comparison: Double-Blind Induction Phase: Placebo BID vs Double-Blind Induction Phase: Upadacitinib 3 mg BID; Week 8; Test type: Superiority; p = 0.830, mixed-effect model repeated measure — [p-value comment as in outcome 15, analysis 1]; LS Mean Difference = 1.7, 95% CI 2-sided [-13.60 to 16.92]
Statistical Analysis 2: Comparison: Double-Blind Induction Phase: Placebo BID vs Double-Blind Induction Phase: Upadacitinib 6 mg BID; Week 8; Test type: Superiority; p = 0.027, mixed-effect model repeated measure — [p-value comment as in outcome 15, analysis 1]; LS Mean Difference = 17.5, 95% CI 2-sided [2.03 to 33.00]
Statistical Analysis 3: Comparison: Double-Blind Induction Phase: Placebo BID vs Double Blind Induction Phase: Upadacitinib 12 mg BID; Week 8; Test type: Superiority; p = 0.263, mixed-effect model repeated measure — [p-value comment as in outcome 15, analysis 1]; LS Mean Difference = 8.9, 95% CI 2-sided [-6.72 to 24.47]
Statistical Analysis 4: Comparison: Double-Blind Induction Phase: Placebo BID vs Double Blind Induction Phase: Upadacitinib 24 mg BID; Week 8; Test type: Superiority; p = 0.008, mixed-effect model repeated measure — [p-value comment as in outcome 15, analysis 1]; LS Mean Difference = 21.6, 95% CI 2-sided [5.68 to 37.52]
Statistical Analysis 5: Comparison: Double-Blind Induction Phase: Placebo BID vs Double Blind Induction Phase: Upadacitinib 24 mg QD; Week 8; Test type: Superiority; p = 0.269, mixed-effect model repeated measure — [p-value comment as in outcome 15, analysis 1]; LS Mean Difference = 8.8, 95% CI 2-sided [-6.88 to 24.53]
Statistical Analysis 6: Comparison: Double-Blind Induction Phase: Placebo BID vs Double-Blind Induction Phase: Upadacitinib 3 mg BID; Week 16; Test type: Superiority; p = 0.231, mixed-effect model repeated measure — [p-value comment as in outcome 15, analysis 1]; LS Mean Difference = 10.3, 95% CI 2-sided [-6.63 to 27.25]
Statistical Analysis 7: Comparison: Double-Blind Induction Phase: Placebo BID vs Double-Blind Induction Phase: Upadacitinib 6 mg BID; Test type: Superiority; p = 0.002, mixed-effect model repeated measure — [p-value comment as in outcome 15, analysis 1]; LS Mean Difference = 27.9, 95% CI 2-sided [10.68 to 45.15]
Statistical Analysis 8: Comparison: Double-Blind Induction Phase: Placebo BID vs Double Blind Induction Phase: Upadacitinib 12 mg BID; Week 16; Test type: Superiority; p = 0.057, mixed-effect model repeated measure — [p-value comment as in outcome 15, analysis 1]; LS Mean Difference = 17.1, 95% CI 2-sided [-0.51 to 34.72]
Statistical Analysis 9: Comparison: Double-Blind Induction Phase: Placebo BID vs Double Blind Induction Phase: Upadacitinib 24 mg BID; Week 16; Test type: Superiority; p = 0.002, mixed-effect model repeated measure — [p-value comment as in outcome 15, analysis 1]; LS Mean Difference = 28.8, 95% CI 2-sided [11.12 to 46.56]
Statistical Analysis 10: Comparison: Double-Blind Induction Phase: Placebo BID vs Double Blind Induction Phase: Upadacitinib 24 mg QD; Test type: Superiority; p = 0.165, mixed-effect model repeated measure — [p-value comment as in outcome 15, analysis 1]; LS Mean Difference = 12.3, 95% CI 2-sided [-5.12 to 29.72]

18. Secondary Outcome: Percentage of Participants With Isolated Ileal Crohn's Disease at Baseline Who Achieve Remission at Week 16
Description: Remission is defined as endoscopic remission AND clinical remission. Endoscopic remission: SES-CD ≤ 4 and at least 2-point reduction versus Baseline and no subscore > 1 in any individual variable. Clinical remission: average daily stool frequency ≤ 1.5 and not worse than Baseline AND average daily abdominal pain ≤ 1.0 and not worse than Baseline. The very soft/liquid stool frequency and abdominal pain scores at a visit were the average of the daily values reported during the 7 usable days preceding the scheduled assessment visit. Abdominal Pain was rated on a 4-point scale from 0 (none) to 3 (severe). Details of the SES-CD scale are provided in the description of the first primary endpoint.
Time Frame: Week 16
Population: mITT Population: all randomized participants who took at least 1 dose of study drug in the Induction Period. Only mITT participants with isolated ileal Crohn's disease at Baseline are included. Non-responder imputation.
Measure: Number; unit: percentage of participants
Arm/Group | Double-Blind Induction Phase: Placebo BID | Double-Blind Induction Phase: Upadacitinib 3 mg BID | Double-Blind Induction Phase: Upadacitinib 6 mg BID | Double Blind Induction Phase: Upadacitinib 12 mg BID | Double Blind Induction Phase: Upadacitinib 24 mg BID | Double Blind Induction Phase: Upadacitinib 24 mg QD
Number analyzed (Participants) | 9 | 10 | 6 | 5 | 6 | 10
percentage of participants | 0.0 | 20.0 | 16.7 | 20.0 | 0.0 | 20.0
Statistical Analysis 1: Comparison: Double-Blind Induction Phase: Placebo BID vs Double-Blind Induction Phase: Upadacitinib 3 mg BID; Test type: Superiority; p = 0.167, Cochran-Mantel-Haenszel — Based on CMH test stratified by baseline SES-CD (SES-CD <15 and SES-CD >=15); Adjusted risk difference from placebo = 20.0, 95% CI 2-sided [-8.4 to 48.4]
Statistical Analysis 2: Comparison: Double-Blind Induction Phase: Placebo BID vs Double-Blind Induction Phase: Upadacitinib 6 mg BID; Test type: Superiority; p = 0.221, Cochran-Mantel-Haenszel — Based on CMH test stratified by baseline SES-CD (SES-CD <15 and SES-CD >=15); Adjusted risk difference from placebo = 16.7, 95% CI 2-sided [-10.0 to 43.3]
Statistical Analysis 3: Comparison: Double-Blind Induction Phase: Placebo BID vs Double Blind Induction Phase: Upadacitinib 12 mg BID; Test type: Superiority; p = 0.18, Cochran-Mantel-Haenszel — Based on CMH test stratified by baseline SES-CD (SES-CD <15 and SES-CD >=15); Adjusted risk difference from placebo = 20.0, 95% CI 2-sided [-9.2 to 49.2]
Statistical Analysis 4: Comparison: Double-Blind Induction Phase: Placebo BID vs Double Blind Induction Phase: Upadacitinib 24 mg QD; Test type: Superiority; p = 0.167, Cochran-Mantel-Haenszel — Based on CMH test stratified by baseline SES-CD (SES-CD <15 and SES-CD >=15); LS Mean Difference = 20.0, 95% CI 2-sided [-8.4 to 48.4]

19. Secondary Outcome: Percentage of Participants With a Decrease in CDAI ≥ 100 Points From Baseline at Week 16
Description: CDAI is used to quantify the signs and symptoms of subjects with Crohn's disease. The score includes the frequency of stools, abdominal pain and general well-being as well as the presence of complications, use of antidiarrheals, presence of abdominal mass, hematocrit and weight. CDAI generally ranges from 0 to 600 where higher scores indicate more severe disease. A score below 150 indicates remission and a score above 450 indicates very severe disease.
Time Frame: Week 16
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Double-Blind Induction Phase: Placebo BID | Double-Blind Induction Phase: Upadacitinib 3 mg BID | Double-Blind Induction Phase: Upadacitinib 6 mg BID | Double Blind Induction Phase: Upadacitinib 12 mg BID | Double Blind Induction Phase: Upadacitinib 24 mg BID | Double Blind Induction Phase: Upadacitinib 24 mg QD
Number analyzed (Participants) | 37 | 39 | 37 | 36 | 36 | 35
percentage of participants | 27.0 | 33.3 | 40.5 | 44.4 | 55.6 | 31.4
Statistical Analysis 1: Comparison: Double-Blind Induction Phase: Placebo BID vs Double-Blind Induction Phase: Upadacitinib 3 mg BID; Test type: Superiority; p = 0.607, Cochran-Mantel-Haenszel — Based on CMH test stratified by baseline SES-CD (SES-CD <15 and SES-CD >=15); Adjusted risk difference from placebo = 5.5, 95% CI 2-sided [-15.5 to 26.5]
Statistical Analysis 2: Comparison: Double-Blind Induction Phase: Placebo BID vs Double-Blind Induction Phase: Upadacitinib 6 mg BID; Test type: Superiority; p = 0.272, Cochran-Mantel-Haenszel — Based on CMH test stratified by baseline SES-CD (SES-CD <15 and SES-CD >=15); Adjusted risk difference from placebo = 12.2, 95% CI 2-sided [-9.6 to 33.9]
Statistical Analysis 3: Comparison: Double-Blind Induction Phase: Placebo BID vs Double Blind Induction Phase: Upadacitinib 12 mg BID; Test type: Superiority; p = -0.157, Cochran-Mantel-Haenszel — Based on CMH test stratified by baseline SES-CD (SES-CD <15 and SES-CD >=15); Adjusted risk difference from placebo = 15.9, 95% CI 2-sided [-6.1 to 37.9]
Statistical Analysis 4: Comparison: Double-Blind Induction Phase: Placebo BID vs Double Blind Induction Phase: Upadacitinib 24 mg BID; Test type: Superiority; p = 0.017, Cochran-Mantel-Haenszel — Based on CMH test stratified by baseline SES-CD (SES-CD <15 and SES-CD >=15); LS Mean Difference = 27.7, 95% CI 2-sided [4.9 to 50.6]
Statistical Analysis 5: Comparison: Double-Blind Induction Phase: Placebo BID vs Double Blind Induction Phase: Upadacitinib 24 mg QD; Test type: Superiority; p = 0.798, Cochran-Mantel-Haenszel — Based on CMH test stratified by baseline SES-CD (SES-CD <15 and SES-CD >=15); Adjusted risk difference from placebo = 2.8, 95% CI 2-sided [-18.4 to 23.9]

20. Secondary Outcome: Percentage of Participants Who Achieve > 50% Reduction From Baseline in SES-CD or Endoscopic Remission at Week 12/16
Description: Endoscopic remission: SES-CD ≤ 4 and at least two point reduction versus Baseline and no subscore > 1 in any individual variable. Details of the SES-CD scale are provided in the description of the first primary endpoint.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Double-Blind Induction Phase: Placebo BID | Double-Blind Induction Phase: Upadacitinib 3 mg BID | Double-Blind Induction Phase: Upadacitinib 6 mg BID | Double Blind Induction Phase: Upadacitinib 12 mg BID | Double Blind Induction Phase: Upadacitinib 24 mg BID | Double Blind Induction Phase: Upadacitinib 24 mg QD
Number analyzed (Participants) | 37 | 39 | 37 | 36 | 36 | 35
percentage of participants | 2.7 | 12.8 | 18.9 | 25.0 | 36.1 | 25.7
Statistical Analysis 1: Comparison: Double-Blind Induction Phase: Placebo BID vs Double-Blind Induction Phase: Upadacitinib 3 mg BID; Test type: Superiority; p = 0.119, Cochran-Mantel-Haenszel — Based on CMH test stratified by baseline SES-CD (SES-CD <15 and SES-CD >=15); Adjusted risk difference from placebo = 9.8, 95% CI 2-sided [-2.5 to 22.1]
Statistical Analysis 2: Comparison: Double-Blind Induction Phase: Placebo BID vs Double-Blind Induction Phase: Upadacitinib 6 mg BID; Test type: Superiority; p = 0.034, Cochran-Mantel-Haenszel — Based on CMH test stratified by baseline SES-CD (SES-CD <15 and SES-CD >=15); Adjusted risk difference from placebo = 15.4, 95% CI 2-sided [1.1 to 29.7]
Statistical Analysis 3: Comparison: Double-Blind Induction Phase: Placebo BID vs Double Blind Induction Phase: Upadacitinib 12 mg BID; Test type: Superiority; p = 0.004, Cochran-Mantel-Haenszel — Based on CMH test stratified by baseline SES-CD (SES-CD <15 and SES-CD >=15); Adjusted risk difference from placebo = 23.2, 95% CI 2-sided [7.3 to 39.2]
Statistical Analysis 4: Comparison: Double-Blind Induction Phase: Placebo BID vs Double Blind Induction Phase: Upadacitinib 24 mg BID; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — Based on CMH test stratified by baseline SES-CD (SES-CD <15 and SES-CD >=15); Adjusted risk difference from placebo = 32.4, 95% CI 2-sided [14.2 to 50.5]
Statistical Analysis 5: Comparison: Double-Blind Induction Phase: Placebo BID vs Double Blind Induction Phase: Upadacitinib 24 mg QD; Test type: Superiority; p < 0.006, Cochran-Mantel-Haenszel — Based on CMH test stratified by baseline SES-CD (SES-CD <15 and SES-CD >=15); Adjusted risk difference from placebo = 22.9, 95% CI 2-sided [6.6 to 39.2]

21. Secondary Outcome: Percentage of Participants Who Achieve Modified Clinical Remission at Week 16 Among Participants With an Average Daily Stool Frequency ≥ 4.0 or Average Daily Abdominal Pain ≥ 2.0 at Baseline
Description: Modified clinical remission was defined as average daily stool frequency <= 2.8 and not worse than Baseline and average daily abdominal pain <= 1.0 and not worse than Induction Baseline. The very soft/liquid stool frequency and abdominal pain scores at a visit were the average of the daily values reported during the 7 usable days preceding the scheduled assessment visit. Abdominal Pain was rated on a 4-point scale from 0 (none) to 3 (severe).
Time Frame: Week 16
Population: mITT Population: all randomized participants who took at least 1 dose of study drug in the Induction Period. Includes only mITT participants with an average daily stool frequency ≥ 4.0 or average daily abdominal pain ≥ 2.0 at Baseline. Non-responder imputation.
Measure: Number; unit: percentage of participants
Arm/Group | Double-Blind Induction Phase: Placebo BID | Double-Blind Induction Phase: Upadacitinib 3 mg BID | Double-Blind Induction Phase: Upadacitinib 6 mg BID | Double Blind Induction Phase: Upadacitinib 12 mg BID | Double Blind Induction Phase: Upadacitinib 24 mg BID | Double Blind Induction Phase: Upadacitinib 24 mg QD
Number analyzed (Participants) | 33 | 38 | 33 | 34 | 30 | 32
percentage of participants | 12.1 | 15.8 | 30.3 | 26.5 | 36.7 | 18.8
Statistical Analysis 1: Comparison: Double-Blind Induction Phase: Placebo BID vs Double-Blind Induction Phase: Upadacitinib 3 mg BID; Test type: Superiority; p = 0.647, Cochran-Mantel-Haenszel — Based on CMH test stratified by baseline SES-CD (SES-CD <15 and SES-CD >=15); Adjusted risk difference from placebo = 3.9, 95% CI 2-sided [-12.7 to 20.5]
Statistical Analysis 2: Comparison: Double-Blind Induction Phase: Placebo BID vs Double-Blind Induction Phase: Upadacitinib 6 mg BID; Test type: Superiority; p = 0.093, Cochran-Mantel-Haenszel — Based on CMH test stratified by baseline SES-CD (SES-CD <15 and SES-CD >=15); Adjusted risk difference from placebo = 17.1, 95% CI 2-sided [-2.9 to 37.1]
Statistical Analysis 3: Comparison: Double-Blind Induction Phase: Placebo BID vs Double Blind Induction Phase: Upadacitinib 12 mg BID; Test type: Superiority; p = 0.165, Cochran-Mantel-Haenszel — Based on CMH test stratified by baseline SES-CD (SES-CD <15 and SES-CD >=15); Adjusted risk difference from placebo = 13.6, 95% CI 2-sided [-5.6 to 32.8]
Statistical Analysis 4: Comparison: Double-Blind Induction Phase: Placebo BID vs Double Blind Induction Phase: Upadacitinib 24 mg BID; Test type: Superiority; p = 0.023, Cochran-Mantel-Haenszel — Based on CMH test stratified by baseline SES-CD (SES-CD <15 and SES-CD >=15); Adjusted risk difference from placebo = 24.9, 95% CI 2-sided [3.4 to 46.3]
Statistical Analysis 5: Comparison: Double-Blind Induction Phase: Placebo BID vs Double Blind Induction Phase: Upadacitinib 24 mg QD; Test type: Superiority; p = 0.448, Cochran-Mantel-Haenszel — Based on CMH test stratified by baseline SES-CD (SES-CD <15 and SES-CD >=15); Adjusted risk difference from placebo = 7.0, 95% CI 2-sided [-11.0 to 25.0]

22. Secondary Outcome: Change From Baseline in Abdominal Pain Rating Scale at Week 12
Description: Abdominal pain was assessed on an abdominal pain rating scale, where subjects rated their average abdominal pain over the last 24 hours on a scale of 0 (none) to 10 (worst pain imaginable).
Time Frame: Baseline, Week 12
Population: mITT Population: all randomized participants who took at least 1 dose of study drug in the Induction Period. Includes only mITT participants with an assessment at baseline and given time point. Non-responder imputation.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Double-Blind Induction Phase: Placebo BID | Double-Blind Induction Phase: Upadacitinib 3 mg BID | Double-Blind Induction Phase: Upadacitinib 6 mg BID | Double Blind Induction Phase: Upadacitinib 12 mg BID | Double Blind Induction Phase: Upadacitinib 24 mg BID | Double Blind Induction Phase: Upadacitinib 24 mg QD
Number analyzed (Participants) | 30 | 35 | 34 | 27 | 29 | 30
units on a scale | -1.1 (1.84) | -1.0 (2.61) | -2.6 (2.53) | -2.4 (3.17) | -2.7 (2.52) | -1.0 (1.99)
Statistical Analysis 1: Comparison: Double-Blind Induction Phase: Placebo BID vs Double-Blind Induction Phase: Upadacitinib 3 mg BID; Test type: Superiority; p = 0.412, mixed-effect model repeated measure — [p-value comment as in outcome 15, analysis 1]; LS Mean Difference = 0.4, 95% CI 2-sided [-0.62 to 1.5]
Statistical Analysis 2: Comparison: Double-Blind Induction Phase: Placebo BID vs Double-Blind Induction Phase: Upadacitinib 6 mg BID; Test type: Superiority; p = 0.01, mixed-effect model repeated measure — [p-value comment as in outcome 15, analysis 1]; LS Mean Difference = -1.4, 95% CI 2-sided [-2.47 to -0.34]
Statistical Analysis 3: Comparison: Double-Blind Induction Phase: Placebo BID vs Double Blind Induction Phase: Upadacitinib 12 mg BID; Test type: Superiority; p = 0.082, mixed-effect model repeated measure — [p-value comment as in outcome 15, analysis 1]; LS Mean Difference = -1.0, 95% CI 2-sided [-2.13 to 0.13]
Statistical Analysis 4: Comparison: Double-Blind Induction Phase: Placebo BID vs Double Blind Induction Phase: Upadacitinib 24 mg BID; Test type: Superiority; p = 0.004, mixed-effect model repeated measure — [p-value comment as in outcome 15, analysis 1]; LS Mean Difference = -1.6, 95% CI 2-sided [-2.73 to -0.52]
Statistical Analysis 5: Comparison: Double-Blind Induction Phase: Placebo BID vs Double Blind Induction Phase: Upadacitinib 24 mg QD; Test type: Superiority; p = 0.766, mixed-effect model repeated measure — [p-value comment as in outcome 15, analysis 1]; LS Mean Difference = 0.2, 95% CI 2-sided [-0.93 to 1.26]

23. Secondary Outcome: Change From Baseline in Abdominal Pain Rating Scale at Week 16
Description: as for outcome 22
Time Frame: Baseline, Week 16
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Double-Blind Induction Phase: Placebo BID | Double-Blind Induction Phase: Upadacitinib 3 mg BID | Double-Blind Induction Phase: Upadacitinib 6 mg BID | Double Blind Induction Phase: Upadacitinib 12 mg BID | Double Blind Induction Phase: Upadacitinib 24 mg BID | Double Blind Induction Phase: Upadacitinib 24 mg QD
Number analyzed (Participants) | 28 | 34 | 33 | 26 | 28 | 28
units on a scale | -0.9 (2.27) | -1.7 (3.02) | -2.8 (2.77) | -1.7 (2.86) | -2.3 (2.42) | -1.4 (2.15)
Statistical Analysis 1: Comparison: Double-Blind Induction Phase: Placebo BID vs Double-Blind Induction Phase: Upadacitinib 3 mg BID; Test type: Superiority; p = 0.314, mixed-effect model repeated measure — [p-value comment as in outcome 15, analysis 1]; LS Mean Difference = -0.6, 95% CI 2-sided [-1.75 to 0.56]
Statistical Analysis 2: Comparison: Double-Blind Induction Phase: Placebo BID vs Double-Blind Induction Phase: Upadacitinib 6 mg BID; Test type: Superiority; p = 0.002, mixed-effect model repeated measure — [p-value comment as in outcome 15, analysis 1]; LS Mean Difference = -1.8, 95% CI 2-sided [-3.01 to -0.68]
Statistical Analysis 3: Comparison: Double-Blind Induction Phase: Placebo BID vs Double Blind Induction Phase: Upadacitinib 12 mg BID; Test type: Superiority; p = 0.255, mixed-effect model repeated measure — [p-value comment as in outcome 15, analysis 1]; LS Mean Difference = -0.7, 95% CI 2-sided [-1.94 to 0.52]
Statistical Analysis 4: Comparison: Double-Blind Induction Phase: Placebo BID vs Double Blind Induction Phase: Upadacitinib 24 mg BID; Test type: Superiority; p = 0.022, mixed-effect model repeated measure — [p-value comment as in outcome 15, analysis 1]; LS Mean Difference = -1.4, 95% CI 2-sided [-2.61 to -0.2]
Statistical Analysis 5: Comparison: Double-Blind Induction Phase: Placebo BID vs Double Blind Induction Phase: Upadacitinib 24 mg QD; Test type: Superiority; p = 0.239, mixed-effect model repeated measure — [p-value comment as in outcome 15, analysis 1]; LS Mean Difference = -0.7, 95% CI 2-sided [-1.92 to 0.48]

24. Secondary Outcome: Percentage of Participants Who Achieve Remission at Week 52
Description: Remission at Week 52 was defined as both endoscopic remission at Week 52 and clinical remission at Week 52. Endoscopic remission: SES-CD ≤ 4 and at least 2-point reduction versus Baseline and no subscore > 1 in any individual variable. Clinical remission: average daily stool frequency ≤ 1.5 and not worse than Baseline AND average daily abdominal pain ≤ 1.0 and not worse than Baseline. The very soft/liquid stool frequency and abdominal pain scores at a visit were the average of the daily values reported during the 7 usable days preceding the scheduled assessment visit. Abdominal Pain was rated on a 4-point scale from 0 (none) to 3 (severe). See SES-CD description details in the first primary endpoint description of this record. See definitions of responder and clinical responder in Outcome Measure 7 of this record.
Time Frame: Week 52
Population: Includes intent-to-treat responder (ITT-R) and non-responder (ITT-NR) analysis sets: all re-randomized participants in the double-blind Extension Phase who were responders and nonresponders at Week 16 of the Induction Period, respectively. Non responder imputation.
Measure: Number; unit: percentage of participants
Groups:
- Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction: Upadacitinib 3 mg BID during the 36-week double-blind Extension Phase. Upadacitinib in Induction Phase.
- Upadacitinib 6 mg BID in Extension/Upadacitinib in Induction: Upadacitinib 6 mg BID during the 36-week double-blind Extension Phase. Upadacitinib in Induction Phase.
- Upadacitinib 12 mg BID in Extension/Upadacitinib in Induction: Upadacitinib 12 mg BID during the 36-week double-blind Extension Phase. Upadacitinib in Induction Phase.
- Upadacitinib 24 mg QD in Extension/Upadacitinib in Induction: Upadacitinib 24 mg QD (consisting of two 12 mg IR doses) during the 36-week double-blind Extension Phase. Upadacitinib in Induction.
- Upadacitinib 3 mg BID in Extension/Placebo in Induction: Upadacitinib 3 mg BID during the 36-week double-blind Extension Phase. Placebo in Induction Phase.
- Upadacitinib 6 mg BID in Extension/Placebo in Induction: Upadacitinib 6 mg BID during the 36-week double-blind Extension Phase. Placebo in Induction Phase.
- Upadacitinib 12 mg BID in Extension/Placebo in Induction: Upadacitinib 12 mg BID during the 36-week double-blind Extension Phase. Placebo in Induction Phase.
- Upadacitinib 24 mg QD in Extension/Placebo in Induction: Upadacitinib 24 mg QD (consisting of two 12 mg IR doses) during the 36-week double-blind Extension Phase. Placebo in Induction.
Arm/Group | Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction | Upadacitinib 6 mg BID in Extension/Upadacitinib in Induction | Upadacitinib 12 mg BID in Extension/Upadacitinib in Induction | Upadacitinib 24 mg QD in Extension/Upadacitinib in Induction | Upadacitinib 3 mg BID in Extension/Placebo in Induction | Upadacitinib 6 mg BID in Extension/Placebo in Induction | Upadacitinib 12 mg BID in Extension/Placebo in Induction | Upadacitinib 24 mg QD in Extension/Placebo in Induction
Number analyzed (Participants) | 52 | 18 | 50 | 33 | 9 | 5 | 9 | 4
percentage of participants
  Responders: number analyzed (Participants) | 20 | 8 | 16 | 10 | 1 | 0 | 0 | 0
  Responders | 20.0 | 12.5 | 25.0 | 0.0 | 0.0 |  |  |
  Non-Responders: number analyzed (Participants) | 32 | 10 | 34 | 23 | 8 | 5 | 9 | 4
  Non-Responders | 0.0 | 0.0 | 2.9 | 13.0 | 0.0 | 0.0 | 0.0 | 25.0
  Clinical Responders: number analyzed (Participants) | 32 | 14 | 29 | 19 | 6 | 1 | 4 | 1
  Clinical Responders | 12.5 | 7.1 | 13.8 | 15.8 | 0.0 | 0.0 | 0.0 | 100
  Clinical Non-Responders: number analyzed (Participants) | 20 | 4 | 21 | 14 | 3 | 4 | 5 | 3
  Clinical Non-Responders | 0.0 | 0.0 | 4.8 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
Statistical Analysis 1: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/Upadacitinib in Induction; Responders; Test type: Superiority; p = 1.000, Chi-squared — P value was calculated based on chi-square test (or Fisher's exact test if >= 20% of the cells have expected cell count < 5); Risk Difference (RD) = -7.5, 95% CI 2-sided [-36.4 to 21.4] — Risk difference = upadacitinib higher dose - upadacitinib lower dose. 95% confidence intervals for risk difference were calculated based on normal approximation using proc freq
Statistical Analysis 2: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/Upadacitinib in Induction; Responders; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 24, analysis 1]; Risk Difference (RD) = 5.0, 95% CI 2-sided [-22.5 to 32.5] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 3: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/Upadacitinib in Induction; Responders; Test type: Superiority; p = 0.272, Chi-squared — [p-value comment as in outcome 24, analysis 1]; Risk Difference (RD) = -20.0, 95% CI 2-sided [-37.5 to -2.5] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 4: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/Upadacitinib in Induction; Non-responders; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 24, analysis 1]; Risk Difference (RD) = 2.9, 95% CI 2-sided [-2.7 to 8.6] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 5: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/Upadacitinib in Induction; Non-responders; Test type: Superiority; p = 0.068, Chi-squared — [p-value comment as in outcome 24, analysis 1]; Risk Difference (RD) = 13.0, 95% CI 2-sided [-0.7 to 26.8] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 6: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/Upadacitinib in Induction; Clinical responders; Test type: Superiority; p = 1.0000, Chi-squared — [p-value comment as in outcome 24, analysis 1]; Risk Difference (RD) = -5.4, 95% CI 2-sided [-23.1 to 12.3] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 7: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/Upadacitinib in Induction; Clinical responders; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 24, analysis 1]; Risk Difference (RD) = 1.3, 95% CI 2-sided [-15.7 to 18.3] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 8: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/Upadacitinib in Induction; Clinical responders; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 24, analysis 1]; Risk Difference (RD) = 3.3, 95% CI 2-sided [-16.7 to 23.3] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 9: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/Upadacitinib in Induction; Clinical non-responders; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 24, analysis 1]; Risk Difference (RD) = 4.8, 95% CI 2-sided [-4.3 to 13.9] — [estimate comment as in outcome 24, analysis 1]

25. Secondary Outcome: Percentage of Participants Who Achieve Endoscopic Remission at Week 52
Description: as for outcome 14
Time Frame: Week 52
Population: as for outcome 24
Measure: Number; unit: percentage of participants
Groups:
- Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction: Upadacitinib 6 mg BID during the 36-week double-blind Extension Phase. Upadacitinib in Induction Phase.
- Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction: Upadacitinib 12 mg BID during the 36-week double-blind Extension Phase. Upadacitinib in Induction Phase.
- Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction: Upadacitinib 24 mg QD (consisting of two 12 mg IR doses) during the 36-week double-blind Extension Phase.
  Upadacitinib in Induction.
- Upadacitinib 3 mg BID in Extension/ Placebo in Induction: Upadacitinib 3 mg BID during the 36-week double-blind Extension Phase. Placebo in Induction Phase.
- Upadacitinib 6 mg BID in Extension/ Placebo in Induction: Upadacitinib 6 mg BID during the 36-week double-blind Extension Phase. Placebo in Induction Phase.
- Upadacitinib 12 mg BID in Extension/ Placebo in Induction: Upadacitinib 12 mg BID during the 36-week double-blind Extension Phase. Placebo in Induction Phase.
- Upadacitinib 24 mg QD in Extension/ Placebo in Induction: Upadacitinib 24 mg QD (consisting of two 12 mg IR doses) during the 36-week double-blind Extension Phase.
  Placebo in Induction.
Arm/Group | Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction | Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction | Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction | Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction | Upadacitinib 3 mg BID in Extension/ Placebo in Induction | Upadacitinib 6 mg BID in Extension/ Placebo in Induction | Upadacitinib 12 mg BID in Extension/ Placebo in Induction | Upadacitinib 24 mg QD in Extension/ Placebo in Induction
Number analyzed (Participants) | 52 | 18 | 50 | 33 | 9 | 5 | 9 | 4
percentage of participants
  Responders: number analyzed (Participants) | 20 | 8 | 16 | 10 | 1 | 0 | 0 | 0
  Responders | 25.0 | 25.0 | 37.5 | 10.0 | 0 |  |  |
  Non-Responders: number analyzed (Participants) | 32 | 10 | 34 | 23 | 8 | 5 | 9 | 4
  Non-Responders | 3.1 | 10.0 | 8.8 | 17.4 | 0 | 0 | 0 | 25.0
  Clinical Responders: number analyzed (Participants) | 32 | 14 | 29 | 19 | 6 | 1 | 4 | 1
  Clinical Responders | 15.6 | 21.4 | 24.1 | 26.3 | 0 | 0 | 0 | 100
  Clinical Non-Responders: number analyzed (Participants) | 20 | 4 | 21 | 14 | 3 | 4 | 5 | 3
  Clinical Non-Responders | 5.0 | 0 | 9.5 | 0 | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Responders; Test type: Superiority; p = 1.000, Chi-squared — P-value was calculated based on chi-square test (or Fisher's exact test if >= 20% of the cells had expected cell count < 5); Risk Difference (RD) = 0.0, 95% CI 2-sided [-35.5 to 35.5] — Risk difference = (upadacitinib higher dose - upadacitinib 3 mg BID). 95% confidence intervals for risk difference were calculated based on normal approximation using proc FREQ
Statistical Analysis 2: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Responders; Test type: Superiority; p = 0.483, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 12.5, 95% CI 2-sided [-17.9 to 42.9] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 3: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Responders; Test type: Superiority; p = 0.633, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -15.0, 95% CI 2-sided [-41.6 to 11.6] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 4: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Non-responders; Test type: Superiority; p = 0.424, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 6.9, 95% CI 2-sided [-12.7 to 26.4] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 5: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Non-responders; Test type: Superiority; p = 0.614, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 5.7, 95% CI 2-sided [-5.6 to 17.0] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 6: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Non-responders; Test type: Superiority; p = 0.149, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 14.3, 95% CI 2-sided [-2.4 to 30.9] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 7: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical responders; Test type: Superiority; p = 0.684, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 5.8, 95% CI 2-sided [-19.1 to 30.7] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 8: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical responders; Test type: Superiority; p = 0.404, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 8.5, 95% CI 2-sided [-11.5 to 28.5] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 9: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical responders; Test type: Superiority; p = 0.470, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 10.7, 95% CI 2-sided [-12.8 to 34.1] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 10: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical non-responders; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -5.0, 95% CI 2-sided [-14.6 to 4.6] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 11: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical non-responders; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 4.5, 95% CI 2-sided [-11.3 to 20.3] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 12: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical non-responders; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -5.0, 95% CI 2-sided [-14.6 to 4.6] — [estimate comment as in outcome 25, analysis 1]

26. Secondary Outcome: Percentage of Participants Who Achieve Both Endoscopic Remission and Modified Clinical Remission at Week 52 Among Subjects With Daily Stool Frequency ≥ 4.0 or Daily Abdominal Pain ≥ 2.0 at Induction Baseline
Description: Endoscopic remission was defined as SES-CD <= 4 and at least 2 points reduction versus induction baseline and no subscore > 1 in any individual variable. Modified clinical remission was defined as average daily stool frequency <= 2.8 and not worse than induction baseline AND average daily abdominal pain <= 1.0 and not worse than induction baseline. The very soft/liquid stool frequency and abdominal pain scores at a visit were the average of the daily values reported during the 7 usable days preceding the scheduled assessment visit. Abdominal Pain was rated on a 4-point scale from 0 (none) to 3 (severe). See SES-CD description details in the first primary endpoint description of this record.
Time Frame: Week 52
Population: Includes intent-to-treat responder (ITT-R) and non-responder (ITT-NR) analysis sets: all re-randomized participants in the double-blind Extension Phase who were responders and nonresponders at Week 16 of the Induction Period, respectively. Participants with daily stool frequency >= 4.0 or daily abdominal pain >= 2.0 at Induction Baseline. Non responder imputation
Measure: Number; unit: percentage of participants
Arm/Group | Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction | Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction | Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction | Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction | Upadacitinib 3 mg BID in Extension/ Placebo in Induction | Upadacitinib 6 mg BID in Extension/ Placebo in Induction | Upadacitinib 12 mg BID in Extension/ Placebo in Induction | Upadacitinib 24 mg QD in Extension/ Placebo in Induction
Number analyzed (Participants) | 45 | 17 | 48 | 30 | 8 | 5 | 8 | 4
percentage of participants
  Responders: number analyzed (Participants) | 17 | 8 | 15 | 10 | 1 | 0 | 0 | 0
  Responders | 29.4 | 12.5 | 33.3 | 10.0 | 0 |  |  |
  Non-responders: number analyzed (Participants) | 28 | 9 | 33 | 20 | 7 | 5 | 8 | 4
  Non-responders | 0 | 0 | 6.1 | 15.0 | 0 | 0 | 0 | 25.0
  Clinical responders: number analyzed (Participants) | 28 | 14 | 27 | 18 | 5 | 1 | 3 | 1
  Clinical responders | 17.9 | 7.1 | 22.2 | 22.2 | 0 | 0 | 0 | 100
  Clinical non-responders: number analyzed (Participants) | 17 | 3 | 21 | 12 | 3 | 4 | 5 | 3
  Clinical non-responders | 0 | 0 | 4.8 | 0 | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Responders; Test type: Superiority; p = 0.624, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -16.9, 95% CI 2-sided [-48.4 to 14.6] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 2: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Responders; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 3.9, 95% CI 2-sided [-28.3 to 36.1] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 3: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Responders; Test type: Superiority; p = 0.363, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -19.4, 95% CI 2-sided [-48.0 to 9.1] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 4: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Non-responders; Test type: Superiority; p = 0.495, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 6.1, 95% CI 2-sided [-2.1 to 14.2] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 5: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Non-responders; Test type: Superiority; p = 0.066, Chi-squared — P-value was calculated based on chi-square test (or Fisher's exact test if >= 20% of the cells had expected cell count < 5). Prespecified significance at the 0.1 level; Risk Difference (RD) = 15.0, 95% CI 2-sided [-0.6 to 30.6] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 6: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical responders; Test type: Superiority; p = 0.645, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -10.7, 95% CI 2-sided [-30.3 to 8.9] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 7: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical responders; Test type: Superiority; p = 0.686, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 4.4, 95% CI 2-sided [-16.8 to 25.5] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 8: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical responders; Test type: Superiority; p = 0.721, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 4.4, 95% CI 2-sided [-19.5 to 28.2] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 9: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical non-responders; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 4.8, 95% CI 2-sided [-4.3 to 13.9] — [estimate comment as in outcome 25, analysis 1]

27. Secondary Outcome: Percentage of Participants Who Achieve Clinical Remission Over Time During Extension Phase in Participants Receiving Upadacitinib in Induction
Description: Clinical remission was defined as average daily stool frequency <= 1.5 and not worse than Induction Baseline and average daily abdominal pain <= 1.0 and not worse than Induction Baseline. The very soft/liquid stool frequency and abdominal pain scores at a visit were the average of the daily values reported during the 7 usable days preceding the scheduled assessment visit. Abdominal Pain was rated on a 4-point scale from 0 (none) to 3 (severe).
Time Frame: Week 20, Week 28, Week 36, Week 44, Week 52
Population: Includes intent-to-treat responder (ITT-R) and non-responder (ITT-NR) analysis sets: all re-randomized participants in the double-blind Extension Phase who were responders and nonresponders at Week 16 of the Induction Period, respectively. Non responder imputation. Participants with an assessment at given time point.
Measure: Number; unit: percentage of participants
Arm/Group | Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction | Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction | Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction | Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction
Number analyzed (Participants) | 52 | 18 | 50 | 33
percentage of participants
  Responders, Week 20: number analyzed (Participants) | 20 | 8 | 16 | 10
  Responders, Week 20 | 45.0 | 37.5 | 50.0 | 40.0
  Responders, Week 28: number analyzed (Participants) | 20 | 8 | 16 | 10
  Responders, Week 28 | 45.0 | 37.5 | 56.3 | 50.0
  Responders, Week 36: number analyzed (Participants) | 20 | 8 | 16 | 10
  Responders, Week 36 | 40.0 | 37.5 | 62.5 | 30.0
  Responders, Week 44: number analyzed (Participants) | 20 | 8 | 16 | 10
  Responders, Week 44 | 40.0 | 12.5 | 68.8 | 40.0
  Responders, Week 52: number analyzed (Participants) | 20 | 8 | 16 | 10
  Responders, Week 52 | 30.0 | 37.5 | 62.5 | 30.0
  Non-responders, Week 20: number analyzed (Participants) | 32 | 10 | 34 | 23
  Non-responders, Week 20 | 12.5 | 40.0 | 8.8 | 8.7
  Non-responders, Week 28: number analyzed (Participants) | 32 | 10 | 34 | 23
  Non-responders, Week 28 | 12.5 | 40.0 | 8.8 | 13.0
  Non-responders, Week 36: number analyzed (Participants) | 32 | 10 | 34 | 23
  Non-responders, Week 36 | 9.4 | 10.0 | 2.9 | 13.0
  Non-responders, Week 44: number analyzed (Participants) | 32 | 10 | 34 | 23
  Non-responders, Week 44 | 12.5 | 20.0 | 5.9 | 8.7
  Non-responders, Week 52: number analyzed (Participants) | 32 | 10 | 34 | 23
  Non-responders, Week 52 | 9.4 | 10.0 | 8.8 | 13.0
  Clinical responders, Week 20: number analyzed (Participants) | 32 | 14 | 29 | 19
  Clinical responders, Week 20 | 40.6 | 50.0 | 37.9 | 31.6
  Clinical responders, Week 28: number analyzed (Participants) | 32 | 14 | 29 | 19
  Clinical responders, Week 28 | 37.5 | 50.0 | 41.4 | 42.1
  Clinical responders, Week 36: number analyzed (Participants) | 32 | 14 | 29 | 19
  Clinical responders, Week 36 | 34.4 | 28.6 | 37.9 | 31.9
  Clinical responders, Week 44: number analyzed (Participants) | 32 | 14 | 29 | 19
  Clinical responders, Week 44 | 34.4 | 21.4 | 44.8 | 31.6
  Clinical responders, Week 52: number analyzed (Participants) | 32 | 14 | 29 | 19
  Clinical responders, Week 52 | 25.0 | 28.6 | 41.4 | 31.6
  Clinical non-responders, Week 20: number analyzed (Participants) | 20 | 4 | 21 | 14
  Clinical non-responders, Week 20 | 0 | 0 | 0 | 0
  Clinical non-responders, Week 28: number analyzed (Participants) | 20 | 4 | 21 | 14
  Clinical non-responders, Week 28 | 5.0 | 0 | 0 | 0
  Clinical non-responders, Week 36: number analyzed (Participants) | 20 | 4 | 21 | 14
  Clinical non-responders, Week 36 | 0 | 0 | 0 | 0
  Clinical non-responders, Week 44: number analyzed (Participants) | 20 | 4 | 21 | 14
  Clinical non-responders, Week 44 | 5.0 | 0 | 0 | 0
  Clinical non-responders, Week 52: number analyzed (Participants) | 20 | 4 | 21 | 14
  Clinical non-responders, Week 52 | 5.0 | 0 | 4.8 | 0
Statistical Analysis 1: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 20; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -7.5, 95% CI 2-sided [-47.5 to 32.5] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 2: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 20; Test type: Superiority; p = 0.765, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 5.0, 95% CI 2-sided [-27.8 to 37.8] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 3: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Responders, Week 20; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -5.0, 95% CI 2-sided [-42.4 to 32.4] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 4: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 28; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -7.5, 95% CI 2-sided [-47.5 to 32.5] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 5: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 28; Test type: Superiority; p = 0.502, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 11.3, 95% CI 2-sided [-21.4 to 43.9] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 6: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Responders, Week 28; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 5.0, 95% CI 2-sided [-32.9 to 42.9] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 7: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 36; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -2.5, 95% CI 2-sided [-42.3 to 37.3] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 8: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 36; Test type: Superiority; p = 0.180, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 22.5, 95% CI 2-sided [-9.5 to 54.5] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 9: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Responders, Week 36; Test type: Superiority; p = 0.702, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -10.0, 95% CI 2-sided [-45.6 to 25.6] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 10: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 44; Test type: Superiority; p = 0.214, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -27.5, 95% CI 2-sided [-58.9 to 3.9] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 11: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 44; Test type: Superiority; p = 0.086, Chi-squared — P-value was calculated based on chi-square test (or Fisher's exact test if >= 20% of the cells had expected cell count < 5). Prespecified statistical significance at the 0.1 level; Risk Difference (RD) = 28.8, 95% CI 2-sided [-2.5 to 60.0] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 12: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Responders, Week 44; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 0.0, 95% CI 2-sided [-37.2 to 37.2] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 13: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 52; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 7.5, 95% CI 2-sided [-31.6 to 46.6] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 14: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 52; Test type: Superiority; p = 0.051, Chi-squared — [p-value comment as in outcome 27, analysis 11]; Risk Difference (RD) = 32.5, 95% CI 2-sided [1.4 to 63.6] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 15: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Responders, Week 52; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 0.0, 95% CI 2-sided [-34.8 to 34.8] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 16: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 20; Test type: Superiority; p = 0.075, Chi-squared — [p-value comment as in outcome 27, analysis 11]; Risk Difference (RD) = 27.5, 95% CI 2-sided [-5.0 to 60.0] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 17: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 20; Test type: Superiority; p = 0.705, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -3.7, 95% CI 2-sided [-18.6 to 11.2] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 18: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Non-responders, Week 20; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -3.8, 95% CI 2-sided [-20.0 to 12.4] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 19: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 28; Test type: Superiority; p = 0.075, Chi-squared — [p-value comment as in outcome 27, analysis 11]; Risk Difference (RD) = 27.5, 95% CI 2-sided [-5.0 to 60.0] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 20: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 28; Test type: Superiority; p = 0.705, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -3.7, 95% CI 2-sided [-18.6 to 11.2] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 21: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Non-responders, Week 28; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 0.5, 95% CI 2-sided [-17.4 to 18.5] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 22: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 36; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 0.6, 95% CI 2-sided [-20.5 to 21.8] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 23: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 36; Test type: Superiority; p = 0.348, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -6.4, 95% CI 2-sided [-18.0 to 5.2] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 24: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Non-responders, Week 36; Test type: Superiority; p = 0.686, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 3.7, 95% CI 2-sided [-13.4 to 20.7] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 25: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 44; Test type: Superiority; p = 0.616, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 7.5, 95% CI 2-sided [-19.8 to 34.8] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 26: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 44; Test type: Superiority; p = 0.420, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -6.6, 95% CI 2-sided [-20.5 to 7.3] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 27: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Non-responders, Week 44; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -3.8, 95% CI 2-sided [-20.0 to 12.4] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 28: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 52; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 0.6, 95% CI 2-sided [-20.5 to 21.8] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 29: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 52; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -0.6, 95% CI 2-sided [-14.4 to 13.3] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 30: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Non-responders, Week 52; Test type: Superiority; p = 0.686, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 3.7, 95% CI 2-sided [-13.4 to 20.7] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 31: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 20; Test type: Superiority; p = 0.555, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 9.4, 95% CI 2-sided [-21.9 to 40.6] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 32: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 20; Test type: Superiority; p = 0.830, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -2.7, 95% CI 2-sided [-27.2 to 21.8] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 33: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical responders, Week 20; Test type: Superiority; p = 0.518, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -9.0, 95% CI 2-sided [-36.0 to 17.9] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 34: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 28; Test type: Superiority; p = 0.428, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 12.5, 95% CI 2-sided [-18.6 to 43.6] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 35: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 28; Test type: Superiority; p = 0.757, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 3.9, 95% CI 2-sided [-20.7 to 28.4] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 36: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical responders, Week 28; Test type: Superiority; p = 0.745, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 4.6, 95% CI 2-sided [-23.2 to 32.4] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 37: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 36; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -5.8, 95% CI 2-sided [-34.6 to 23.0] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 38: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 36; Test type: Superiority; p = 0.773, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 3.6, 95% CI 2-sided [-20.6 to 27.7] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 39: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical responders, Week 36; Test type: Superiority; p = 0.838, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -2.8, 95% CI 2-sided [-29.4 to 23.8] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 40: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 44; Test type: Superiority; p = 0.497, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -12.9, 95% CI 2-sided [-40.0 to 14.1] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 41: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 44; Test type: Superiority; p = 0.404, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 10.5, 95% CI 2-sided [-14.0 to 34.9] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 42: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical responders, Week 44; Test type: Superiority; p = 0.838, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -2.8, 95% CI 2-sided [-29.4 to 23.8] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 43: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 52; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 3.6, 95% CI 2-sided [-24.4 to 31.6] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 44: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 52; Test type: Superiority; p = 0.174, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 16.4, 95% CI 2-sided [-7.0 to 39.8] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 45: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical responders, Week 52; Test type: Superiority; p = 0.611, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 6.6, 95% CI 2-sided [-19.1 to 32.3] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 46: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 28; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -5.0, 95% CI 2-sided [-14.6 to 4.6] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 47: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 28; Test type: Superiority; p = 0.488, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -5.0, 95% CI 2-sided [-14.6 to 4.6] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 48: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 28; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -5.0, 95% CI 2-sided [-14.6 to 4.6] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 49: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 44; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -5.0, 95% CI 2-sided [-14.6 to 4.6] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 50: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 44; Test type: Superiority; p = 0.488, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -5.0, 95% CI 2-sided [-14.6 to 4.6] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 51: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 44; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -5.0, 95% CI 2-sided [-14.6 to 4.6] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 52: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 52; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -5.0, 95% CI 2-sided [-14.6 to 4.6] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 53: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 52; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -0.2, 95% CI 2-sided [-13.4 to 13.0] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 54: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 52; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -5.0, 95% CI 2-sided [-14.6 to 4.6] — [estimate comment as in outcome 25, analysis 1]

28. Secondary Outcome: Percentage of Participants Who Maintain Clinical Remission Over Time Among Participants in Clinical Remission at Week 16 in Participants Receiving Upadacitinib in Induction
Description: as for outcome 27
Time Frame: Week 20, Week 28, Week 36, Week 44, Week 52
Population: Includes intent-to-treat responder (ITT-R) and non-responder (ITT-NR) analysis sets: all re-randomized participants in the double-blind Extension Phase who were responders and nonresponders at Week 16 of the Induction Period, respectively, and in clinical remission at Week 16. Non responder imputation. Participants with an assessment at given time point.
Measure: Number; unit: percentage of participants
Arm/Group | Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction | Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction | Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction | Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction
Number analyzed (Participants) | 13 | 6 | 9 | 4
percentage of participants
  Responders, Week 20: number analyzed (Participants) | 10 | 3 | 7 | 3
  Responders, Week 20 | 80.0 | 66.7 | 71.4 | 100
  Responders, Week 28: number analyzed (Participants) | 10 | 3 | 7 | 3
  Responders, Week 28 | 90.0 | 66.7 | 57.1 | 100
  Responders, Week 36: number analyzed (Participants) | 10 | 3 | 7 | 3
  Responders, Week 36 | 80.0 | 100 | 71.4 | 66.7
  Responders, Week 44: number analyzed (Participants) | 10 | 3 | 7 | 3
  Responders, Week 44 | 80.0 | 33.3 | 71.4 | 66.7
  Responders, Week 52: number analyzed (Participants) | 10 | 3 | 7 | 3
  Responders, Week 52 | 60.0 | 66.7 | 71.4 | 66.7
  Non-responders, Week 20: number analyzed (Participants) | 3 | 3 | 2 | 1
  Non-responders, Week 20 | 66.7 | 100 | 50.0 | 100
  Non-responders, Week 28: number analyzed (Participants) | 3 | 3 | 2 | 1
  Non-responders, Week 28 | 66.7 | 100 | 50.0 | 100
  Non-responders, Week 36: number analyzed (Participants) | 3 | 3 | 2 | 1
  Non-responders, Week 36 | 66.7 | 33.3 | 50.0 | 100
  Non-responders, Week 44: number analyzed (Participants) | 3 | 3 | 2 | 1
  Non-responders, Week 44 | 66.7 | 66.7 | 50.0 | 100
  Non-responders, Week 52: number analyzed (Participants) | 3 | 3 | 2 | 1
  Non-responders, Week 52 | 33.3 | 33.3 | 0 | 100
  Clinical responders, Week 20 | 76.9 | 83.3 | 66.7 | 100
  Clinical responders, Week 28 | 84.6 | 83.3 | 55.6 | 100
  Clinical responders, Week 36 | 76.9 | 66.7 | 66.7 | 75.0
  Clinical responders, Week 44 | 76.9 | 50.0 | 66.7 | 75.0
  Clinical responders, Week 52 | 53.8 | 50.0 | 55.6 | 75.0
  Clinical non-responders, Week 20: number analyzed (Participants) | 0 | 0 | 0 | 0
  Clinical non-responders, Week 28: number analyzed (Participants) | 0 | 0 | 0 | 0
  Clinical non-responders, Week 36: number analyzed (Participants) | 0 | 0 | 0 | 0
  Clinical non-responders, Week 44: number analyzed (Participants) | 0 | 0 | 0 | 0
  Clinical non-responders, Week 52: number analyzed (Participants) | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 20; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -13.3, 95% CI 2-sided [-72.2 to 45.5] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 2: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 20; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -8.6, 95% CI 2-sided [-50.2 to 33.1] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 3: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Responders, Week 20; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 20.0, 95% CI 2-sided [-4.8 to 44.8] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 4: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 28; Test type: Superiority; p = 0.423, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -23.3, 95% CI 2-sided [-79.8 to 33.2] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 5: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 28; Test type: Superiority; p = 0.250, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -32.9, 95% CI 2-sided [-74.0 to 8.2] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 6: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Responders, Week 28; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 10.0, 95% CI 2-sided [-8.6 to 28.6] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 7: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 36; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 20.0, 95% CI 2-sided [-4.8 to 44.8] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 8: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 36; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -8.6, 95% CI 2-sided [-50.2 to 33.1] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 9: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Responders, Week 36; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -13.3, 95% CI 2-sided [-72.2 to 45.5] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 10: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 44; Test type: Superiority; p = 0.203, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -46.7, 95% CI 2-sided [-100.0 to 12.2] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 11: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 44; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -8.6, 95% CI 2-sided [-50.2 to 33.1] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 12: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Responders, Week 44; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -13.3, 95% CI 2-sided [-72.2 to 45.5] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 13: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 52; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 6.7, 95% CI 2-sided [-54.7 to 68.0] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 14: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 52; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 11.4, 95% CI 2-sided [-33.8 to 56.6] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 15: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Responders, Week 52; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 6.7, 95% CI 2-sided [-54.7 to 68.0] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 16: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 20; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 33.3, 95% CI 2-sided [-20.0 to 86.7] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 17: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 20; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -16.7, 95% CI 2-sided [-100.0 to 70.8] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 18: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Non-responders, Week 20; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 33.3, 95% CI 2-sided [-20.0 to 86.7] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 19: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 28; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 33.3, 95% CI 2-sided [-20.0 to 86.7] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 20: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 28; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -16.7, 95% CI 2-sided [-100.0 to 70.8] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 21: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Non-responders, Week 28; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 33.3, 95% CI 2-sided [-20.0 to 86.7] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 22: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 36; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -33.3, 95% CI 2-sided [-100.0 to 42.1] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 23: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 36; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -16.7, 95% CI 2-sided [-100.0 to 70.8] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 24: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Non-responders, Week 36; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 33.3, 95% CI 2-sided [-20.0 to 86.7] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 25: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 44; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 0.0, 95% CI 2-sided [-75.4 to 75.4] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 26: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 44; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -16.7, 95% CI 2-sided [-100.0 to 70.8] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 27: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Non-responders, Week 44; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 33.3, 95% CI 2-sided [-20.0 to 86.7] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 28: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 52; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 0.0, 95% CI 2-sided [-75.4 to 75.4] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 29: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 52; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -33.3, 95% CI 2-sided [-86.7 to 20.0] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 30: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Non-responders, Week 52; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 66.7, 95% CI 2-sided [13.3 to 100.0] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 31: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 20; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 6.4, 90% CI 2-sided [-31.2 to 44.0] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 32: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 20; Test type: Superiority; p = 0.655, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -10.3, 95% CI 2-sided [-48.6 to 28.1] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 33: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical responders, Week 20; Test type: Superiority; p = 0.541, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 23.1, 95% CI 2-sided [0.2 to 46.0] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 34: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 28; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -1.3, 95% CI 2-sided [-37.0 to 34.4] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 35: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 28; Test type: Superiority; p = 0.178, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -29.1, 95% CI 2-sided [-67.0 to 8.9] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 36: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical responders, Week 28; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 15.4, 95% CI 2-sided [-4.2 to 35.0] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 37: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 36; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -10.3, 95% CI 2-sided [-54.4 to 33.9] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 38: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 36; Test type: Superiority; p = 0.655, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -10.3, 95% CI 2-sided [-48.6 to 28.1] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 39: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical responders, Week 36; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -1.9, 95% CI 2-sided [-50.1 to 46.3] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 40: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 44; Test type: Superiority; p = 0.320, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -26.9, 95% CI 2-sided [-73.0 to 19.2] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 41: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 44; Test type: Superiority; p = 0.655, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -10.3, 95% CI 2-sided [-48.6 to 28.1] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 42: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical responders, Week 44; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -1.9, 95% CI 2-sided [-50.1 to 46.3] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 43: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 52; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -3.8, 95% CI 2-sided [-52.2 to 44.5] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 44: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 52; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 1.7, 95% CI 2-sided [-40.6 to 44.0] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 45: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical responders, Week 52; Test type: Superiority; p = 0.603, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 21.2, 95% CI 2-sided [-29.2 to 71.5] — [estimate comment as in outcome 25, analysis 1]

29. Secondary Outcome: Percentage of Participants Who Achieve Modified Clinical Remission Over Time During Extension Phase Among Participants With Daily Stool Frequency ≥ 4.0 or Daily Abdominal Pain ≥ 2.0 at Induction Baseline
Description: Modified clinical remission was defined as average daily stool frequency <= 2.8 and not worse than Induction Baseline and average daily abdominal pain <= 1.0 and not worse than Induction Baseline. The very soft/liquid stool frequency and abdominal pain scores at a visit were the average of the daily values reported during the 7 usable days preceding the scheduled assessment visit. Abdominal Pain was rated on a 4-point scale from 0 (none) to 3 (severe).
Time Frame: Week 20, Week 28, Week 36, Week 44, Week 52
Population: Includes intent-to-treat responder (ITT-R) and non-responder (ITT-NR) analysis sets: all re-randomized participants in the double-blind Extension Phase who were responders and nonresponders at Week 16 of the Induction Period, respectively, and with daily stool frequency >= 4.0 or daily abdominal pain >= 2.0 at Induction Baseline. Non responder imputation. Participants with an assessment at given time point.
Measure: Number; unit: percentage of participants
Groups:
- Upadacitinib 24 mg QD in Extension/ Placebo in Induction: Upadacitinib 24 mg QD (consisting of two 12 mg IR doses) during the 36-week double-blind Extension Phase. Placebo in Induction Phase.
Arm/Group | Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction | Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction | Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction | Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction | Upadacitinib 3 mg BID in Extension/ Placebo in Induction | Upadacitinib 6 mg BID in Extension/ Placebo in Induction | Upadacitinib 12 mg BID in Extension/ Placebo in Induction | Upadacitinib 24 mg QD in Extension/ Placebo in Induction
Number analyzed (Participants) | 45 | 17 | 48 | 30 | 8 | 5 | 8 | 4
percentage of participants
  Responders, Week 20: number analyzed (Participants) | 17 | 8 | 15 | 10 | 1 | 0 | 0 | 0
  Responders, Week 20 | 47.1 | 62.5 | 66.7 | 60.0 | 0 |  |  |
  Responders, Week 28: number analyzed (Participants) | 17 | 8 | 15 | 10 | 1 | 0 | 0 | 0
  Responders, Week 28 | 70.6 | 50.0 | 66.7 | 60.0 | 0 |  |  |
  Responders, Week 36: number analyzed (Participants) | 17 | 8 | 15 | 10 | 1 | 0 | 0 | 0
  Responders, Week 36 | 58.8 | 87.5 | 73.3 | 30.0 | 0 |  |  |
  Responders, Week 44: number analyzed (Participants) | 17 | 8 | 15 | 10 | 1 | 0 | 0 | 0
  Responders, Week 44 | 47.1 | 37.5 | 73.3 | 40.0 | 0 |  |  |
  Responders, Week 52: number analyzed (Participants) | 17 | 8 | 15 | 10 | 1 | 0 | 0 | 0
  Responders, Week 52 | 41.2 | 62.5 | 73.3 | 40.0 | 0 |  |  |
  Non-responders, Week 20: number analyzed (Participants) | 28 | 9 | 33 | 20 | 7 | 5 | 8 | 4
  Non-responders, Week 20 | 17.9 | 44.4 | 12.1 | 10.0 | 42.9 | 20.0 | 25.0 | 25.0
  Non-responders, Week 28: number analyzed (Participants) | 28 | 9 | 33 | 20 | 7 | 5 | 8 | 4
  Non-responders, Week 28 | 21.4 | 44.4 | 9.1 | 15.0 | 42.9 | 20.0 | 25.0 | 50.0
  Non-responders, Week 36: number analyzed (Participants) | 28 | 9 | 33 | 20 | 7 | 5 | 8 | 4
  Non-responders, Week 36 | 14.3 | 11.1 | 6.1 | 15.0 | 57.1 | 20.0 | 25.0 | 25.0
  Non-responders, Week 44: number analyzed (Participants) | 28 | 9 | 33 | 20 | 7 | 5 | 8 | 4
  Non-responders, Week 44 | 14.3 | 22.2 | 6.1 | 10.0 | 42.9 | 20.0 | 37.5 | 25.0
  Non-responders, Week 52: number analyzed (Participants) | 28 | 9 | 33 | 20 | 7 | 5 | 8 | 4
  Non-responders, Week 52 | 7.1 | 11.1 | 12.1 | 15.0 | 28.6 | 0 | 37.5 | 50.0
  Clinical responders, Week 20: number analyzed (Participants) | 28 | 14 | 27 | 18 | 5 | 1 | 3 | 1
  Clinical responders, Week 20 | 42.9 | 64.3 | 51.9 | 44.4 | 60.0 | 100 | 33.3 | 100
  Clinical responders, Week 28: number analyzed (Participants) | 28 | 14 | 27 | 18 | 5 | 1 | 3 | 1
  Clinical responders, Week 28 | 57.1 | 57.1 | 48.1 | 50.0 | 60.0 | 100 | 33.3 | 100
  Clinical responders, Week 36: number analyzed (Participants) | 28 | 14 | 27 | 18 | 5 | 1 | 3 | 1
  Clinical responders, Week 36 | 46.4 | 57.1 | 48.1 | 33.3 | 80.0 | 100 | 33.3 | 100
  Clinical responders, Week 44: number analyzed (Participants) | 28 | 14 | 27 | 18 | 5 | 1 | 3 | 1
  Clinical responders, Week 44 | 39.3 | 35.7 | 48.1 | 33.3 | 60.0 | 100 | 33.3 | 100
  Clinical responders, Week 52: number analyzed (Participants) | 28 | 14 | 27 | 18 | 5 | 1 | 3 | 1
  Clinical responders, Week 52 | 28.6 | 42.9 | 51.9 | 38.9 | 40.0 | 0 | 33.3 | 100
  Clinical non-responders, Week 20: number analyzed (Participants) | 17 | 3 | 21 | 12 | 3 | 4 | 5 | 3
  Clinical non-responders, Week 20 | 5.9 | 0 | 0 | 0 | 0 | 0 | 20.0 | 0
  Clinical non-responders, Week 28: number analyzed (Participants) | 17 | 3 | 21 | 12 | 3 | 4 | 5 | 3
  Clinical non-responders, Week 28 | 11.8 | 0 | 0 | 0 | 0 | 0 | 20.0 | 33.3
  Clinical non-responders, Week 36: number analyzed (Participants) | 17 | 3 | 21 | 12 | 3 | 4 | 5 | 3
  Clinical non-responders, Week 36 | 5.9 | 0 | 0 | 0 | 0 | 0 | 20.0 | 0
  Clinical non-responders, Week 44: number analyzed (Participants) | 17 | 3 | 21 | 12 | 3 | 4 | 5 | 3
  Clinical non-responders, Week 44 | 5.9 | 0 | 0 | 0 | 0 | 0 | 40.0 | 0
  Clinical non-responders, Week 52: number analyzed (Participants) | 17 | 3 | 21 | 12 | 3 | 4 | 5 | 3
  Clinical non-responders, Week 52 | 5.9 | 0 | 4.8 | 0 | 0 | 0 | 40.0 | 33.3
Statistical Analysis 1: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 20; Test type: Superiority; p = 0.673, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 15.4, 95% CI 2-sided [-25.6 to 56.5] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 2: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 20; Test type: Superiority; p = 0.265, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 19.6, 95% CI 2-sided [-14.0 to 53.3] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 3: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Responders, Week 20; Test type: Superiority; p = 0.695, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 12.9, 95% CI 2-sided [-25.6 to 51.5] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 4: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 28; Test type: Superiority; p = 0.394, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -20.6, 95% CI 2-sided [-61.4 to 20.3] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 5: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 28; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -3.9, 95% CI 2-sided [-36.1 to 28.3] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 6: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Responders, Week 28; Test type: Superiority; p = 0.683, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -10.6, 95% CI 2-sided [-47.9 to 26.7] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 7: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 36; Test type: Superiority; p = 0.205, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 28.7, 95% CI 2-sided [-4.1 to 61.4] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 8: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 36; Test type: Superiority; p = 0.388, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 14.5, 95% CI 2-sided [-17.9 to 46.9] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 9: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Responders, Week 36; Test type: Superiority; p = 0.236, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -28.8, 95% CI 2-sided [-65.6 to 8.0] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 10: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 44; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -9.6, 95% CI 2-sided [-50.6 to 31.5] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 11: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 44; Test type: Superiority; p = 0.131, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 26.3, 95% CI 2-sided [-6.3 to 58.9] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 12: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Responders, Week 44; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -7.1, 95% CI 2-sided [-45.6 to 31.5] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 13: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 52; Test type: Superiority; p = 0.411, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 21.3, 95% CI 2-sided [-19.6 to 62.2] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 14: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 52; Test type: Superiority; p = 0.067, Chi-squared — [p-value comment as in outcome 27, analysis 11]; Risk Difference (RD) = 32.2, 95% CI 2-sided [-0.2 to 64.5] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 15: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Responders, Week 52; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -1.2, 95% CI 2-sided [-39.5 to 37.2] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 16: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 20; Test type: Superiority; p = 0.178, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 26.6, 95% CI 2-sided [-8.8 to 62.0] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 17: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 20; Test type: Superiority; p = 0.720, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -5.7, 95% CI 2-sided [-23.8 to 12.3] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 18: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Non-responders, Week 20; Test type: Superiority; p = 0.683, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -7.9, 95% CI 2-sided [-27.2 to 11.5] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 19: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 28; Test type: Superiority; p = 0.215, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 23.0, 95% CI 2-sided [-12.8 to 58.9] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 20: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 28; Test type: Superiority; p = 0.279, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -12.3, 95% CI 2-sided [-30.4 to 5.8] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 21: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Non-responders, Week 28; Test type: Superiority; p = 0.716, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -6.4, 95% CI 2-sided [-28.2 to 15.4] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 22: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 36; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -3.2, 95% CI 2-sided [-27.5 to 21.1] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 23: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 36; Test type: Superiority; p = 0.400, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -8.2, 95% CI 2-sided [-23.5 to 7.1] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 24: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Non-responders, Week 36; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 0.7, 95% CI 2-sided [-19.6 to 21.0] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 25: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 44; Test type: Superiority; p = 0.620, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 7.9, 95% CI 2-sided [-22.2 to 38.0] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 26: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 44; Test type: Superiority; p = 0.400, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -8.2, 95% CI 2-sided [-23.5 to 7.1] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 27: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Non-responders, Week 44; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -4.3, 95% CI 2-sided [-22.7 to 14.2] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 28: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 52; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 4.0, 95% CI 2-sided [-18.7 to 26.6] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 29: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 52; Test type: Superiority; p = 0.678, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 5.0, 95% CI 2-sided [-9.7 to 19.6] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 30: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Non-responders, Week 52; Test type: Superiority; p = 0.636, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 7.9, 95% CI 2-sided [-10.5 to 26.2] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 31: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 20; Test type: Superiority; p = 0.190, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 21.4, 95% CI 2-sided [-9.7 to 52.5] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 32: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 20; Test type: Superiority; p = 0.504, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 9.0, 95% CI 2-sided [-17.3 to 35.3] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 33: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical responders, Week 20; Test type: Superiority; p = 0.916, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 1.6, 95% CI 2-sided [-27.8 to 31.0] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 34: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 28; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 0.0, 95% CI 2-sided [-31.7 to 31.7] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 35: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 28; Test type: Superiority; p = 0.504, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -9.0, 95% CI 2-sided [-35.3 to 17.3] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 36: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical responders, Week 28; Test type: Superiority; p = 0.635, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -7.1, 95% CI 2-sided [-36.6 to 22.3] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 37: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 36; Test type: Superiority; p = 0.513, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 10.7, 95% CI 2-sided [-21.1 to 42.5] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 38: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 36; Test type: Superiority; p = 0.898, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 1.7, 95% CI 2-sided [-24.7 to 28.1] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 39: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical responders, Week 36; Test type: Superiority; p = 0.379, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -13.1, 95% CI 2-sided [-41.7 to 15.5] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 40: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 44; Test type: Superiority; p = 0.822, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -3.6, 95% CI 2-sided [-34.5 to 27.4] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 41: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 44; Test type: Superiority; p = 0.508, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 8.9, 95% CI 2-sided [-17.3 to 35.0] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 42: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical responders, Week 44; Test type: Superiority; p = 0.683, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -6.0, 95% CI 2-sided [-34.3 to 22.4] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 43: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 52; Test type: Superiority; p = 0.490, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 14.3, 95% CI 2-sided [-16.6 to 45.1] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 44: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 52; Test type: Superiority; p = 0.078, Chi-squared — [p-value comment as in outcome 27, analysis 11]; Risk Difference (RD) = 23.3, 95% CI 2-sided [-1.9 to 48.5] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 45: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical responders, Week 52; Test type: Superiority; p = 0.466, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 10.3, 95% CI 2-sided [-17.7 to 38.4] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 46: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 20; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -5.9, 95% CI 2-sided [-17.1 to 5.3] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 47: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 20; Test type: Superiority; p = 0.447, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -5.9, 95% CI 2-sided [-17.1 to 5.3] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 48: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 20; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -5.9, 95% CI 2-sided [-17.1 to 5.3] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 49: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 28; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -11.8, 95% CI 2-sided [-27.1 to 3.6] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 50: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 28; Test type: Superiority; p = 0.193, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -11.8, 95% CI 2-sided [-27.1 to 3.6] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 51: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 28; Test type: Superiority; p = 0.498, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -11.8, 95% CI 2-sided [-27.1 to 3.6] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 52: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 36; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -5.9, 95% CI 2-sided [-17.1 to 5.3] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 53: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 36; Test type: Superiority; p = 0.447, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -5.9, 95% CI 2-sided [-17.1 to 5.3] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 54: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 36; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -5.9, 95% CI 2-sided [-17.1 to 5.3] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 55: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 44; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -5.9, 95% CI 2-sided [-17.1 to 5.3] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 56: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 44; Test type: Superiority; p = 0.447, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -5.9, 95% CI 2-sided [-17.1 to 5.3] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 57: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 44; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -5.9, 95% CI 2-sided [-17.1 to 5.3] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 58: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 52; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -5.9, 95% CI 2-sided [-17.1 to 5.3] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 59: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 52; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -1.1, 95% CI 2-sided [-15.5 to 13.3] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 60: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 52; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -5.9, 95% CI 2-sided [-17.1 to 5.3] — [estimate comment as in outcome 25, analysis 1]

30. Secondary Outcome: Percentage of Participants Who Achieve Modified Clinical Remission Over Time During Extension Phase Among Participants In Modified Clinical Remission At Week 16 and Daily Stool Frequency ≥ 4.0 or Daily Abdominal Pain ≥ 2.0 at Induction Baseline
Description: as for outcome 29
Time Frame: Week 20, Week 28, Week 36, Week 44, Week 52
Population: Includes intent-to-treat responder (ITT-R) and non-responder (ITT-NR) analysis sets: all re-randomized participants in the double-blind Extension Phase who were responders and nonresponders at Week 16 of the Induction Period, respectively, and with modified clinical remission at Week 16 and daily stool frequency >= 4.0 or daily abdominal pain >= 2.0 at Induction Baseline. Non responder imputation. Participants with an assessment at given time point.
Measure: Number; unit: percentage of participants
Arm/Group | Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction | Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction | Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction | Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction | Upadacitinib 3 mg BID in Extension/ Placebo in Induction | Upadacitinib 6 mg BID in Extension/ Placebo in Induction | Upadacitinib 12 mg BID in Extension/ Placebo in Induction | Upadacitinib 24 mg QD in Extension/ Placebo in Induction
Number analyzed (Participants) | 15 | 10 | 12 | 5 | 2 | 0 | 1 | 1
percentage of participants
  Responders, Week 20: number analyzed (Participants) | 12 | 5 | 10 | 4 | 0 | 0 | 0 | 0
  Responders, Week 20 | 66.7 | 60.0 | 90.0 | 100 |  |  |  |
  Responders, Week 28: number analyzed (Participants) | 12 | 5 | 10 | 4 | 0 | 0 | 0 | 0
  Responders, Week 28 | 91.7 | 60.0 | 90.0 | 100 |  |  |  |
  Responders, Week 36: number analyzed (Participants) | 12 | 5 | 10 | 4 | 0 | 0 | 0 | 0
  Responders, Week 36 | 66.7 | 100 | 90.0 | 75.0 |  |  |  |
  Responders, Week 44: number analyzed (Participants) | 12 | 5 | 10 | 4 | 0 | 0 | 0 | 0
  Responders, Week 44 | 66.7 | 40.0 | 90.0 | 75.0 |  |  |  |
  Responders, Week 52: number analyzed (Participants) | 12 | 5 | 10 | 4 | 0 | 0 | 0 | 0
  Responders, Week 52 | 58.3 | 80.0 | 90.0 | 75.0 |  |  |  |
  Non-responders, Week 20: number analyzed (Participants) | 3 | 5 | 2 | 1 | 2 | 0 | 1 | 1
  Non-responders, Week 20 | 66.7 | 80.0 | 50.0 | 100 | 100 |  | 100 | 100
  Non-responders, Week 28: number analyzed (Participants) | 3 | 5 | 2 | 1 | 2 | 0 | 1 | 1
  Non-responders, Week 28 | 100 | 60.0 | 50.0 | 100 | 100 |  | 100 | 100
  Non-responders, Week 36: number analyzed (Participants) | 3 | 5 | 2 | 1 | 2 | 0 | 1 | 1
  Non-responders, Week 36 | 66.7 | 20.0 | 50.0 | 100 | 100 |  | 100 | 100
  Non-responders, Week 44: number analyzed (Participants) | 3 | 5 | 2 | 1 | 2 | 0 | 1 | 1
  Non-responders, Week 44 | 66.7 | 40.0 | 50.0 | 100 | 50.0 |  | 100 | 100
  Non-responders, Week 52: number analyzed (Participants) | 3 | 5 | 2 | 1 | 2 | 0 | 1 | 1
  Non-responders, Week 52 | 33.3 | 20.0 | 50.0 | 100 | 50.0 |  | 100 | 100
  Clinical responders, Week 20 | 66.7 | 70.0 | 83.3 | 100 | 100 |  | 100 | 100
  Clinical responders, Week 28 | 93.3 | 60.0 | 83.3 | 100 | 100 |  | 100 | 100
  Clinical responders, Week 36 | 66.7 | 60.0 | 83.3 | 80.0 | 100 |  | 100 | 100
  Clinical responders, Week 44 | 66.7 | 40.0 | 83.3 | 80.0 | 50.0 |  | 100 | 100
  Clinical responders, Week 52 | 53.3 | 50.0 | 83.3 | 80.0 | 50.0 |  | 100 | 100
  Clinical non- responders, Week 20: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Clinical non- responders, Week 28: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Clinical non- responders, Week 36: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Clinical non- responders, Week 44: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Clinical non- responders, Week 52: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 20; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -6.7, 95% CI 2-sided [-57.2 to 43.9] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 2: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 20; Test type: Superiority; p = 0.323, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 23.3, 95% CI 2-sided [-9.2 to 55.8] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 3: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Responders, Week 20; Test type: Superiority; p = 0.516, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 33.3, 95% CI 2-sided [6.7 to 60.0] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 4: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 28; Test type: Superiority; p = 0.191, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -31.7, 95% CI 2-sided [-77.4 to 14.0] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 5: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 28; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -1.7, 95% CI 2-sided [-26.0 to 22.6] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 6: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Responders, Week 28; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 8.3, 95% CI 2-sided [-7.3 to 24.0] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 7: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 36; Test type: Superiority; p = 0.261, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 33.3, 95% CI 2-sided [6.7 to 60.0] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 8: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 36; Test type: Superiority; p = 0.323, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 23.3, 95% CI 2-sided [-9.2 to 55.8] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 9: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Responders, Week 36; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 8.3, 95% CI 2-sided [-41.8 to 58.5] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 10: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 44; Test type: Superiority; p = 0.593, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -26.7, 95% CI 2-sided [-77.2 to 23.9] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 11: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 44; Test type: Superiority; p = 0.323, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 23.3, 95% CI 2-sided [-9.2 to 55.8] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 12: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Responders, Week 44; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 8.3, 95% CI 2-sided [-41.8 to 58.5] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 13: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 52; Test type: Superiority; p = 0.600, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 21.7, 95% CI 2-sided [-23.1 to 66.5] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 14: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 52; Test type: Superiority; p = 0.162, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 31.7, 95% CI 2-sided [-1.9 to 65.2] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 15: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Responders, Week 52; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 16.7, 95% CI 2-sided [-34.1 to 67.4] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 16: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 20; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 13.3, 95% CI 2-sided [-50.5 to 77.2] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 17: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 20; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -16.7, 95% CI 2-sided [-100.0 to 70.8] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 18: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Non-responders, Week 20; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 33.3, 95% CI 2-sided [-20.0 to 86.7] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 19: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 28; Test type: Superiority; p = 0.464, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -40.0, 95% CI 2-sided [-82.9 to 2.9] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 20: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 28; Test type: Superiority; p = 0.400, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -50.0, 95% CI 2-sided [-100.0 to 19.3] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 21: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 36; Test type: Superiority; p = 0.464, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -46.7, 95% CI 2-sided [-100.0 to 17.2] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 22: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 36; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -16.7, 95% CI 2-sided [-100.0 to 70.8] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 23: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Non-responders, Week 36; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 33.3, 95% CI 2-sided [-20.0 to 86.7] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 24: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 44; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -26.7, 95% CI 2-sided [-95.1 to 41.8] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 25: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 44; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -16.7, 95% CI 2-sided [-100.0 to 70.8] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 26: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Non-responders, Week 44; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 33.3, 95% CI 2-sided [-20.0 to 86.7] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 27: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 52; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -13.3, 95% CI 2-sided [-77.2 to 50.5] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 28: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 52; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 16.7, 95% CI 2-sided [-70.8 to 100.0] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 29: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Non-responders, Week 52; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 66.7, 95% CI 2-sided [13.3 to 100.0] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 30: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 20; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 3.3, 95% CI 2-sided [-33.8 to 40.4] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 31: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 20; Test type: Superiority; p = 0.408, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 16.7, 95% CI 2-sided [-15.2 to 48.5] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 32: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical responders, Week 20; Test type: Superiority; p = 0.266, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 33.3, 95% CI 2-sided [9.5 to 57.2] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 33: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 28; Test type: Superiority; p = 0.121, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -33.3, 95% CI 2-sided [-66.2 to -0.5] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 34: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 28; Test type: Superiority; p = -10.0, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -10.0, 95% CI 2-sided [-34.6 to 14.6] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 35: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical responders, Week 28; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 6.7, 95% CI 2-sided [-6.0 to 19.3] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 36: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 36; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -6.7, 95% CI 2-sided [-45.3 to 31.9] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 37: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 36; Test type: Superiority; p = 0.408, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 16.7, 95% CI 2-sided [-15.2 to 48.5] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 38: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical responders, Week 36; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 13.3, 95% CI 2-sided [-29.1 to 55.7] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 39: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 44; Test type: Superiority; p = 0.241, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -26.7, 95% CI 2-sided [-65.3 to 11.9] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 40: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 44; Test type: Superiority; p = 0.408, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 16.7, 95% CI 2-sided [-15.2 to 48.5] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 41: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical responders, Week 44; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 13.3, 95% CI 2-sided [-29.1 to 55.7] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 42: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 52; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -3.3, 95% CI 2-sided [-43.3 to 36.6] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 43: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 52; Test type: Superiority; p = 0.217, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 30.0, 95% CI 2-sided [-2.9 to 62.9] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 44: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical responders, Week 52; Test type: Superiority; p = 0.603, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 26.7, 95% CI 2-sided [-16.5 to 69.9] — [estimate comment as in outcome 25, analysis 1]

31. Secondary Outcome: Percentage of Participants Who Achieve Response at Week 52
Description: Response at Week 52 was defined as both endoscopic response at Week 52 and clinical response at Week 52. Endoscopic response: SES-CD at least 25% reduction from Baseline. Clinical response: average daily stool frequency at least 30% reduction from Induction Baseline and average daily abdominal pain not worse than Induction Baseline OR average daily abdominal pain at least 30% reduction from Induction Baseline and average daily stool frequency not worse than Induction Baseline.
  The very soft/liquid stool frequency and abdominal pain scores at a visit were the average of the daily values reported during the 7 usable days preceding the scheduled assessment visit. Abdominal Pain was rated on a 4-point scale from 0 (none) to 3 (severe). Details of the SES-CD scale are provided in the description of the first primary endpoint.
Time Frame: Week 52
Population: Includes intent-to-treat responder (ITT-R) and non-responder (ITT-NR) analysis sets: all re-randomized participants in the double-blind Extension Phase who were responders and nonresponders at Week 16 of the Induction Period, respectively. Non-responder imputation.
Measure: Number; unit: percentage of participants
Arm/Group | Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction | Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction | Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction | Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction | Upadacitinib 3 mg BID in Extension/ Placebo in Induction | Upadacitinib 6 mg BID in Extension/ Placebo in Induction | Upadacitinib 12 mg BID in Extension/ Placebo in Induction | Upadacitinib 24 mg QD in Extension/ Placebo in Induction
Number analyzed (Participants) | 52 | 18 | 50 | 33 | 9 | 5 | 9 | 4
percentage of participants
  Responders: number analyzed (Participants) | 20 | 8 | 16 | 10 | 1 | 0 | 0 | 0
  Responders | 50.0 | 62.5 | 68.8 | 40.0 | 100 |  |  |
  Non-responders: number analyzed (Participants) | 32 | 10 | 34 | 23 | 8 | 5 | 9 | 4
  Non-responders | 6.3 | 10.0 | 14.7 | 13.0 | 0 | 20.0 | 22.2 | 25.0
  Clinical responders: number analyzed (Participants) | 32 | 14 | 29 | 19 | 6 | 1 | 4 | 1
  Clinical responders | 34.4 | 42.9 | 51.7 | 36.8 | 16.7 | 0 | 0 | 100
  Clinical non-responders: number analyzed (Participants) | 20 | 4 | 21 | 14 | 3 | 4 | 5 | 3
  Clinical non-responders | 5.0 | 0 | 4.8 | 0 | 0 | 25.0 | 40.0 | 0
Statistical Analysis 1: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Responders; Test type: Superiority; p = 0.686, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 12.5, 95% CI 2-sided [-27.6 to 52.6] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 2: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Responders; Test type: Superiority; p = 0.257, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 18.8, 95% CI 2-sided [-12.8 to 50.3] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 3: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Responders; Test type: Superiority; p = 0.709, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -10.0, 95% CI 2-sided [-47.4 to 27.4] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 4: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Non-responders; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 3.7, 95% CI 2-sided [-16.6 to 24.1] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 5: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Non-responders; Test type: Superiority; p = 0.428, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 8.5, 95% CI 2-sided [-6.1 to 23.0] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 6: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Non-responders; Test type: Superiority; p = 0.639, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 6.8, 95% CI 2-sided [-9.3 to 22.9] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 7: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical responders; Test type: Superiority; p = 0.583, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 8.5, 95% CI 2-sided [-22.2 to 39.2] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 8: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical responders; Test type: Superiority; p = 0.171, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 17.3, 95% CI 2-sided [-7.2 to 41.9] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 9: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical responders; Test type: Superiority; p = 0.859, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 2.5, 95% CI 2-sided [-24.8 to 29.7] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 10: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical non-responders; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -5.0, 95% CI 2-sided [-14.6 to 4.6] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 11: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical non-responders; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -0.2, 95% CI 2-sided [-13.4 to 13.0] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 12: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical non-responders; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -5.0, 95% CI 2-sided [-14.6 to 4.6] — [estimate comment as in outcome 25, analysis 1]

32. Secondary Outcome: Percentage of Participants With SES-CD ≤ 2 at Week 52
Description: SES-CD subscores assess the following: presence and size of ulcers in 5 visualized bowel segments; extent of ulcerated surface in 5 visualized bowel segments; extent of affected surface in 5 visualized bowel segments; presence and type of narrowings in 5 visualized bowel segments. Subscores range from 0 to 15, and are summed for a total SES-CD score ranging from 0 to 56; higher scores indicate greater severity of mucosal inflammation.
Time Frame: Week 52
Population: as for outcome 31
Measure: Number; unit: percentage of participants
Arm/Group | Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction | Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction | Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction | Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction | Upadacitinib 3 mg BID in Extension/ Placebo in Induction | Upadacitinib 6 mg BID in Extension/ Placebo in Induction | Upadacitinib 12 mg BID in Extension/ Placebo in Induction | Upadacitinib 24 mg QD in Extension/ Placebo in Induction
Number analyzed (Participants) | 52 | 18 | 50 | 33 | 9 | 5 | 9 | 4
percentage of participants
  Responders: number analyzed (Participants) | 20 | 8 | 16 | 10 | 1 | 0 | 0 | 0
  Responders | 10.0 | 12.5 | 31.3 | 0 | 0 |  |  |
  Non-responders: number analyzed (Participants) | 32 | 10 | 34 | 23 | 8 | 5 | 9 | 4
  Non-responders | 6.3 | 0 | 8.8 | 8.7 | 0 | 0 | 0 | 25.0
  Clinical responders: number analyzed (Participants) | 32 | 14 | 29 | 19 | 6 | 1 | 4 | 1
  Clinical responders | 6.3 | 7.1 | 20.7 | 10.5 | 0 | 0 | 0 | 100
  Clinical non-responders: number analyzed (Participants) | 20 | 4 | 21 | 14 | 3 | 4 | 5 | 3
  Clinical non-responders | 10.0 | 0 | 9.5 | 0 | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Responders; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 2.5, 95% CI 2-sided [-23.9 to 28.9] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 2: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Responders; Test type: Superiority; p = 0.204, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 21.3, 95% CI 2-sided [-5.0 to 47.5] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 3: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Responders; Test type: Superiority; p = 0.540, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -10.0, 95% CI 2-sided [-23.1 to 3.1] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 4: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Non-responders; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -6.3, 95% CI 2-sided [-14.6 to 2.1] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 5: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Non-responders; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 2.6, 95% CI 2-sided [-10.1 to 15.3] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 6: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Non-responders; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 2.4, 95% CI 2-sided [-11.8 to 16.7] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 7: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical responders; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 0.9, 95% CI 2-sided [-15.0 to 16.8] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 8: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical responders; Test type: Superiority; p = 0.135, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 14.4, 95% CI 2-sided [-2.5 to 31.4] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 9: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical responders; Test type: Superiority; p = 0.623, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 4.3, 95% CI 2-sided [-11.9 to 20.4] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 10: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical non-responders; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -10.0, 95% CI 2-sided [-23.1 to 3.1] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 11: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical non-responders; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -0.5, 95% CI 2-sided [-18.7 to 17.7] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 12: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical non-responders; Test type: Superiority; p = 0.501, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -10.0, 95% CI 2-sided [-23.1 to 3.1] — [estimate comment as in outcome 25, analysis 1]

33. Secondary Outcome: Percentage of Participants With SES-CD = 0 at Week 52
Description: as for outcome 32
Time Frame: Week 52
Population: as for outcome 31
Measure: Number; unit: percentage of participants
Arm/Group | Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction | Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction | Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction | Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction | Upadacitinib 3 mg BID in Extension/ Placebo in Induction | Upadacitinib 6 mg BID in Extension/ Placebo in Induction | Upadacitinib 12 mg BID in Extension/ Placebo in Induction | Upadacitinib 24 mg QD in Extension/ Placebo in Induction
Number analyzed (Participants) | 52 | 18 | 50 | 33 | 9 | 5 | 9 | 4
percentage of participants
  Responders: number analyzed (Participants) | 20 | 8 | 16 | 10 | 1 | 0 | 0 | 0
  Responders | 10.0 | 12.5 | 31.3 | 0 | 0 |  |  |
  Non-responders: number analyzed (Participants) | 32 | 10 | 34 | 23 | 8 | 5 | 9 | 4
  Non-responders | 3.1 | 0 | 8.8 | 4.3 | 0 | 0 | 0 | 0
  Clinical responders: number analyzed (Participants) | 32 | 14 | 29 | 19 | 6 | 1 | 4 | 1
  Clinical responders | 6.3 | 7.1 | 20.7 | 5.3 | 0 | 0 | 0 | 0
  Clinical non-responders: number analyzed (Participants) | 20 | 4 | 21 | 14 | 3 | 4 | 5 | 3
  Clinical non-responders | 5.0 | 0 | 9.5 | 0 | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Responders; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 2.5, 95% CI 2-sided [-23.9 to 28.9] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 2: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Responders; Test type: Superiority; p = 0.204, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 21.3, 95% CI 2-sided [-5.0 to 47.5] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 3: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Responders; Test type: Superiority; p = 0.540, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -10.0, 95% CI 2-sided [-23.1 to 3.1] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 4: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Non-responders; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -3.1, 95% CI 2-sided [-9.2 to 2.9] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 5: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Non-responders; Test type: Superiority; p = 0.614, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 5.7, 95% CI 2-sided [-5.6 to 17.0] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 6: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Non-responders; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 1.2, 95% CI 2-sided [-9.1 to 11.5] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 7: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical responders; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 0.9, 95% CI 2-sided [-15.0 to 16.8] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 8: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical responders; Test type: Superiority; p = 0.135, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 14.4, 95% CI 2-sided [-2.5 to 31.4] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 9: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical responders; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -1.0, 95% CI 2-sided [-14.1 to 12.1] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 10: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical non-responders; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -5.0, 95% CI 2-sided [-14.6 to 4.6] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 11: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical non-responders; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 4.5, 95% CI 2-sided [-11.3 to 20.3] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 12: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical non-responders; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -5.0, 95% CI 2-sided [-14.6 to 4.6] — [estimate comment as in outcome 25, analysis 1]

34. Secondary Outcome: Percentage of Participants Who Achieve Endoscopic Response at Week 52
Description: Endoscopic response was defined as SES-CD at least 25% reduction from Induction Baseline. SES-CD subscores assess the following: presence and size of ulcers in 5 visualized bowel segments; extent of ulcerated surface in 5 visualized bowel segments; extent of affected surface in 5 visualized bowel segments; presence and type of narrowings in 5 visualized bowel segments. Subscores range from 0 to 15, and are summed for a total SES-CD score ranging from 0 to 56; higher scores indicate greater severity of mucosal inflammation.
Time Frame: Week 52
Population: as for outcome 31
Measure: Number; unit: percentage of participants
Arm/Group | Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction | Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction | Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction | Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction | Upadacitinib 3 mg BID in Extension/ Placebo in Induction | Upadacitinib 6 mg BID in Extension/ Placebo in Induction | Upadacitinib 12 mg BID in Extension/ Placebo in Induction | Upadacitinib 24 mg QD in Extension/ Placebo in Induction
Number analyzed (Participants) | 52 | 18 | 50 | 33 | 9 | 5 | 9 | 4
percentage of participants
  Responders: number analyzed (Participants) | 20 | 8 | 16 | 10 | 1 | 0 | 0 | 0
  Responders | 60.0 | 75.0 | 75.0 | 40.0 | 100 |  |  |
  Non-responders: number analyzed (Participants) | 32 | 10 | 34 | 23 | 8 | 5 | 9 | 4
  Non-responders | 15.6 | 20.0 | 20.6 | 17.4 | 0 | 20.0 | 22.2 | 25.0
  Clinical responders: number analyzed (Participants) | 32 | 14 | 29 | 19 | 6 | 1 | 4 | 1
  Clinical responders | 40.6 | 57.1 | 55.2 | 42.1 | 16.7 | 0 | 0 | 100
  Clinical non-responders: number analyzed (Participants) | 20 | 4 | 21 | 14 | 3 | 4 | 5 | 3
  Clinical non-responders | 20.0 | 0 | 14.3 | 0 | 0 | 25.0 | 40.0 | 0
Statistical Analysis 1: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Responders; Test type: Superiority; p = 0.669, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 15.0, 95% CI 2-sided [-21.9 to 51.9] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 2: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Responders; Test type: Superiority; p = 0.343, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 15.0, 95% CI 2-sided [-15.2 to 45.2] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 3: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Responders; Test type: Superiority; p = 0.442, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -20.0, 95% CI 2-sided [-57.2 to 17.2] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 4: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Non-responders; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 4.4, 95% CI 2-sided [-23.4 to 32.2] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 5: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Non-responders; Test type: Superiority; p = 0.601, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 5.0, 95% CI 2-sided [-13.6 to 23.5] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 6: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Non-responders; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 1.8, 95% CI 2-sided [-18.2 to 21.7] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 7: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical responders; Test type: Superiority; p = 0.301, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 16.5, 95% CI 2-sided [-14.5 to 47.5] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 8: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical responders; Test type: Superiority; p = 0.256, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 14.5, 95% CI 2-sided [-10.3 to 39.4] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 9: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical responders; Test type: Superiority; p = 0.917, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 1.5, 95% CI 2-sided [-26.5 to 29.5] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 10: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical non-responders; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -20.2, 95% CI 2-sided [-37.5 to -2.5] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 11: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical non-responders; Test type: Superiority; p = 0.697, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -5.7, 95% CI 2-sided [-28.8 to 17.3] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 12: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical non-responders; Test type: Superiority; p = 0.126, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -20.0, 95% CI 2-sided [-37.5 to -2.5] — [estimate comment as in outcome 25, analysis 1]

35. Secondary Outcome: Percentage of Participants Who Achieve Enhanced Endoscopic Response at Week 52
Description: Enhanced endoscopic response was defined as SES-CD reduction from Induction Baseline > 50% (or for an Induction Baseline SES-CD of 4, at least a 2 point reduction from Induction Baseline). SES-CD subscores assess the following: presence and size of ulcers in 5 visualized bowel segments; extent of ulcerated surface in 5 visualized bowel segments; extent of affected surface in 5 visualized bowel segments; presence and type of narrowings in 5 visualized bowel segments. Subscores range from 0 to 15, and are summed for a total SES-CD score ranging from 0 to 56; higher scores indicate greater severity of mucosal inflammation.
Time Frame: Week 52
Population: as for outcome 31
Measure: Number; unit: percentage of participants
Arm/Group | Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction | Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction | Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction | Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction | Upadacitinib 3 mg BID in Extension/ Placebo in Induction | Upadacitinib 6 mg BID in Extension/ Placebo in Induction | Upadacitinib 12 mg BID in Extension/ Placebo in Induction | Upadacitinib 24 mg QD in Extension/ Placebo in Induction
Number analyzed (Participants) | 52 | 18 | 50 | 33 | 9 | 5 | 9 | 4
percentage of participants
  Responders: number analyzed (Participants) | 20 | 8 | 16 | 10 | 1 | 0 | 0 | 0
  Responders | 40.0 | 50.0 | 68.8 | 30.0 | 100 |  |  |
  Non-responders: number analyzed (Participants) | 32 | 10 | 34 | 23 | 8 | 5 | 9 | 4
  Non-responders | 12.5 | 0 | 11.8 | 17.4 | 0 | 20.0 | 11.1 | 25.0
  Clinical responders: number analyzed (Participants) | 32 | 14 | 29 | 19 | 6 | 1 | 4 | 1
  Clinical responders | 28.1 | 28.6 | 44.8 | 36.8 | 16.7 | 0 | 0 | 100
  Clinical non-responders: number analyzed (Participants) | 20 | 4 | 21 | 14 | 3 | 4 | 5 | 3
  Clinical non-responders | 15.0 | 0 | 9.5 | 0 | 0 | 25.0 | 20.0 | 0
Statistical Analysis 1: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Responders; Test type: Superiority; p = 0.691, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 10.0, 95% CI 2-sided [-30.8 to 50.8] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 2: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Responders; Test type: Superiority; p = 0.086, Chi-squared — [p-value comment as in outcome 27, analysis 11]; Risk Difference (RD) = 28.8, 95% CI 2-sided [-2.5 to 60.0] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 3: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Responders; Test type: Superiority; p = 0.702, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -10.0, 95% CI 2-sided [-45.6 to 25.6] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 4: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Non-responders; Test type: Superiority; p = 0.557, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -12.5, 95% CI 2-sided [-24.0 to -1.0] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 5: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Non-responders; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -0.7, 95% CI 2-sided [-16.5 to 15.0] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 6: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Non-responders; Test type: Superiority; p = 0.707, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 4.9, 95% CI 2-sided [-14.4 to 24.2] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 7: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical responders; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 0.4, 95% CI 2-sided [-27.9 to 28.8] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 8: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical responders; Test type: Superiority; p = 0.175, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 16.7, 95% CI 2-sided [-7.2 to 40.6] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 9: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical responders; Test type: Superiority; p = 0.517, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 8.7, 95% CI 2-sided [-18.0 to 35.4] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 10: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical non-responders; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -15.0, 95% CI 2-sided [-30.6 to 0.6] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 11: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical non-responders; Test type: Superiority; p = 0.663, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -5.5, 95% CI 2-sided [-25.5 to 14.6] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 12: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical non-responders; Test type: Superiority; p = 0.251, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -15.0, 95% CI 2-sided [-30.6 to 0.6] — [estimate comment as in outcome 25, analysis 1]

36. Secondary Outcome: Percentage of Participants Who Achieve Endoscopic Improvement at Week 52
Description: Endoscopic Improvement: SES-CD reduction from Induction Baseline > 50% or endoscopic remission. Endoscopic remission was defined as SES-CD <= 4 and at least 2 points reduction versus Induction Baseline and no subscore > 1 in any individual variable. SES-CD subscores assess the following: presence and size of ulcers in 5 visualized bowel segments; extent of ulcerated surface in 5 visualized bowel segments; extent of affected surface in 5 visualized bowel segments; presence and type of narrowings in 5 visualized bowel segments. Subscores range from 0 to 15, and are summed for a total SES-CD score ranging from 0 to 56; higher scores indicate greater severity of mucosal inflammation.
Time Frame: Week 52
Population: as for outcome 31
Measure: Number; unit: percentage of participants
Arm/Group | Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction | Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction | Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction | Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction | Upadacitinib 3 mg BID in Extension/ Placebo in Induction | Upadacitinib 6 mg BID in Extension/ Placebo in Induction | Upadacitinib 12 mg BID in Extension/ Placebo in Induction | Upadacitinib 24 mg QD in Extension/ Placebo in Induction
Number analyzed (Participants) | 52 | 18 | 50 | 33 | 9 | 5 | 9 | 4
percentage of participants
  Responders: number analyzed (Participants) | 20 | 8 | 16 | 10 | 1 | 0 | 0 | 0
  Responders | 50.0 | 50.0 | 68.8 | 30.0 | 100 |  |  |
  Non-responders: number analyzed (Participants) | 32 | 10 | 34 | 23 | 8 | 5 | 9 | 4
  Non-responders | 12.5 | 10.0 | 11.8 | 17.4 | 0 | 20.0 | 11.1 | 25.0
  Clinical responders: number analyzed (Participants) | 32 | 14 | 29 | 19 | 6 | 1 | 4 | 1
  Clinical responders | 34.4 | 35.7 | 44.8 | 36.8 | 16.7 | 0 | 0 | 100
  Clinical non-responders: number analyzed (Participants) | 20 | 4 | 21 | 14 | 3 | 4 | 5 | 3
  Clinical non-responders | 15.0 | 0 | 9.5 | 0 | 0 | 25.0 | 20.0 | 0
Statistical Analysis 1: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Responders; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 0.0, 95% CI 2-sided [-41.0 to 41.0] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 2: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Responders; Test type: Superiority; p = 0.257, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 18.8, 95% CI 2-sided [-12.8 to 50.3] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 3: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Responders; Test type: Superiority; p = 0.440, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -20.0, 95% CI 2-sided [-55.9 to 15.9] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 4: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Non-responders; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -2.5, 95% CI 2-sided [-24.3 to 19.3] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 5: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Non-responders; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -0.7, 95% CI 2-sided [-16.5 to 15.0] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 6: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Non-responders; Test type: Superiority; p = 0.440, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -20.0, 95% CI 2-sided [-55.9 to 15.9] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 7: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical responders; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 1.3, 95% CI 2-sided [-28.7 to 31.4] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 8: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical responders; Test type: Superiority; p = 0.404, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 10.5, 95% CI 2-sided [-14.0 to 34.9] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 9: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical responders; Test type: Superiority; p = 0.859, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 2.5, 95% CI 2-sided [-24.8 to 29.7] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 10: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical non-responders; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -15.0, 95% CI 2-sided [-30.6 to 0.6] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 11: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical non-responders; Test type: Superiority; p = 0.663, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -5.5, 95% CI 2-sided [-25.5 to 14.6] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 12: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical non-responders; Test type: Superiority; p = 0.251, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -15.0, 95% CI 2-sided [-30.6 to 0.6] — [estimate comment as in outcome 25, analysis 1]

37. Secondary Outcome: Percentage of Participants Who Achieve Endoscopic Healing at Week 52
Description: Endoscopic healing was defined as SES-CD ulcerated surface subscore of 0 in subjects with SES-CD ulcerated surface subscore >= 1 at Induction Baseline. SES-CD subscores assess the following: presence and size of ulcers in 5 visualized bowel segments; extent of ulcerated surface in 5 visualized bowel segments; extent of affected surface in 5 visualized bowel segments; presence and type of narrowings in 5 visualized bowel segments. Subscores range from 0 to 15, and are summed for a total SES-CD score ranging from 0 to 56; higher scores indicate greater severity of mucosal inflammation.
Time Frame: Week 52
Population: as for outcome 31
Measure: Number; unit: percentage of participants
Arm/Group | Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction | Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction | Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction | Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction | Upadacitinib 3 mg BID in Extension/ Placebo in Induction | Upadacitinib 6 mg BID in Extension/ Placebo in Induction | Upadacitinib 12 mg BID in Extension/ Placebo in Induction | Upadacitinib 24 mg QD in Extension/ Placebo in Induction
Number analyzed (Participants) | 52 | 18 | 50 | 33 | 9 | 5 | 9 | 4
percentage of participants
  Responders: number analyzed (Participants) | 20 | 8 | 16 | 10 | 1 | 0 | 0 | 0
  Responders | 15.0 | 25.0 | 50.0 | 0 | 0 |  |  |
  Non-responders: number analyzed (Participants) | 32 | 10 | 34 | 23 | 8 | 5 | 9 | 4
  Non-responders | 9.4 | 10.0 | 8.8 | 8.7 | 0 | 20.0 | 0 | 0
  Clinical responders: number analyzed (Participants) | 32 | 14 | 29 | 19 | 6 | 1 | 4 | 1
  Clinical responders | 9.4 | 21.4 | 31.0 | 10.5 | 0 | 0 | 0 | 0
  Clinical non-responders: number analyzed (Participants) | 20 | 4 | 21 | 14 | 3 | 4 | 5 | 3
  Clinical non-responders | 15.0 | 0 | 9.5 | 0 | 0 | 25.0 | 0 | 0
Statistical Analysis 1: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Responders; Test type: Superiority; p = 0.606, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 10.0, 95% CI 2-sided [-23.8 to 43.8] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 2: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Responders; Test type: Superiority; p = 0.034, Chi-squared — P-value was calculated based on chi-square test (or Fisher's exact test if >= 20% of the cells had expected cell count < 5). Prespecified significant at the 0.5 level; Risk Difference (RD) = 35.0, 95% CI 2-sided [5.9 to 64.1] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 3: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Responders; Test type: Superiority; p = 0.532, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -15.0, 95% CI 2-sided [-30.6 to 0.6] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 4: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Non-responders; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 0.6, 95% CI 2-sided [-20.5 to 21.8] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 5: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Non-responders; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -0.6, 95% CI 2-sided [-14.4 to 13.3] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 6: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Non-responders; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -0.7, 95% CI 2-sided [-16.0 to 14.6] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 7: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical responders; Test type: Superiority; p = 0.350, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 12.1, 95% CI 2-sided [-11.7 to 35.8] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 8: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical responders; Test type: Superiority; p = 0.034, Chi-squared — [p-value comment as in outcome 37, analysis 2]; Risk Difference (RD) = 21.7, 95% CI 2-sided [2.0 to 41.3] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 9: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical responders; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 1.2, 95% CI 2-sided [-15.9 to 18.3] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 10: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical non-responders; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -15.0, 95% CI 2-sided [-30.6 to 0.6] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 11: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical non-responders; Test type: Superiority; p = 0.663, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -5.5, 95% CI 2-sided [-25.5 to 14.6] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 12: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical non-responders; Test type: Superiority; p = 0.251, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -15.0, 95% CI 2-sided [-30.6 to 0.6] — [estimate comment as in outcome 25, analysis 1]

38. Secondary Outcome: Percentage of Participants Who Achieve Clinical Response Over Time During Extension Phase
Description: Clinical response was defined as average daily stool frequency at least 30% reduction from Induction Baseline and average daily abdominal pain not worse than Induction Baseline OR average daily abdominal pain at least 30% reduction from Induction Baseline and average daily stool frequency not worse than Induction Baseline. The very soft/liquid stool frequency and abdominal pain scores at a visit were the average of the daily values reported during the 7 usable days preceding the scheduled assessment visit. Abdominal Pain was rated on a 4-point scale from 0 (none) to 3 (severe).
Time Frame: Week 20, Week 28, Week 36, Week 44, Week 52
Population: as for outcome 31
Measure: Number; unit: percentage of participants
Arm/Group | Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction | Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction | Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction | Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction | Upadacitinib 3 mg BID in Extension/ Placebo in Induction | Upadacitinib 6 mg BID in Extension/ Placebo in Induction | Upadacitinib 12 mg BID in Extension/ Placebo in Induction | Upadacitinib 24 mg QD in Extension/ Placebo in Induction
Number analyzed (Participants) | 52 | 18 | 50 | 33 | 9 | 5 | 9 | 4
percentage of participants
  Responders, Week 20: number analyzed (Participants) | 20 | 8 | 16 | 10 | 1 | 0 | 0 | 0
  Responders, Week 20 | 85.0 | 100 | 100 | 80.0 | 100 |  |  |
  Responders, Week 28: number analyzed (Participants) | 20 | 8 | 16 | 10 | 1 | 0 | 0 | 0
  Responders, Week 28 | 85.0 | 75.0 | 81.3 | 60.0 | 0 |  |  |
  Responders, Week 36: number analyzed (Participants) | 20 | 8 | 16 | 10 | 1 | 0 | 0 | 0
  Responders, Week 36 | 75.0 | 100 | 75.0 | 50.0 | 100 |  |  |
  Responders, Week 44: number analyzed (Participants) | 20 | 8 | 16 | 10 | 1 | 0 | 0 | 0
  Responders, Week 44 | 50.0 | 87.5 | 81.3 | 40.0 | 0 |  |  |
  Responders, Week 52: number analyzed (Participants) | 20 | 8 | 16 | 10 | 1 | 0 | 0 | 0
  Responders, Week 52 | 55.0 | 87.5 | 68.8 | 50.0 | 100 |  |  |
  Non-responders, Week 20: number analyzed (Participants) | 32 | 10 | 34 | 23 | 8 | 5 | 9 | 4
  Non-responders, Week 20 | 43.8 | 60.0 | 41.2 | 39.1 | 75.0 | 20.0 | 33.3 | 50.0
  Non-responders, Week 28: number analyzed (Participants) | 32 | 10 | 34 | 23 | 8 | 5 | 9 | 4
  Non-responders, Week 28 | 40.6 | 60.0 | 29.4 | 26.1 | 50.0 | 20.0 | 22.2 | 50.0
  Non-responders, Week 36: number analyzed (Participants) | 32 | 10 | 34 | 23 | 8 | 5 | 9 | 4
  Non-responders, Week 36 | 28.1 | 40.0 | 26.5 | 17.4 | 50.0 | 20.0 | 33.3 | 25.0
  Non-responders, Week 44: number analyzed (Participants) | 32 | 10 | 34 | 23 | 8 | 5 | 9 | 4
  Non-responders, Week 44 | 25.0 | 30.0 | 26.5 | 21.7 | 37.5 | 40.0 | 33.3 | 50.0
  Non-responders, Week 52: number analyzed (Participants) | 32 | 10 | 34 | 23 | 8 | 5 | 9 | 4
  Non-responders, Week 52 | 21.9 | 30.0 | 26.5 | 13.0 | 37.5 | 40.0 | 33.3 | 50.0
  Clinical responders, Week 20: number analyzed (Participants) | 32 | 14 | 29 | 19 | 6 | 1 | 4 | 1
  Clinical responders, Week 20 | 78.1 | 100 | 93.1 | 78.9 | 100 | 100 | 25.0 | 100
  Clinical responders, Week 28: number analyzed (Participants) | 32 | 14 | 29 | 19 | 6 | 1 | 4 | 1
  Clinical responders, Week 28 | 78.1 | 78.6 | 69.0 | 57.9 | 66.7 | 100 | 25.0 | 100
  Clinical responders, Week 36: number analyzed (Participants) | 32 | 14 | 29 | 19 | 6 | 1 | 4 | 1
  Clinical responders, Week 36 | 65.6 | 78.6 | 65.5 | 47.4 | 83.3 | 100 | 25.0 | 100
  Clinical responders, Week 44: number analyzed (Participants) | 32 | 14 | 29 | 19 | 6 | 1 | 4 | 1
  Clinical responders, Week 44 | 50.0 | 71.4 | 72.4 | 42.1 | 50.0 | 100 | 25.0 | 100
  Clinical responders, Week 52: number analyzed (Participants) | 32 | 14 | 29 | 19 | 6 | 1 | 4 | 1
  Clinical responders, Week 52 | 50.0 | 71.4 | 62.1 | 42.1 | 66.7 | 100 | 25.0 | 100
  Non-clinical responders, Week 20: number analyzed (Participants) | 20 | 4 | 21 | 14 | 3 | 4 | 5 | 3
  Non-clinical responders, Week 20 | 30.0 | 0 | 14.3 | 14.3 | 33.3 | 0 | 40.0 | 33.3
  Non-clinical responders, Week 28: number analyzed (Participants) | 20 | 4 | 21 | 14 | 3 | 4 | 5 | 3
  Non-clinical responders, Week 28 | 25.0 | 25.0 | 14.3 | 7.1 | 0 | 0 | 20.0 | 33.3
  Non-clinical responders, Week 36: number analyzed (Participants) | 20 | 4 | 21 | 14 | 3 | 4 | 5 | 3
  Non-clinical responders, Week 36 | 15.0 | 25.0 | 9.5 | 0 | 0 | 0 | 40.0 | 0
  Non-clinical responders, Week 44: number analyzed (Participants) | 20 | 4 | 21 | 14 | 3 | 4 | 5 | 3
  Non-clinical responders, Week 44 | 10.0 | 0 | 4.8 | 7.1 | 0 | 25.0 | 40.0 | 33.3
  Non-clinical responders, Week 52: number analyzed (Participants) | 20 | 4 | 21 | 14 | 3 | 4 | 5 | 3
  Non-clinical responders, Week 52 | 10.0 | 0 | 9.5 | 0 | 0 | 25.0 | 40.0 | 33.3
Statistical Analysis 1: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 20; Test type: Superiority; p = 0.536, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 15.0, 95% CI 2-sided [-0.6 to 30.6] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 2: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 20; Test type: Superiority; p = 0.238, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 15.0, 95% CI 2-sided [-0.6 to 30.6] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 3: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Responders, Week 20; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -5.0, 95% CI 2-sided [-34.3 to 24.3] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 4: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 28; Test type: Superiority; p = 0.606, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -10.0, 95% CI 2-sided [-43.8 to 23.8] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 5: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 28; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -3.8, 95% CI 2-sided [-28.5 to 21.0] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 6: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Responders, Week 28; Test type: Superiority; p = 0.181, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -25.0, 95% CI 2-sided [-59.2 to 9.2] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 7: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 36; Test type: Superiority; p = 0.281, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 25.0, 95% CI 2-sided [6.0 to 44.0] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 8: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 36; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 0.0, 95% CI 2-sided [-28.5 to 28.5] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 9: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Responders, Week 36; Test type: Superiority; p = 0.231, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -25.0, 95% CI 2-sided [-61.3 to 11.3] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 10: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 44; Test type: Superiority; p = 0.099, Chi-squared — [p-value comment as in outcome 26, analysis 5]; Risk Difference (RD) = 37.5, 95% CI 2-sided [5.8 to 69.2] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 11: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 44; Test type: Superiority; p = 0.052, Chi-squared — [p-value comment as in outcome 26, analysis 5]; Risk Difference (RD) = 31.3, 95% CI 2-sided [2.2 to 60.3] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 12: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Responders, Week 44; Test type: Superiority; p = 0.709, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -10.0, 95% CI 2-sided [-47.4 to 27.4] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 13: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 52; Test type: Superiority; p = 0.194, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 32.5, 95% CI 2-sided [0.9 to 64.1] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 14: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 52; Test type: Superiority; p = 0.400, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 13.8, 95% CI 2-sided [-17.7 to 45.2] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 15: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Responders, Week 52; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -5.0, 95% CI 2-sided [-42.9 to 32.9] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 16: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 20; Test type: Superiority; p = 0.477, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 16.3, 95% CI 2-sided [-18.6 to 51.1] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 17: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 20; Test type: Superiority; p = 0.833, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -2.6, 95% CI 2-sided [-26.4 to 21.3] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 18: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Non-responders, Week 20; Test type: Superiority; p = 0.732, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -4.6, 95% CI 2-sided [-30.9 to 21.7] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 19: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 28; Test type: Superiority; p = 0.468, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 19.4, 95% CI 2-sided [-15.4 to 54.2] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 20: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 28; Test type: Superiority; p = 0.339, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -11.2, 95% CI 2-sided [-34.1 to 11.7] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 21: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Non-responders, Week 28; Test type: Superiority; p = 0.263, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -14.5, 95% CI 2-sided [-39.3 to 10.2] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 22: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 36; Test type: Superiority; p = 0.697, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 11.9, 95% CI 2-sided [-22.3 to 46.0] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 23: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 36; Test type: Superiority; p = 0.880, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -1.7, 95% CI 2-sided [-23.2 to 19.9] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 24: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Non-responders, Week 36; Test type: Superiority; p = 0.355, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -10.7, 95% CI 2-sided [-32.7 to 11.2] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 25: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 44; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 5.0, 95% CI 2-sided [-27.1 to 37.1] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 26: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 44; Test type: Superiority; p = 0.891, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 1.5, 95% CI 2-sided [-19.6 to 22.6] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 27: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Non-responders, Week 44; Test type: Superiority; p = 0.779, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -3.3, 95% CI 2-sided [-25.8 to 19.3] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 28: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 52; Test type: Superiority; p = 0.678, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 8.1, 95% CI 2-sided [-23.7 to 39.9] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 29: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 52; Test type: Superiority; p = 0.663, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 4.6, 95% CI 2-sided [-16.0 to 25.2] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 30: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Non-responders, Week 52; Test type: Superiority; p = 0.494, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -8.8, 95% CI 2-sided [-28.7 to 11.0] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 31: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 20; Test type: Superiority; p = 0.083, Chi-squared — [p-value comment as in outcome 26, analysis 5]; Risk Difference (RD) = 21.9, 95% CI 2-sided [7.6 to 36.2] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 32: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 20; Test type: Superiority; p = 0.151, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 15.0, 95% CI 2-sided [-2.1 to 32.0] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 33: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical responders, Week 20; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 0.8, 95% CI 2-sided [-22.4 to 24.1] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 34: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 28; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 0.4, 95% CI 2-sided [-25.4 to 26.3] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 35: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 28; Test type: Superiority; p = 0.417, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -9.2, 95% CI 2-sided [-31.3 to 12.9] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 36: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical responders, Week 28; Test type: Superiority; p = 0.125, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -20.2, 95% CI 2-sided [-46.7 to 6.2] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 37: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 36; Test type: Superiority; p = 0.497, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 12.9, 95% CI 2-sided [-14.1 to 40.0] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 38: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 36; Test type: Superiority; p = 0.993, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -0.1, 95% CI 2-sided [-24.0 to 23.8] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 39: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical responders, Week 36; Test type: Superiority; p = 0.200, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -18.3, 95% CI 2-sided [-46.1 to 9.6] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 40: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 44; Test type: Superiority; p = 0.177, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 21.4, 95% CI 2-sided [-7.9 to 50.8] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 41: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 44; Test type: Superiority; p = 0.074, Chi-squared — [p-value comment as in outcome 26, analysis 5]; Risk Difference (RD) = 22.4, 95% CI 2-sided [-1.4 to 46.2] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 42: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical responders, Week 44; Test type: Superiority; p = 0.585, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -7.9, 95% CI 2-sided [-36.1 to 20.3] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 43: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 52; Test type: Superiority; p = 0.177, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 21.4, 95% CI 2-sided [-7.9 to 50.8] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 44: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 52; Test type: Superiority; p = 0.343, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 12.1, 95% CI 2-sided [-12.7 to 36.8] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 45: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical responders, Week 52; Test type: Superiority; p = 0.585, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -7.9, 95% CI 2-sided [-36.1 to 20.3] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 46: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 20; Test type: Superiority; p = 0.539, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -30.0, 95% CI 2-sided [-50.1 to -9.9] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 47: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 20; Test type: Superiority; p = 0.277, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -15.7, 95% CI 2-sided [-40.8 to 9.3] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 48: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 20; Test type: Superiority; p = 0.422, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -15.7, 95% CI 2-sided [-42.9 to 11.5] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 49: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 28; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 0.0, 95% CI 2-sided [-46.5 to 46.5] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 50: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 28; Test type: Superiority; p = 0.454, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -10.7, 95% CI 2-sided [-34.9 to 13.5] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 51: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 28; Test type: Superiority; p = 0.364, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -17.9, 95% CI 2-sided [-41.1 to 5.4] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 52: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 36; Test type: Superiority; p = 0.544, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 10.0, 95% CI 2-sided [-35.2 to 55.2] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 53: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 36; Test type: Superiority; p = 0.663, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -5.5, 95% CI 2-sided [-25.5 to 14.6] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 54: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 36; Test type: Superiority; p = 0.251, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -15.0, 95% CI 2-sided [-30.6 to 0.6] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 55: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 44; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -10.0, 95% CI 2-sided [-23.1 to 3.1]
Statistical Analysis 56: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 44; Test type: Superiority; p = 0.606, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -5.2, 95% CI 2-sided [-21.2 to 10.8] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 57: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 44; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -2.9, 95% CI 2-sided [-21.7 to 16.0] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 58: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 52; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -10.0, 95% CI 2-sided [-23.1 to 3.1] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 59: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 52; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -0.5, 95% CI 2-sided [-18.7 to 17.7] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 60: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 52; Test type: Superiority; p = 0.501, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -10.0, 95% CI 2-sided [-23.1 to 3.1] — [estimate comment as in outcome 25, analysis 1]

39. Secondary Outcome: Percentage of Participants Who Achieve Enhanced Clinical Response Over Time During Extension Phase
Description: Enhanced clinical response was defined as average daily stool frequency at least 60% reduction from Induction Baseline and average daily abdominal pain not worse than Induction Baseline OR average daily abdominal pain at least 35% reduction from Induction Baseline and average daily stool frequency not worse than Induction Baseline or modified clinical remission (average daily stool frequency ≤ 2.8 and not worse than Induction baseline AND average daily abdominal pain ≤ 1.0 and not worse than Induction baseline). The very soft/liquid stool frequency and abdominal pain scores at a visit were the average of the daily values reported during the 7 usable days preceding the scheduled assessment visit. Abdominal Pain was rated on a 4-point scale from 0 (none) to 3 (severe).
Time Frame: Week 20, Week 28, Week 36, Week 44, Week 52
Population: as for outcome 31
Measure: Number; unit: percentage of participants
Arm/Group | Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction | Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction | Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction | Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction | Upadacitinib 3 mg BID in Extension/ Placebo in Induction | Upadacitinib 6 mg BID in Extension/ Placebo in Induction | Upadacitinib 12 mg BID in Extension/ Placebo in Induction | Upadacitinib 24 mg QD in Extension/ Placebo in Induction
Number analyzed (Participants) | 52 | 18 | 50 | 33 | 9 | 5 | 9 | 4
percentage of participants
  Responders, Week 20: number analyzed (Participants) | 20 | 8 | 16 | 10 | 1 | 0 | 0 | 0
  Responders, Week 20 | 70.0 | 87.5 | 100 | 70.0 | 100 |  |  |
  Responders, Week 28: number analyzed (Participants) | 20 | 8 | 16 | 10 | 1 | 0 | 0 | 0
  Responders, Week 28 | 80.0 | 75.0 | 81.3 | 60.0 | 0 |  |  |
  Responders, Week 36: number analyzed (Participants) | 20 | 8 | 16 | 10 | 1 | 0 | 0 | 0
  Responders, Week 36 | 75.0 | 100 | 75.0 | 40.0 | 100 |  |  |
  Responders, Week 44: number analyzed (Participants) | 20 | 8 | 16 | 10 | 1 | 0 | 0 | 0
  Responders, Week 44 | 50.0 | 62.5 | 75.0 | 40.0 | 0 |  |  |
  Responders, Week 52: number analyzed (Participants) | 20 | 8 | 16 | 10 | 1 | 0 | 0 | 0
  Responders, Week 52 | 50.0 | 87.5 | 68.8 | 50.0 | 100 |  |  |
  Non-responders, Week 20: number analyzed (Participants) | 32 | 10 | 34 | 23 | 8 | 5 | 9 | 4
  Non-responders, Week 20 | 34.4 | 50.0 | 38.2 | 26.1 | 50.0 | 20.0 | 33.3 | 25.0
  Non-responders, Week 28: number analyzed (Participants) | 32 | 10 | 34 | 23 | 8 | 5 | 9 | 4
  Non-responders, Week 28 | 37.5 | 60.0 | 29.4 | 21.7 | 70.0 | 20.0 | 22.2 | 50.0
  Non-responders, Week 36: number analyzed (Participants) | 32 | 10 | 34 | 23 | 8 | 5 | 9 | 4
  Non-responders, Week 36 | 28.1 | 40.0 | 26.5 | 17.4 | 50.0 | 20.0 | 33.3 | 25.0
  Non-responders, Week 44: number analyzed (Participants) | 32 | 10 | 34 | 23 | 8 | 5 | 9 | 4
  Non-responders, Week 44 | 21.9 | 30.0 | 23.5 | 21.7 | 37.5 | 20.0 | 33.3 | 50.0
  Non-responders, Week 52: number analyzed (Participants) | 32 | 10 | 34 | 23 | 8 | 5 | 9 | 4
  Non-responders, Week 52 | 21.9 | 30.0 | 26.5 | 13.0 | 37.5 | 40.0 | 33.3 | 50.0
  Clinical responders, Week 20: number analyzed (Participants) | 32 | 14 | 29 | 19 | 6 | 1 | 4 | 1
  Clinical responders, Week 20 | 62.5 | 85.7 | 93.1 | 63.2 | 83.3 | 100 | 25.0 | 100
  Clinical responders, Week 28: number analyzed (Participants) | 32 | 14 | 29 | 19 | 6 | 1 | 4 | 1
  Clinical responders, Week 28 | 71.9 | 78.6 | 69.0 | 57.9 | 66.7 | 100 | 25.0 | 100
  Clinical responders, Week 36: number analyzed (Participants) | 32 | 14 | 29 | 19 | 6 | 1 | 4 | 1
  Clinical responders, Week 36 | 65.6 | 78.6 | 65.5 | 42.1 | 83.3 | 100 | 25.0 | 100
  Clinical responders, Week 44: number analyzed (Participants) | 32 | 14 | 29 | 19 | 6 | 1 | 4 | 1
  Clinical responders, Week 44 | 50.0 | 57.1 | 65.5 | 42.1 | 50.0 | 100 | 25.0 | 100
  Clinical responders, Week 52: number analyzed (Participants) | 32 | 14 | 29 | 19 | 6 | 1 | 4 | 1
  Clinical responders, Week 52 | 46.9 | 71.4 | 62.1 | 42.1 | 66.7 | 100 | 25.0 | 100
  Clinical non-responders, Week 20: number analyzed (Participants) | 20 | 4 | 21 | 14 | 3 | 4 | 5 | 3
  Clinical non-responders, Week 20 | 25.0 | 0 | 9.5 | 7.1 | 0 | 0 | 40.0 | 0
  Clinical non-responders, Week 28: number analyzed (Participants) | 20 | 4 | 21 | 14 | 3 | 4 | 5 | 3
  Clinical non-responders, Week 28 | 25.0 | 25.0 | 14.3 | 0 | 0 | 0 | 20.0 | 33.3
  Clinical non-responders, Week 36: number analyzed (Participants) | 20 | 4 | 21 | 14 | 3 | 4 | 5 | 3
  Clinical non-responders, Week 36 | 15.0 | 25.0 | 9.5 | 0 | 0 | 0 | 40.0 | 0
  Clinical non-responders, Week 44: number analyzed (Participants) | 20 | 4 | 21 | 14 | 3 | 4 | 5 | 3
  Clinical non-responders, Week 44 | 5.0 | 0 | 4.8 | 7.1 | 0 | 0 | 40.0 | 33.3
  Clinical non-responders, Week 52: number analyzed (Participants) | 20 | 4 | 21 | 14 | 3 | 4 | 5 | 3
  Clinical non-responders, Week 52 | 10.0 | 0 | 9.5 | 0 | 0 | 25.0 | 40.0 | 33.3
Statistical Analysis 1: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 20; Test type: Superiority; p = 0.633, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 17.5, 95% CI 2-sided [-13.0 to 48.0] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 2: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 20; Test type: Superiority; p = 0.0024, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 30.0, 95% CI 2-sided [9.9 to 50.1] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 3: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Responders, Week 20; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 0.0, 95% CI 2-sided [-34.8 to 34.8] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 4: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 28; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -5.0, 95% CI 2-sided [-39.8 to 29.8] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 5: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 28; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 1.3, 95% CI 2-sided [-24.7 to 27.2] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 6: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Responders, Week 28; Test type: Superiority; p = 0.384, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -20.0, 95% CI 2-sided [-55.1 to 15.1] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 7: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 36; Test type: Superiority; p = 0.281, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 25.0, 95% CI 2-sided [6.0 to 44.0] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 8: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 36; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 0.0, 95% CI 2-sided [-28.5 to 28.5] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 9: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Responders, Week 36; Test type: Superiority; p = 0.108, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -35.0, 95% CI 2-sided [-70.8 to 0.8] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 10: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 44; Test type: Superiority; p = 0.686, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 12.5, 95% CI 2-sided [-27.6 to 52.6] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 11: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 44; Test type: Superiority; p = 0.126, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 25.0, 95% CI 2-sided [-5.5 to 55.5] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 12: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Responders, Week 44; Test type: Superiority; p = 0.709, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -10.0, 95% CI 2-sided [-47.4 to 27.4] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 13: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 52; Test type: Superiority; p = 0.099, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 37.5, 95% CI 2-sided [5.8 to 69.2] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 14: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 52; Test type: Superiority; p = 0.257, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 18.8, 95% CI 2-sided [-12.8 to 50.3] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 15: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Responders, Week 52; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 0.0, 95% CI 2-sided [-38.0 to 38.0] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 16: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 20; Test type: Superiority; p = 0.465, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 15.6, 95% CI 2-sided [-19.5 to 50.7] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 17: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 20; Test type: Superiority; p = 0.745, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 3.9, 95% CI 2-sided [-19.3 to 27.0] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 18: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Non-responders, Week 20; Test type: Superiority; p = 0.512, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -8.3, 95% CI 2-sided [-32.6 to 16.1] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 19: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 28; Test type: Superiority; p = 0.281, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 22.5, 95% CI 2-sided [-12.2 to 57.2] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 20: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 28; Test type: Superiority; p = 0.486, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -8.1, 95% CI 2-sided [-30.8 to 14.6] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 21: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Non-responders, Week 28; Test type: Superiority; p = 0.212, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -15.8, 95% CI 2-sided [-39.5 to 8.0] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 22: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 36; Test type: Superiority; p = 0.697, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 11.9, 95% CI 2-sided [-22.3 to 46.0] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 23: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 36; Test type: Superiority; p = 0.880, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -1.7, 95% CI 2-sided [-23.2 to 19.9] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 24: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Non-responders, Week 36; Test type: Superiority; p = 0.355, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -10.7, 95% CI 2-sided [-32.7 to 11.2] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 25: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 44; Test type: Superiority; p = 0.678, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 8.1, 95% CI 2-sided [-23.7 to 39.9] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 26: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 44; Test type: Superiority; p = 0.873, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 1.7, 95% CI 2-sided [-18.6 to 21.9] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 27: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Non-responders, Week 44; Test type: Superiority; p = 0.990, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -0.1, 95% CI 2-sided [-22.3 to 22.0] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 28: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 52; Test type: Superiority; p = 0.678, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 8.1, 95% CI 2-sided [-23.7 to 39.9] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 29: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 52; Test type: Superiority; p = 0.663, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 4.6, 95% CI 2-sided [-16.0 to 25.2] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 30: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Non-responders, Week 52; Test type: Superiority; p = 0.494, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -8.8, 95% CI 2-sided [-28.7 to 11.0] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 31: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 20; Test type: Superiority; p = 0.169, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 23.2, 95% CI 2-sided [-1.6 to 48.1] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 32: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 20; Test type: Superiority; p = 0.005, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 30.6, 95% CI 2-sided [11.5 to 49.7] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 33: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical responders, Week 20; Test type: Superiority; p = 0.963, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 0.7, 95% CI 2-sided [-26.8 to 28.1] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 34: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 28; Test type: Superiority; p = 0.729, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 6.7, 95% CI 2-sided [-19.8 to 33.2] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 35: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 28; Test type: Superiority; p = 0.804, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -2.9, 95% CI 2-sided [-25.8 to 20.0] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 36: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical responders, Week 28; Test type: Superiority; p = 0.306, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -14.0, 95% CI 2-sided [-41.1 to 13.1] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 37: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 36; Test type: Superiority; p = 0.497, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 12.9, 95% CI 2-sided [-14.1 to 40.0] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 38: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 36; Test type: Superiority; p = 0.993, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -0.1, 95% CI 2-sided [-24.0 to 23.8] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 39: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical responders, Week 36; Test type: Superiority; p = 0.101, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -23.5, 95% CI 2-sided [-51.2 to 4.1] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 40: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 44; Test type: Superiority; p = 0.655, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 7.1, 95% CI 2-sided [-24.0 to 38.3] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 41: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 44; Test type: Superiority; p = 0.221, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 15.5, 95% CI 2-sided [-9.0 to 40.0] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 42: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical responders, Week 44; Test type: Superiority; p = 0.585, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -7.9, 95% CI 2-sided [-36.1 to 20.3] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 43: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 52; Test type: Superiority; p = 0.124, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 24.6, 95% CI 2-sided [-4.8 to 53.9] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 44: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 52; Test type: Superiority; p = 0.234, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 15.2, 95% CI 2-sided [-9.5 to 39.9] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 45: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical responders, Week 52; Test type: Superiority; p = 0.741, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -4.8, 95% CI 2-sided [-32.9 to 23.4] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 46: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 20; Test type: Superiority; p = 0.544, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -25.0, 95% CI 2-sided [-44.0 to -6.0] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 47: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 20; Test type: Superiority; p = 0.238, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -15.5, 95% CI 2-sided [-38.2 to 7.3] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 48: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 20; Test type: Superiority; p = 0.364, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -17.9, 95% CI 2-sided [-41.1 to 5.4] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 49: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 28; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 0.0, 95% CI 2-sided [-46.5 to 46.5] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 50: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 28; Test type: Superiority; p = 0.454, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -10.7, 95% CI 2-sided [-34.9 to 13.5] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 51: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 28; Test type: Superiority; p = 0.063, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -25.0, 95% CI 2-sided [-44.0 to -6.0] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 52: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 36; Test type: Superiority; p = 0.544, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 10.0, 95% CI 2-sided [-35.2 to 55.2] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 53: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 36; Test type: Superiority; p = 0.663, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -5.5, 95% CI 2-sided [-25.5 to 14.6] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 54: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 36; Test type: Superiority; p = 0.251, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -15.0, 95% CI 2-sided [-30.6 to 0.6] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 55: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 44; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -5.0, 95% CI 2-sided [-14.6 to 4.6] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 56: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 44; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -0.2, 95% CI 2-sided [-13.4 to 13.0] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 57: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 44; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 2.1, 95% CI 2-sided [-14.4 to 18.7] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 58: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 52; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -10.0, 95% CI 2-sided [-23.1 to 3.1] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 59: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 52; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -0.5, 95% CI 2-sided [-18.7 to 17.7] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 60: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 52; Test type: Superiority; p = 0.501, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -10.0, 95% CI 2-sided [-23.1 to 3.1] — [estimate comment as in outcome 25, analysis 1]

40. Secondary Outcome: Percentage of Participants Who Achieve Enhanced Clinical Response Over Time During Extension Phase Among Participants In Enhanced Clinical Response At Week 16
Description: as for outcome 39
Time Frame: Week 20, Week 28, Week 36, Week 44, Week 52
Population: Subjects from ITT population with enhanced clinical response at Week 16. Non responder imputation.
Measure: Number; unit: percentage of participants
Arm/Group | Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction | Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction | Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction | Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction | Upadacitinib 3 mg BID in Extension/ Placebo in Induction | Upadacitinib 6 mg BID in Extension/ Placebo in Induction | Upadacitinib 12 mg BID in Extension/ Placebo in Induction | Upadacitinib 24 mg QD in Extension/ Placebo in Induction
Number analyzed (Participants) | 30 | 13 | 28 | 16 | 4 | 1 | 2 | 1
percentage of participants
  Responders, Week 20: number analyzed (Participants) | 20 | 7 | 16 | 9 | 0 | 0 | 0 | 0
  Responders, Week 20 | 70.0 | 100 | 100 | 66.7 |  |  |  |
  Responders, Week 28: number analyzed (Participants) | 20 | 7 | 16 | 9 | 0 | 0 | 0 | 0
  Responders, Week 28 | 80.0 | 71.4 | 81.3 | 55.6 |  |  |  |
  Responders, Week 36: number analyzed (Participants) | 20 | 7 | 16 | 9 | 0 | 0 | 0 | 0
  Responders, Week 36 | 75.0 | 100 | 75.0 | 33.3 |  |  |  |
  Responders, Week 44: number analyzed (Participants) | 20 | 7 | 16 | 9 | 0 | 0 | 0 | 0
  Responders, Week 44 | 50.0 | 71.4 | 75.0 | 33.3 |  |  |  |
  Responders, Week 52: number analyzed (Participants) | 20 | 7 | 16 | 9 | 0 | 0 | 0 | 0
  Responders, Week 52 | 50.0 | 85.7 | 68.8 | 44.4 |  |  |  |
  Non-responders, Week 20: number analyzed (Participants) | 10 | 6 | 12 | 7 | 4 | 1 | 2 | 1
  Non-responders, Week 20 | 50.0 | 83.3 | 83.3 | 57.1 | 100 | 100 | 50.0 | 100
  Non-responders, Week 28: number analyzed (Participants) | 10 | 6 | 12 | 7 | 4 | 1 | 2 | 1
  Non-responders, Week 28 | 70.0 | 83.3 | 58.3 | 57.1 | 100 | 100 | 50.0 | 100
  Non-responders, Week 36: number analyzed (Participants) | 10 | 6 | 12 | 7 | 4 | 1 | 2 | 1
  Non-responders, Week 36 | 50.0 | 50.0 | 58.3 | 57.1 | 100 | 100 | 50.0 | 100
  Non-responders, Week 44: number analyzed (Participants) | 10 | 6 | 12 | 7 | 4 | 1 | 2 | 1
  Non-responders, Week 44 | 50.0 | 50.0 | 58.3 | 57.1 | 75.0 | 100 | 50.0 | 100
  Non-responders, Week 52: number analyzed (Participants) | 10 | 6 | 12 | 7 | 4 | 1 | 2 | 1
  Non-responders, Week 52 | 40.0 | 50.0 | 58.3 | 42.9 | 75.0 | 100 | 50.0 | 100
  Clinical Responders, Week 20: number analyzed (Participants) | 30 | 13 | 28 | 15 | 4 | 1 | 2 | 1
  Clinical Responders, Week 20 | 63.3 | 92.3 | 92.9 | 66.7 | 100 | 100 | 50.0 | 100
  Clinical Responders, Week 28: number analyzed (Participants) | 30 | 13 | 28 | 15 | 4 | 1 | 2 | 1
  Clinical Responders, Week 28 | 76.7 | 76.9 | 71.4 | 60.0 | 100 | 100 | 50.0 | 100
  Clinical Responders, Week 36: number analyzed (Participants) | 30 | 13 | 28 | 15 | 4 | 1 | 2 | 1
  Clinical Responders, Week 36 | 66.7 | 76.9 | 67.9 | 46.7 | 100 | 100 | 50.0 | 100
  Clinical Responders, Week 44: number analyzed (Participants) | 30 | 13 | 28 | 15 | 4 | 1 | 2 | 1
  Clinical Responders, Week 44 | 50.0 | 61.5 | 67.9 | 46.7 | 75.0 | 100 | 50.0 | 100
  Clinical Responders, Week 52: number analyzed (Participants) | 30 | 13 | 28 | 15 | 4 | 1 | 2 | 1
  Clinical Responders, Week 52 | 46.7 | 69.2 | 64.3 | 46.7 | 75.0 | 100 | 50.0 | 100
  Clinical Non-responders, Week 20: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Clinical Non-responders, Week 20 |  |  |  | 0 |  |  |  |
  Clinical Non-responders, Week 28: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Clinical Non-responders, Week 28 |  |  |  | 0 |  |  |  |
  Clinical Non-responders, Week 36: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Clinical Non-responders, Week 36 |  |  |  | 0 |  |  |  |
  Clinical Non-responders, Week 44: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Clinical Non-responders, Week 44 |  |  |  | 0 |  |  |  |
  Clinical Non-responders, Week 52: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Clinical Non-responders, Week 52 |  |  |  | 0 |  |  |  |
Statistical Analysis 1: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 20; Test type: Superiority; p = 0.155, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 30.0, 95% CI 2-sided [9.9 to 50.1] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 2: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 20; Test type: Superiority; p = 0.024, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 30.0, 95% CI 2-sided [9.9 to 50.1] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 3: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Responders, Week 20; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -3.3, 95% CI 2-sided [-40.1 to 33.4] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 4: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 28; Test type: Superiority; p = 0.633, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -8.6, 95% CI 2-sided [-46.4 to 29.2] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 5: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 28; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 1.3, 95% CI 2-sided [-24.7 to 27.2] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 6: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Responders, Week 28; Test type: Superiority; p = 0.209, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -24.4, 95% CI 2-sided [-61.3 to 12.5] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 7: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 36; Test type: Superiority; p = 0.283, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 25.0, 95% CI 2-sided [6.0 to 44.0] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 8: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 36; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 0.0, 95% CI 2-sided [-28.5 to 28.5] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 9: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Responders, Week 36; Test type: Superiority; p = 0.048, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -41.7, 95% CI 2-sided [-77.8 to -5.5] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 10: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 44; Test type: Superiority; p = 0.408, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 21.4, 95% CI 2-sided [-18.6 to 61.4] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 11: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 44; Test type: Superiority; p = 0.126, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 25.0, 95% CI 2-sided [-5.5 to 55.5] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 12: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Responders, Week 44; Test type: Superiority; p = 0.454, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -16.7, 95% CI 2-sided [-54.5 to 21.1] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 13: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 52; Test type: Superiority; p = 0.183, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 35.7, 95% CI 2-sided [1.8 to 69.7] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 14: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 52; Test type: Superiority; p = 0.257, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 18.8, 95% CI 2-sided [-12.8 to 50.3] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 15: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Responders, Week 52; Test type: Superiority; p = 1.000, ANOVA — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -5.6, 95% CI 2-sided [-44.7 to 33.6] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 16: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 20; Test type: Superiority; p = 0.307, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 33.3, 95% CI 2-sided [-9.7 to 76.3] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 17: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 20; Test type: Superiority; p = 0.172, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 33.3, 95% CI 2-sided [-4.1 to 70.8] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 18: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Non-responders, Week 20; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 7.1, 95% CI 2-sided [-40.9 to 55.1] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 19: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 28; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 13.3, 95% CI 2-sided [-27.8 to 54.5] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 20: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 28; Test type: Superiority; p = 0.675, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -11.7, 95% CI 2-sided [-51.5 to 28.1] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 21: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Non-responders, Week 28; Test type: Superiority; p = 0.644, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -12.9, 95% CI 2-sided [-59.2 to 33.5] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 22: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 36; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 0.0, 95% CI 2-sided [-50.6 to 50.6] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 23: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 36; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 8.3, 95% CI 2-sided [-33.4 to 50.0] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 24: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Non-responders, Week 36; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 7.1, 95% CI 2-sided [-40.9 to 55.1] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 25: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 44; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 0.0, 95% CI 2-sided [-50.6 to 50.6] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 26: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 44; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 8.3, 95% CI 2-sided [-33.4 to 50.0] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 27: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Non-responders, Week 44; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 7.1, 95% CI 2-sided [-40.9 to 55.1] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 28: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 52; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 10.0, 95% CI 2-sided [-40.2 to 60.2] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 29: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 52; Test type: Superiority; p = 0.392, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 18.3, 95% CI 2-sided [-22.9 to 59.6] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 30: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Non-responders, Week 52; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 2.9, 95% CI 2-sided [-44.7 to 50.5] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 31: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 20; Test type: Superiority; p = 0.070, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 29.0, 95% CI 2-sided [6.5 to 51.5] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 32: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 20; Test type: Superiority; p = 0.007, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 29.5, 95% CI 2-sided [9.8 to 49.2] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 33: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical responders, Week 20; Test type: Superiority; p = 0.826, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 3.3, 95% CI 2-sided [-26.1 to 32.8] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 34: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 28; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 0.3, 95% CI 2-sided [-27.2 to 27.7] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 35: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 28; Test type: Superiority; p = 0.649, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -5.2, 95% CI 2-sided [-27.8 to 17.3] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 36: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical responders, Week 28; Test type: Superiority; p = 0.304, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -16.7, 95% CI 2-sided [-45.7 to 12.4] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 37: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 36; Test type: Superiority; p = 0.720, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 10.3, 95% CI 2-sided [-18.2 to 38.7] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 38: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 36; Test type: Superiority; p = 0.923, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 1.2, 95% CI 2-sided [-23.0 to 25.4] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 39: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical responders, Week 36; Test type: Superiority; p = 0.197, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -20.0, 95% CI 2-sided [-50.4 to 10.4] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 40: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 44; Test type: Superiority; p = 0.486, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 11.5, 95% CI 2-sided [-20.4 to 43.5] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 41: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 44; Test type: Superiority; p = 0.168, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 17.9, 95% CI 2-sided [-7.0 to 42.7] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 42: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical responders, Week 44; Test type: Superiority; p = 0.833, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -3.3, 95% CI 2-sided [-34.3 to 27.6] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 43: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 52; Test type: Superiority; p = 0.173, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 22.6, 95% CI 2-sided [-8.2 to 53.4] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 44: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 52; Test type: Superiority; p = 0.178, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 17.6, 95% CI 2-sided [-7.6 to 42.8] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 45: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical responders, Week 52; Test type: Superiority; p = 1.000, ANCOVA — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 0.0, 95% CI 2-sided [-30.9 to 30.9] — [estimate comment as in outcome 25, analysis 1]

41. Secondary Outcome: Percentage of Participants Who Achieve Clinical Remission Over Time During Extension Phase Among Participants With an Average Daily Stool Frequency ≥ 2.5 and Average Daily Abdominal Pain ≥ 2.0 at Induction Baseline
Description: as for outcome 27
Time Frame: Week 20, Week 28, Week 36, Week 44, Week 52
Population: Participants from ITT population with man average daily stool frequency >= 2.5 and average daily abdominal pain >= 2.0 at Induction Baseline. Participants Receiving Upadacitinib in Induction. Non responder imputation.
Measure: Number; unit: percentage of participants
Arm/Group | Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction | Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction | Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction | Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction
Number analyzed (Participants) | 23 | 11 | 23 | 14
percentage of participants
  Responders, Week 20: number analyzed (Participants) | 9 | 6 | 8 | 5
  Responders, Week 20 | 44.4 | 16.7 | 37.5 | 20.0
  Responders, Week 28: number analyzed (Participants) | 9 | 6 | 8 | 5
  Responders, Week 28 | 55.6 | 16.7 | 50.0 | 40.0
  Responders, Week 36: number analyzed (Participants) | 9 | 6 | 8 | 5
  Responders, Week 36 | 44.4 | 16.7 | 50.0 | 20.0
  Responders, Week 44: number analyzed (Participants) | 9 | 6 | 8 | 5
  Responders, Week 44 | 44.4 | 0 | 50.0 | 40.0
  Responders, Week 52: number analyzed (Participants) | 9 | 6 | 8 | 5
  Responders, Week 52 | 33.3 | 33.3 | 50.0 | 20.0
  Non-responders, Week 20: number analyzed (Participants) | 14 | 5 | 15 | 9
  Non-responders, Week 20 | 21.4 | 40.0 | 6.7 | 11.1
  Non-responders, Week 28: number analyzed (Participants) | 14 | 5 | 15 | 9
  Non-responders, Week 28 | 21.4 | 40.0 | 6.7 | 22.2
  Non-responders, Week 36: number analyzed (Participants) | 14 | 5 | 15 | 9
  Non-responders, Week 36 | 21.4 | 20.0 | 0 | 22.2
  Non-responders, Week 44: number analyzed (Participants) | 14 | 5 | 15 | 9
  Non-responders, Week 44 | 14.3 | 20.0 | 6.7 | 11.1
  Non-responders, Week 52: number analyzed (Participants) | 14 | 5 | 15 | 9
  Non-responders, Week 52 | 7.1 | 20.0 | 13.3 | 22.2
  Clinical responders, Week 20: number analyzed (Participants) | 17 | 10 | 15 | 9
  Clinical responders, Week 20 | 41.2 | 30.0 | 26.7 | 22.2
  Clinical responders, Week 28: number analyzed (Participants) | 17 | 10 | 15 | 9
  Clinical responders, Week 28 | 47.1 | 30.0 | 33.3 | 44.4
  Clinical responders, Week 36: number analyzed (Participants) | 17 | 10 | 15 | 9
  Clinical responders, Week 36 | 41.2 | 20.0 | 26.7 | 33.3
  Clinical responders, Week 44: number analyzed (Participants) | 17 | 10 | 15 | 9
  Clinical responders, Week 44 | 35.3 | 10.0 | 33.3 | 33.3
  Clinical responders, Week 52: number analyzed (Participants) | 17 | 10 | 15 | 9
  Clinical responders, Week 52 | 23.5 | 30.0 | 40.0 | 33.3
  Clinical non-responders, Week 20: number analyzed (Participants) | 6 | 1 | 8 | 5
  Clinical non-responders, Week 20 | 0 | 0 | 0 | 0
  Clinical non-responders, Week 28: number analyzed (Participants) | 6 | 1 | 8 | 5
  Clinical non-responders, Week 28 | 0 | 0 | 0 | 0
  Clinical non-responders, Week 36: number analyzed (Participants) | 6 | 1 | 8 | 5
  Clinical non-responders, Week 36 | 0 | 0 | 0 | 0
  Clinical non-responders, Week 44: number analyzed (Participants) | 6 | 1 | 8 | 5
  Clinical non-responders, Week 44 | 0 | 0 | 0 | 0
  Clinical non-responders, Week 52: number analyzed (Participants) | 6 | 1 | 8 | 5
  Clinical non-responders, Week 52 | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 20; Test type: Superiority; p = 0.580, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -27.8, 95% CI 2-sided [-71.9 to 16.3] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 2: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 20; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -6.9, 95% CI 2-sided [-53.6 to 39.7] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 3: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Responders, Week 20; Test type: Superiority; p = 0.580, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -24.4, 95% CI 2-sided [-72.2 to 23.3] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 4: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 28; Test type: Superiority; p = 0.287, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -38.9, 95% CI 2-sided [-83.0 to 5.2] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 5: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 28; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -5.6, 95% CI 2-sided [-53.0 to 41.9] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 6: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Responders, Week 28; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -15.6, 95% CI 2-sided [-69.4 to 38.3] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 7: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 36; Test type: Superiority; p = 0.580, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -27.8, 95% CI 2-sided [-71.9 to 16.3] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 8: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 36; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 5.6, 95% CI 2-sided [-41.9 to 53.0] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 9: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Responders, Week 36; Test type: Superiority; p = 0.580, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -24.4, 95% CI 2-sided [-72.2 to 23.3] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 10: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 44; Test type: Superiority; p = 0.103, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -44.4, 95% CI 2-sided [-76.9 to -12.0] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 11: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 44; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 5.6, 95% CI 2-sided [-41.9 to 53.0] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 12: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Responders, Week 44; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -4.4, 95% CI 2-sided [-58.3 to 49.4] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 13: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 52; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 0.0, 95% CI 2-sided [-48.7 to 48.7] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 14: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 52; Test type: Superiority; p = 0.637, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 16.7, 95% CI 2-sided [-29.7 to 63.0] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 15: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Responders, Week 52; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -13.3, 95% CI 2-sided [-60.0 to 33.3] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 16: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 20; Test type: Superiority; p = 0.570, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 18.6, 95% CI 2-sided [-29.4 to 66.6] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 17: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 20; Test type: Superiority; p = 0.330, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -14.8, 95% CI 2-sided [-39.7 to 10.2] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 18: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Non-responders, Week 20; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -10.3, 95% CI 2-sided [-40.0 to 19.4] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 19: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 28; Test type: Superiority; p = 0.570, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 18.6, 95% CI 2-sided [-29.4 to 66.6] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 20: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 28; Test type: Superiority; p = 0.330, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -14.8, 95% CI 2-sided [-39.7 to 10.2] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 21: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Non-responders, Week 28; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 0.8, 95% CI 2-sided [-33.8 to 35.4] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 22: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 36; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -1.4, 95% CI 2-sided [-42.6 to 39.7] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 23: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 36; Test type: Superiority; p = 0.100, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -21.4, 95% CI 2-sided [-42.9 to 0.1] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 24: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Non-responders, Week 36; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 0.8, 95% CI 2-sided [-33.8 to 35.4] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 25: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 44; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 5.7, 95% CI 2-sided [-33.8 to 45.3] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 26: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 44; Test type: Superiority; p = 0.598, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -7.6, 95% CI 2-sided [-29.9 to 14.6] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 27: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Non-responders, Week 44; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -3.2, 95% CI 2-sided [-30.7 to 24.3] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 28: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 52; Test type: Superiority; p = 0.468, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 12.9, 95% CI 2-sided [-24.7 to 50.4]; Risk difference = (upadacitinib higher dose - upadacitinib 3 mg BID). 95% confidence intervals for risk difference were calculated based on normal approximation using proc FREQ
Statistical Analysis 29: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 52; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 6.2, 95% CI 2-sided [-15.7 to 28.1] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 30: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Non-responders, Week 52; Test type: Superiority; p = 0.538, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 15.1, 95% CI 2-sided [-15.2 to 45.4] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 31: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 20; Test type: Superiority; p = 0.692, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -11.2, 95% CI 2-sided [-48.0 to 25.6] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 32: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 20; Test type: Superiority; p = 0.388, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -14.5, 95% CI 2-sided [-46.9 to 17.9] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 33: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical responders, Week 20; Test type: Superiority; p = 0.418, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -19.0, 95% CI 2-sided [-54.8 to 16.9] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 34: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 28; Test type: Superiority; p = 0.448, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -17.1, 95% CI 2-sided [-54.1 to 20.0] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 35: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 28; Test type: Superiority; p = 0.430, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -13.7, 95% CI 2-sided [-47.4 to 19.9] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 36: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical responders, Week 28; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -2.6, 95% CI 2-sided [-42.8 to 37.6] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 37: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 36; Test type: Superiority; p = 0.406, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -21.2, 95% CI 2-sided [-55.3 to 12.9] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 38: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 36; Test type: Superiority; p = 0.388, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -14.5, 95% CI 2-sided [-46.9 to 17.9] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 39: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical responders, Week 36; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -7.8, 95% CI 2-sided [-46.5 to 30.8] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 40: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 44; Test type: Superiority; p = 0.204, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -25.3, 95% CI 2-sided [-54.7 to 4.1] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 41: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 44; Test type: Superiority; p = 0.907, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -2.0, 95% CI 2-sided [-34.9 to 31.0] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 42: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical responders, Week 44; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -2.0, 95% CI 2-sided [-40.2 to 36.3] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 43: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 52; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 6.5, 95% CI 2-sided [-28.4 to 41.3] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 44: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 52; Test type: Superiority; p = 0.450, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 16.5, 95% CI 2-sided [-15.5 to 48.4] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 45: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical responders, Week 52; Test type: Superiority; p = 0.661, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 9.8, 95% CI 2-sided [-27.0 to 46.6] — [estimate comment as in outcome 25, analysis 1]

42. Secondary Outcome: Percentage of Participants Taking Corticosteroids at Induction Baseline Who Discontinued Corticosteroid Use and Achieve CDAI < 150 Over Time
Description: as for outcome 3
Time Frame: Week 20, Week 28, Week 36, Week 44, Week 52
Population: Participants from ITT population taking corticosteroids at Induction Baseline. Non responder imputation.
Measure: Number; unit: percentage of participants
Arm/Group | Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction | Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction | Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction | Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction | Upadacitinib 3 mg BID in Extension/ Placebo in Induction | Upadacitinib 6 mg BID in Extension/ Placebo in Induction | Upadacitinib 12 mg BID in Extension/ Placebo in Induction | Upadacitinib 24 mg QD in Extension/ Placebo in Induction
Number analyzed (Participants) | 23 | 7 | 20 | 14 | 5 | 0 | 3 | 3
percentage of participants
  Responders, Week 20: number analyzed (Participants) | 8 | 2 | 8 | 5 | 0 | 0 | 0 | 0
  Responders, Week 20 | 50.0 | 50.0 | 75.0 | 0 |  |  |  |
  Responders, Week 28: number analyzed (Participants) | 8 | 2 | 8 | 5 | 0 | 0 | 0 | 0
  Responders, Week 28 | 50.0 | 50.0 | 50.0 | 20.0 |  |  |  |
  Responders, Week 36: number analyzed (Participants) | 8 | 2 | 8 | 5 | 0 | 0 | 0 | 0
  Responders, Week 36 | 50.0 | 100 | 50.0 | 0 |  |  |  |
  Responders, Week 44: number analyzed (Participants) | 8 | 2 | 8 | 5 | 0 | 0 | 0 | 0
  Responders, Week 44 | 37.5 | 50.0 | 50.0 | 20.0 |  |  |  |
  Responders, Week 52: number analyzed (Participants) | 8 | 2 | 8 | 5 | 0 | 0 | 0 | 0
  Responders, Week 52 | 50.0 | 100 | 62.5 | 0 |  |  |  |
  Non-responders, Week 20: number analyzed (Participants) | 15 | 5 | 12 | 9 | 5 | 0 | 3 | 3
  Non-responders, Week 20 | 13.3 | 40.0 | 8.3 | 0 | 0 |  | 0 | 0
  Non-responders, Week 28: number analyzed (Participants) | 15 | 5 | 12 | 9 | 5 | 0 | 3 | 3
  Non-responders, Week 28 | 6.7 | 40.0 | 16.7 | 11.1 | 0 |  | 0 | 0
  Non-responders, Week 36: number analyzed (Participants) | 15 | 5 | 12 | 9 | 5 | 0 | 3 | 3
  Non-responders, Week 36 | 13.3 | 40.0 | 8.3 | 11.1 | 0 |  | 0 | 0
  Non-responders, Week 44: number analyzed (Participants) | 15 | 5 | 12 | 9 | 5 | 0 | 3 | 3
  Non-responders, Week 44 | 26.7 | 40.0 | 25.0 | 11.1 | 0 |  | 0 | 0
  Non-responders, Week 52: number analyzed (Participants) | 15 | 5 | 12 | 9 | 5 | 0 | 3 | 3
  Non-responders, Week 52 | 20.0 | 40.0 | 25.0 | 11.1 | 0 |  | 0 | 0
  Clinical responders, Week 20: number analyzed (Participants) | 15 | 6 | 14 | 8 | 2 | 0 | 1 | 0
  Clinical responders, Week 20 | 40.0 | 50.0 | 50.0 | 0 | 0 |  | 0 |
  Clinical responders, Week 28: number analyzed (Participants) | 15 | 6 | 14 | 8 | 2 | 0 | 1 | 0
  Clinical responders, Week 28 | 33.3 | 50.0 | 42.9 | 25.0 | 0 |  | 0 |
  Clinical responders, Week 36: number analyzed (Participants) | 15 | 6 | 14 | 8 | 2 | 0 | 1 | 0
  Clinical responders, Week 36 | 40.0 | 66.7 | 35.7 | 12.5 | 0 |  | 0 |
  Clinical responders, Week 44: number analyzed (Participants) | 15 | 6 | 14 | 8 | 2 | 0 | 1 | 0
  Clinical responders, Week 44 | 40.0 | 50.0 | 50.0 | 25.0 | 0 |  | 0 |
  Clinical responders, Week 52: number analyzed (Participants) | 15 | 6 | 14 | 8 | 2 | 0 | 1 | 0
  Clinical responders, Week 52 | 46.7 | 66.7 | 57.1 | 12.5 | 0 |  | 0 |
  Clinical non-responders, Week 20: number analyzed (Participants) | 8 | 1 | 6 | 6 | 3 | 0 | 2 | 3
  Clinical non-responders, Week 20 | 0 | 0 | 0 | 0 | 0 |  | 0 | 0
  Clinical non-responders, Week 28: number analyzed (Participants) | 8 | 1 | 6 | 6 | 3 | 0 | 2 | 3
  Clinical non-responders, Week 28 | 0 | 0 | 0 | 0 | 0 |  | 0 | 0
  Clinical non-responders, Week 36: number analyzed (Participants) | 8 | 1 | 6 | 6 | 3 | 0 | 2 | 3
  Clinical non-responders, Week 36 | 0 | 0 | 0 | 0 | 0 |  | 0 | 0
  Clinical non-responders, Week 44: number analyzed (Participants) | 8 | 1 | 6 | 6 | 3 | 0 | 2 | 3
  Clinical non-responders, Week 44 | 12.5 | 0 | 0 | 0 | 0 |  | 0 | 0
  Clinical non-responders, Week 52: number analyzed (Participants) | 8 | 1 | 6 | 6 | 3 | 0 | 2 | 3
  Clinical non-responders, Week 52 | 0 | 0 | 0 | 0 | 0 |  | 0 | 0
Statistical Analysis 1: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 20; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 0.0, 95% CI 2-sided [-77.5 to 77.5] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 2: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 20; Test type: Superiority; p = 0.608, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 25.0, 95% CI 2-sided [-20.8 to 70.8] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 3: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Responders, Week 20; Test type: Superiority; p = 0.105, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -50.0, 95% CI 2-sided [-84.6 to -15.4] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 4: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 28; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 0.0, 95% CI 2-sided [-77.5 to 77.5] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 5: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 28; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 0.0, 95% CI 2-sided [-49.0 to 49.0] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 6: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Responders, Week 28; Test type: Superiority; p = 0.565, ANOVA — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -30.0, 95% CI 2-sided [-79.3 to 19.3] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 7: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 36; Test type: Superiority; p = 0.467, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 50.0, 95% CI 2-sided [15.4 to 84.6] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 8: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 36; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 0.0, 95% CI 2-sided [-49.0 to 49.0] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 9: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Responders, Week 36; Test type: Superiority; p = 0.105, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -50.0, 95% CI 2-sided [-84.6 to -15.4] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 10: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 44; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 12.5, 95% CI 2-sided [-64.5 to 89.5] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 11: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 44; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 12.5, 95% CI 2-sided [-35.7 to 60.7] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 12: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Responders, Week 44; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -17.5, 95% CI 2-sided [-66.0 to 31.0] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 13: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 52; Test type: Superiority; p = 0.467, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 50.0, 95% CI 2-sided [15.4 to 84.6] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 14: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 52; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 12.5, 95% CI 2-sided [-35.7 to 60.7] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 15: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Responders, Week 52; Test type: Superiority; p = 0.105, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -50.0, 95% CI 2-sided [-84.6 to -15.4] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 16: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 20; Test type: Superiority; p = 0.249, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 26.7, 95% CI 2-sided [-19.6 to 72.9] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 17: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 20; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -5.0, 95% CI 2-sided [-28.2 to 18.2] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 18: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Non-responders, Week 20; Test type: Superiority; p = 0.511, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -13.3, 95% CI 2-sided [-30.5 to 3.9] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 19: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 28; Test type: Superiority; p = 0.140, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 33.3, 95% CI 2-sided [-11.4 to 78.1] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 20: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 28; Test type: Superiority; p = 0.569, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 10.0, 95% CI 2-sided [-14.6 to 34.6] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 21: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Non-responders, Week 28; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 4.4, 95% CI 2-sided [-19.7 to 28.5] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 22: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 36; Test type: Superiority; p = 0.249, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 26.7, 95% CI 2-sided [-19.6 to 72.9] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 23: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 36; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -5.0, 95% CI 2-sided [-28.2 to 18.2] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 24: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Non-responders, Week 36; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -2.2, 95% CI 2-sided [-29.0 to 24.6] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 25: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 44; Test type: Superiority; p = 0.613, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 13.3, 95% CI 2-sided [-35.1 to 61.8] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 26: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 44; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -1.7, 95% CI 2-sided [-34.8 to 31.5] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 27: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Non-responders, Week 44; Test type: Superiority; p = 0.615, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -15.6, 95% CI 2-sided [-45.9 to 14.8] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 28: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 52; Test type: Superiority; p = 0.560, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 20.0, 95% CI 2-sided [-27.5 to 67.5] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 29: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 52; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 5.0, 95% CI 2-sided [-26.8 to 36.8]
Statistical Analysis 30: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Non-responders, Week 52; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -8.9, 95% CI 2-sided [-37.7 to 19.9] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 31: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 20; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 10.0, 95% CI 2-sided [-37.1 to 57.1] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 32: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 20; Test type: Superiority; p = 0.588, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 10.0, 95% CI 2-sided [-26.1 to 46.1] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 33: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical responders, Week 20; Test type: Superiority; p = 0.058, Chi-squared — [p-value comment as in outcome 27, analysis 11]; Risk Difference (RD) = -40.0, 95% CI 2-sided [-64.8 to -15.2] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 34: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 28; Test type: Superiority; p = 0.631, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 16.7, 95% CI 2-sided [-29.9 to 63.2] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 35: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 28; Test type: Superiority; p = 0.597, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 9.5, 95% CI 2-sided [-25.7 to 44.8] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 36: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical responders, Week 28; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -8.3, 95% CI 2-sided [-46.7 to 30.0] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 37: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 36; Test type: Superiority; p = 0.361, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 26.7, 95% CI 2-sided [-18.5 to 71.8] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 38: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 36; Test type: Superiority; p = 0.812, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -4.3, 95% CI 2-sided [-39.6 to 31.0] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 39: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical responders, Week 36; Test type: Superiority; p = 0.345, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -27.5, 95% CI 2-sided [-61.3 to 6.3] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 40: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 44; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 10.0, 95% CI 2-sided [-37.1 to 57.1] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 41: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 44; Test type: Superiority; p = 0.588, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 10.0, 95% CI 2-sided [-26.1 to 46.1] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 42: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical responders, Week 44; Test type: Superiority; p = 0.657, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -15.0, 95% CI 2-sided [-53.9 to 23.9] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 43: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 52; Test type: Superiority; p = 0.635, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 20.0, 95% CI 2-sided [-25.4 to 65.4] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 44: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 52; Test type: Superiority; p = 0.573, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 10.5, 95% CI 2-sided [-25.7 to 46.7] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 45: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical responders, Week 52; Test type: Superiority; p = 0.176, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -34.2, 95% CI 2-sided [-68.3 to -0.1] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 46: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 44; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -12.5, 95% CI 2-sided [-35.4 to 10.4] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 47: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 44; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -12.5, 95% CI 2-sided [-35.4 to 10.4] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 48: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 44; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -12.5, 95% CI 2-sided [-35.4 to 10.4] — [estimate comment as in outcome 25, analysis 1]

43. Secondary Outcome: Percentage of Participants Taking Corticosteroids at Induction Baseline Who Discontinued Corticosteroid Use and Achieve Remission At Week 52
Description: Steroid-free remission at Week 52 was defined as both endoscopic remission at Week 52 and clinical remission at Week 52. Endoscopic remission: SES-CD ≤ 4 and at least 2 point reduction versus Induction Baseline and no subscore > 1 in any individual variable. Clinical remission: Average daily stool frequency ≤ 1.5 and not worse than baseline AND average daily abdominal pain ≤ 1.0 and not worse than Induction Baseline. The very soft/liquid stool frequency and abdominal pain scores at a visit were the average of the daily values reported during the 7 usable days preceding the scheduled assessment visit. Abdominal Pain was rated on a 4-point scale from 0 (none) to 3 (severe). See SES-CD description details in the first primary endpoint description of this record.
Time Frame: Baseline, Week 52
Population: Participants from ITT population taking corticosteroids at Induction Baseline. Non responder imputation.
Measure: Number; unit: percentage of participants
Arm/Group | Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction | Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction | Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction | Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction | Upadacitinib 3 mg BID in Extension/ Placebo in Induction | Upadacitinib 6 mg BID in Extension/ Placebo in Induction | Upadacitinib 12 mg BID in Extension/ Placebo in Induction | Upadacitinib 24 mg QD in Extension/ Placebo in Induction
Number analyzed (Participants) | 23 | 7 | 20 | 14 | 5 | 0 | 3 | 3
percentage of participants
  Responders: number analyzed (Participants) | 8 | 2 | 8 | 5 | 0 | 0 | 0 | 0
  Responders | 25.0 | 0 | 37.5 | 0 |  |  |  |
  Non-responders: number analyzed (Participants) | 15 | 5 | 12 | 9 | 5 | 0 | 3 | 3
  Non-responders | 0 | 0 | 0 | 11.1 | 0 |  | 0 | 0
  Clinical Responders: number analyzed (Participants) | 15 | 6 | 14 | 8 | 2 | 0 | 1 | 0
  Clinical Responders | 13.3 | 0 | 21.4 | 12.5 | 0 |  | 0 |
  Clinical non-responders: number analyzed (Participants) | 8 | 1 | 6 | 6 | 3 | 0 | 2 | 3
  Clinical non-responders | 0 | 0 | 0 | 0 | 0 |  | 0 | 0
Statistical Analysis 1: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Responders; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -25.0, 95% CI 2-sided [-55.0 to 5.0] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 2: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Responders; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 12.5, 95% CI 2-sided [-32.5 to 57.5] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 3: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Responders; Test type: Superiority; p = 0.487, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -25.0, 95% CI 2-sided [-55.0 to 5.0] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 4: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Non-respoonders; Test type: Superiority; p = 0.375, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 11.1, 95% CI 2-sided [-9.4 to 31.6] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 5: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical responders; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -13.3, 95% CI 2-sided [-30.5 to 3.9] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 6: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical responders; Test type: Superiority; p = 0.651, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 8.1, 95% CI 2-sided [-19.4 to 35.6] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 7: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical responders; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -0.8, 95% CI 2-sided [-29.5 to 27.8] — [estimate comment as in outcome 25, analysis 1]

44. Secondary Outcome: Percentage of Participants Taking Corticosteroids at Induction Baseline Who Discontinued Corticosteroid Use and Achieve Clinical Remission Over Time
Description: Steroid-free clinical remission was defined as average daily stool frequency <= 1.5 and not worse than Induction Baseline AND average daily abdominal pain <= 1.0 and not worse than Induction Baseline. The very soft/liquid stool frequency and abdominal pain scores at a visit were the average of the daily values reported during the 7 usable days preceding the scheduled assessment visit. Abdominal Pain was rated on a 4-point scale from 0 (none) to 3 (severe).
Time Frame: Week 20, Week 28, Week 36, Week 44, Week 52
Population: Participants from ITT population taking corticosteroids at Induction Baseline. Non responder imputation.
Measure: Number; unit: percentage of participants
Arm/Group | Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction | Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction | Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction | Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction | Upadacitinib 3 mg BID in Extension/ Placebo in Induction | Upadacitinib 6 mg BID in Extension/ Placebo in Induction | Upadacitinib 12 mg BID in Extension/ Placebo in Induction | Upadacitinib 24 mg QD in Extension/ Placebo in Induction
Number analyzed (Participants) | 23 | 7 | 20 | 14 | 5 | 0 | 3 | 3
percentage of participants
  Responders, Week 20: number analyzed (Participants) | 8 | 2 | 8 | 5 | 0 | 0 | 0 | 0
  Responders, Week 20 | 50.0 | 50.0 | 50.0 | 0 |  |  |  |
  Responders, Week 28: number analyzed (Participants) | 8 | 2 | 8 | 5 | 0 | 0 | 0 | 0
  Responders, Week 28 | 37.5 | 50.0 | 50.0 | 20.0 |  |  |  |
  Responders, Week 36: number analyzed (Participants) | 8 | 2 | 8 | 5 | 0 | 0 | 0 | 0
  Responders, Week 36 | 37.5 | 100 | 62.5 | 0 |  |  |  |
  Responders, Week 44: number analyzed (Participants) | 8 | 2 | 8 | 5 | 0 | 0 | 0 | 0
  Responders, Week 44 | 37.5 | 0 | 62.5 | 20.0 |  |  |  |
  Responders, Week 52: number analyzed (Participants) | 8 | 2 | 8 | 5 | 0 | 0 | 0 | 0
  Responders, Week 52 | 25.0 | 100 | 62.5 | 0 |  |  |  |
  Non-responders, Week 20: number analyzed (Participants) | 15 | 5 | 12 | 9 | 5 | 0 | 3 | 3
  Non-responders, Week 20 | 13.3 | 40.0 | 0 | 0 | 0 |  | 0 | 0
  Non-responders, Week 28: number analyzed (Participants) | 15 | 5 | 12 | 9 | 5 | 0 | 3 | 3
  Non-responders, Week 28 | 6.7 | 40.0 | 16.7 | 11.1 | 0 |  | 0 | 0
  Non-responders, Week 36: number analyzed (Participants) | 15 | 5 | 12 | 9 | 5 | 0 | 3 | 3
  Non-responders, Week 36 | 6.7 | 20.0 | 0 | 11.1 | 0 |  | 0 | 0
  Non-responders, Week 44: number analyzed (Participants) | 15 | 5 | 12 | 9 | 5 | 0 | 3 | 3
  Non-responders, Week 44 | 20.0 | 40.0 | 0 | 11.1 | 0 |  | 0 | 0
  Non-responders, Week 52: number analyzed (Participants) | 15 | 5 | 12 | 9 | 5 | 0 | 3 | 3
  Non-responders, Week 52 | 13.3 | 20.0 | 8.3 | 11.1 | 0 |  | 0 | 0
  Clinical responders, Week 20: number analyzed (Participants) | 15 | 6 | 14 | 8 | 2 | 0 | 1 | 0
  Clinical responders, Week 20 | 40.0 | 50.0 | 28.6 | 0 | 0 |  | 0 |
  Clinical responders, Week 28: number analyzed (Participants) | 15 | 6 | 14 | 8 | 2 | 0 | 1 | 0
  Clinical responders, Week 28 | 26.7 | 50.0 | 42.9 | 25.0 | 0 |  | 0 |
  Clinical responders, Week 36: number analyzed (Participants) | 15 | 6 | 14 | 8 | 2 | 0 | 1 | 0
  Clinical responders, Week 36 | 26.7 | 50.0 | 35.7 | 12.5 | 0 |  | 0 |
  Clinical responders, Week 44: number analyzed (Participants) | 15 | 6 | 14 | 8 | 2 | 0 | 1 | 0
  Clinical responders, Week 44 | 40.0 | 33.3 | 35.7 | 25.0 | 0 |  | 0 |
  Clinical responders, Week 52: number analyzed (Participants) | 15 | 6 | 14 | 8 | 2 | 0 | 1 | 0
  Clinical responders, Week 52 | 26.7 | 50.0 | 42.9 | 12.5 | 0 |  | 0 |
  Clinical non-responders, Week 20: number analyzed (Participants) | 8 | 1 | 6 | 6 | 3 | 0 | 2 | 3
  Clinical non-responders, Week 20 | 0 | 0 | 0 | 0 | 0 |  | 0 | 0
  Clinical non-responders, Week 28: number analyzed (Participants) | 8 | 1 | 6 | 6 | 3 | 0 | 2 | 3
  Clinical non-responders, Week 28 | 0 | 0 | 0 | 0 | 0 |  | 0 | 0
  Clinical non-responders, Week 36: number analyzed (Participants) | 8 | 1 | 6 | 6 | 3 | 0 | 2 | 3
  Clinical non-responders, Week 36 | 0 | 0 | 0 | 0 | 0 |  | 0 | 0
  Clinical non-responders, Week 44: number analyzed (Participants) | 8 | 1 | 6 | 6 | 3 | 0 | 2 | 3
  Clinical non-responders, Week 44 | 0 | 0 | 0 | 0 | 0 |  | 0 | 0
  Clinical non-responders, Week 52: number analyzed (Participants) | 8 | 1 | 6 | 6 | 3 | 0 | 2 | 3
  Clinical non-responders, Week 52 | 0 | 0 | 0 | 0 | 0 |  | 0 | 0
Statistical Analysis 1: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 20; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 0.0, 95% CI 2-sided [-77.5 to 77.5] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 2: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 20; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 0.0, 95% CI 2-sided [-49.0 to 49.0] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 3: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Responders, Week 20; Test type: Superiority; p = 0.105, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -50.0, 95% CI 2-sided [-84.6 to -15.4] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 4: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 28; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 12.5, 95% CI 2-sided [-64.5 to 89.5] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 5: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 28; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 12.5, 95% CI 2-sided [-35.7 to 60.7] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 6: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Responders, Week 28; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -17.5, 95% CI 2-sided [-66.0 to 31.0] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 7: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 36; Test type: Superiority; p = 0.444, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 62.5, 95% CI 2-sided [29.0 to 96.0] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 8: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 36; Test type: Superiority; p = 0.619, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 25.0, 95% CI 2-sided [-22.4 to 72.4] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 9: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Responders, Week 36; Test type: Superiority; p = 0.231, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -37.5, 95% CI 2-sided [-71.0 to -4.0] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 10: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 44; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -37.5, 95% CI 2-sided [-71.0 to -4.0] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 11: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 44; Test type: Superiority; p = 0.619, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 25.0, 95% CI 2-sided [-22.4 to 72.4] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 12: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Responders, Week 44; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -17.5, 95% CI 2-sided [-66.0 to 31.0] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 13: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 52; Test type: Superiority; p = 0.133, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 75.0, 95% CI 2-sided [45.0 to 100.0] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 14: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 52; Test type: Superiority; p = 0.315, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 37.5, 95% CI 2-sided [-7.5 to 82.5] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 15: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Responders, Week 52; Test type: Superiority; p = 0.487, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -25.0, 95% CI 2-sided [-55.0 to 5.0] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 16: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 20; Test type: Superiority; p = 0.249, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 26.7, 95% CI 2-sided [-19.6 to 72.9] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 17: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 20; Test type: Superiority; p = 0.487, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -13.3, 95% CI 2-sided [-30.5 to 3.9] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 18: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Non-responders, Week 20; Test type: Superiority; p = 0.511, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -13.3, 95% CI 2-sided [-30.5 to 3.9] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 19: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 28; Test type: Superiority; p = 0.140, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 33.3, 95% CI 2-sided [-11.4 to 78.1] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 20: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 28; Test type: Superiority; p = 0.569, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 10.0, 95% CI 2-sided [-14.6 to 34.6] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 21: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Non-responders, Week 28; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 4.4, 95% CI 2-sided [-19.7 to 28.5] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 22: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 36; Test type: Superiority; p = 0.447, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 13.3, 95% CI 2-sided [-23.9 to 50.6] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 23: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 36; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -6.7, 95% CI 2-sided [-19.3 to 6.0] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 24: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Non-responders, Week 36; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 4.4, 95% CI 2-sided [-19.7 to 28.5] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 25: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 44; Test type: Superiority; p = 0.560, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 20.0, 95% CI 2-sided [-27.5 to 67.5] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 26: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 44; Test type: Superiority; p = 0.231, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -20.0, 95% CI 2-sided [-40.2 to 0.2] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 27: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Non-responders, Week 44; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -8.9, 95% CI 2-sided [-37.7 to 19.9] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 28: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 52; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 6.7, 95% CI 2-sided [-32.4 to 45.7] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 29: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 52; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -5.0, 95% CI 2-sided [-28.2 to 18.2] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 30: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Non-responders, Week 52; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -2.2, 95% CI 2-sided [-29.0 to 24.6] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 31: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 20; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 10.0, 95% CI 2-sided [-37.1 to 57.1] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 32: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 20; Test type: Superiority; p = 0.700, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -11.4, 95% CI 2-sided [-45.7 to 22.8] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 33: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical responders, Week 20; Test type: Superiority; p = 0.058, Chi-squared — [p-value comment as in outcome 27, analysis 11]; Risk Difference (RD) = -40.0, 95% CI 2-sided [-64.8 to -15.2] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 34: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 28; Test type: Superiority; p = 0.354, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 23.3, 95% CI 2-sided [-22.5 to 69.2] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 35: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 28; Test type: Superiority; p = 0.450, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 16.2, 95% CI 2-sided [-18.1 to 50.4] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 36: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical responders, Week 28; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -1.7, 95% CI 2-sided [-39.1 to 35.8] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 37: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 36; Test type: Superiority; p = 0.354, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 23.3, 95% CI 2-sided [-22.5 to 69.2] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 38: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 36; Test type: Superiority; p = 0.700, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 9.0, 95% CI 2-sided [-24.6 to 42.7] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 39: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical responders, Week 36; Test type: Superiority; p = 0.621, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -14.2, 95% CI 2-sided [-46.2 to 17.9] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 40: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 44; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -6.7, 95% CI 2-sided [-51.8 to 38.5] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 41: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 44; Test type: Superiority; p = 0.812, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -4.3, 95% CI 2-sided [-39.6 to 31.0] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 42: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical responders, Week 44; Test type: Superiority; p = 0.657, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -15.0, 95% CI 2-sided [-53.9 to 23.9] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 43: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 52; Test type: Superiority; p = 0.354, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 23.3, 95% CI 2-sided [-22.5 to 69.2] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 44: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 52; Test type: Superiority; p = 0.450, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 16.2, 95% CI 2-sided [-18.1 to 50.4] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 45: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical responders, Week 52; Test type: Superiority; p = 0.621, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -14.2, 95% CI 2-sided [-46.2 to 17.9] — [estimate comment as in outcome 25, analysis 1]

45. Secondary Outcome: Percentage of Participants Taking Corticosteroids at Induction Baseline and With Daily Stool Frequency ≥ 4.0 or Daily Abdominal Pain ≥ 2.0 at Induction Baseline Who Discontinued Corticosteroid Use and Achieve Modified Clinical Remission Over Time
Description: Steroid-free modified clinical remission was defined as average daily stool frequency <= 2.8 and not worse than Induction Baseline AND average daily abdominal pain <= 1.0 and not worse than Induction Baseline. The very soft/liquid stool frequency and abdominal pain scores at a visit were the average of the daily values reported during the 7 usable days preceding the scheduled assessment visit. Abdominal Pain was rated on a 4-point scale from 0 (none) to 3 (severe).
Time Frame: Week 20, Week 28, Week 36, Week 44, Week 52
Population: Participants from ITT population taking corticosteroids at Induction Baseline and Daily Stool Frequency >= 4.0 OR Daily Abdominal Pain >= 2.0 at Induction Baseline. Non responder imputation.
Measure: Number; unit: percentage of participants
Arm/Group | Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction | Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction | Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction | Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction | Upadacitinib 3 mg BID in Extension/ Placebo in Induction | Upadacitinib 6 mg BID in Extension/ Placebo in Induction | Upadacitinib 12 mg BID in Extension/ Placebo in Induction | Upadacitinib 24 mg QD in Extension/ Placebo in Induction
Number analyzed (Participants) | 18 | 7 | 20 | 13 | 4 | 0 | 3 | 3
percentage of participants
  Responders, Week 20: number analyzed (Participants) | 6 | 2 | 8 | 5 | 0 | 0 | 0 | 0
  Responders, Week 20 | 33.3 | 50.0 | 62.5 | 20.0 |  |  |  |
  Responders, Week 28: number analyzed (Participants) | 6 | 2 | 8 | 5 | 0 | 0 | 0 | 0
  Responders, Week 28 | 50.0 | 50.0 | 62.5 | 20.0 |  |  |  |
  Responders, Week 36: number analyzed (Participants) | 6 | 2 | 8 | 5 | 0 | 0 | 0 | 0
  Responders, Week 36 | 50.0 | 100 | 62.5 | 0 |  |  |  |
  Responders, Week 44: number analyzed (Participants) | 6 | 2 | 8 | 5 | 0 | 0 | 0 | 0
  Responders, Week 44 | 33.3 | 50.0 | 62.5 | 20.0 |  |  |  |
  Responders, Week 52: number analyzed (Participants) | 6 | 2 | 8 | 5 | 0 | 0 | 0 | 0
  Responders, Week 52 | 33.3 | 100 | 62.5 | 0 |  |  |  |
  Non-responders, Week 20: number analyzed (Participants) | 12 | 5 | 12 | 8 | 4 | 0 | 3 | 3
  Non-responders, Week 20 | 8.3 | 40.0 | 8.3 | 0 | 0 |  | 0 | 0
  Non-responders, Week 28: number analyzed (Participants) | 12 | 5 | 12 | 8 | 4 | 0 | 3 | 3
  Non-responders, Week 28 | 16.7 | 40.0 | 16.7 | 12.5 | 0 |  | 0 | 0
  Non-responders, Week 36: number analyzed (Participants) | 12 | 5 | 12 | 8 | 4 | 0 | 3 | 3
  Non-responders, Week 36 | 8.3 | 20.0 | 8.3 | 12.5 | 0 |  | 0 | 0
  Non-responders, Week 44: number analyzed (Participants) | 12 | 5 | 12 | 8 | 4 | 0 | 3 | 3
  Non-responders, Week 44 | 16.7 | 40.0 | 0 | 12.5 | 0 |  | 0 | 0
  Non-responders, Week 52: number analyzed (Participants) | 12 | 5 | 12 | 8 | 4 | 0 | 3 | 3
  Non-responders, Week 52 | 8.3 | 20.0 | 16.7 | 12.5 | 0 |  | 0 | 0
  Clinical responders, Week 20: number analyzed (Participants) | 12 | 6 | 14 | 7 | 1 | 0 | 1 | 0
  Clinical responders, Week 20 | 25.0 | 50.0 | 42.9 | 14.3 | 0 |  | 0 |
  Clinical responders, Week 28: number analyzed (Participants) | 12 | 6 | 14 | 7 | 1 | 0 | 1 | 0
  Clinical responders, Week 28 | 41.7 | 50.0 | 50.0 | 28.6 | 0 |  | 0 |
  Clinical responders, Week 36: number analyzed (Participants) | 12 | 6 | 14 | 7 | 1 | 0 | 1 | 0
  Clinical responders, Week 36 | 33.3 | 50.0 | 42.9 | 14.3 | 0 |  | 0 |
  Clinical responders, Week 44: number analyzed (Participants) | 12 | 6 | 14 | 7 | 1 | 0 | 1 | 0
  Clinical responders, Week 44 | 33.3 | 50.0 | 35.7 | 28.6 | 0 |  | 0 |
  Clinical responders, Week 52: number analyzed (Participants) | 12 | 6 | 14 | 7 | 1 | 0 | 1 | 0
  Clinical responders, Week 52 | 25.0 | 50.0 | 50.0 | 14.3 | 0 |  | 0 |
  Clinical non-responders, Week 20: number analyzed (Participants) | 6 | 1 | 6 | 6 | 3 | 0 | 2 | 3
  Clinical non-responders, Week 20 | 0 | 0 | 0 | 0 | 0 |  | 0 | 0
  Clinical non-responders, Week 28: number analyzed (Participants) | 6 | 1 | 6 | 6 | 3 | 0 | 2 | 3
  Clinical non-responders, Week 28 | 0 | 0 | 0 | 0 | 0 |  | 0 | 0
  Clinical non-responders, Week 36: number analyzed (Participants) | 6 | 1 | 6 | 6 | 3 | 0 | 2 | 3
  Clinical non-responders, Week 36 | 0 | 0 | 0 | 0 | 0 |  | 0 | 0
  Clinical non-responders, Week 44: number analyzed (Participants) | 6 | 1 | 6 | 6 | 3 | 0 | 2 | 3
  Clinical non-responders, Week 44 | 0 | 0 | 0 | 0 | 0 |  | 0 | 0
  Clinical non-responders, Week 52: number analyzed (Participants) | 6 | 1 | 6 | 6 | 3 | 0 | 2 | 3
  Clinical non-responders, Week 52 | 0 | 0 | 0 | 0 | 0 |  | 0 | 0
Statistical Analysis 1: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 20; Test type: Superiority; p = 1.000, Chi-squared — P-value was calculated based on chi-square test (or Fisher's exact test if >= 20%of the cells have expected cell count <5); Risk Difference (RD) = 16.7, 95% CI 2-sided [-62.2 to 95.6] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 2: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 20; Test type: Superiority; p = 0.592, Chi-squared — P-value was calculated based on chi-square test (or Fisher's exact test if >= 20% of the cells have expected cell count < 5); Risk Difference (RD) = 29.2, 95% CI 2-sided [-21.3 to 79.6] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 3: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Responders, Week 20; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = -13.3, 95% CI 2-sided [-64.8 to 38.2] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 4: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 28; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = 0.0, 95% CI 2-sided [-80.0 to 80.0] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 5: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 28; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = 12.5, 95% CI 2-sided [-39.7 to 64.7] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 6: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Responders, Week 28; Test type: Superiority; p = 0.545, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = -30.0, 95% CI 2-sided [-83.2 to 23.2] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 7: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 36; Test type: Superiority; p = 0.464, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = 50.0, 95% CI 2-sided [10.0 to 90.0] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 8: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 36; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = 12.5, 95% CI 2-sided [-39.7 to 64.7] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 9: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Responders, Week 36; Test type: Superiority; p = 0.182, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = -50.0, 95% CI 2-sided [-90.0 to -10.0] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 10: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 44; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = 16.7, 95% CI 2-sided [-62.2 to 95.6] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 11: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 44; Test type: Superiority; p = 0.592, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = 29.2, 95% CI 2-sided [-21.3 to 79.6] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 12: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Responders, Week 44; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = -13.3, 95% CI 2-sided [-64.8 to 38.2] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 13: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 52; Test type: Superiority; p = 0.429, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = 66.7, 95% CI 2-sided [28.9 to 100.0] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 14: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 52; Test type: Superiority; p = 0.592, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = 29.2, 95% CI 2-sided [-21.3 to 79.6] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 15: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Responders, Week 52; Test type: Superiority; p = 0.455, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = -33.3, 95% CI 2-sided [-71.1 to 4.4] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 16: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 20; Test type: Superiority; p = 0.191, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = 31.7, 95% CI 2-sided [-14.0 to 77.4] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 17: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 20; Test type: Superiority; p = 1.000, Chi-squared; P-value was calculated based on chi-square test (or Fisher's exact test if >= 20% of the cells have expected cell count < 5); Risk Difference (RD) = 0.0, 95% CI 2-sided [-22.1 to 22.1] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 18: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Non-responders, Week 20; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = -8.3, 95% CI 2-sided [-24.0 to 7.3] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 19: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 28; Test type: Superiority; p = 0.538, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = 23.3, 95% CI 2-sided [-24.5 to 71.2] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 20: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 28; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = 0.0, 95% CI 2-sided [-29.8 to 29.8] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 21: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Non-responders, Week 28; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = -4.2, 95% CI 2-sided [-35.3 to 27.0] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 22: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 36; Test type: Superiority; p = 0.515, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = 11.7, 95% CI 2-sided [-26.7 to 50.1] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 23: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 36; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = 0.0, 95% CI 2-sided [-22.1 to 22.1] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 24: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Non-responders, Week 36; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = 4.2, 95% CI 2-sided [-23.6 to 31.9] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 25: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 44; Test type: Superiority; p = 0.538, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = 23.3, 95% CI 2-sided [-24.5 to 71.2] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 26: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 44; Test type: Superiority; p = 0.478, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = -16.7, 95% CI 2-sided [-37.8 to 4.4] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 27: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Non-responders, Week 44; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = -4.2, 95% CI 2-sided [-35.3 to 27.0] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 28: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 52; Test type: Superiority; p = 0.515, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = 11.7, 95% CI 2-sided [-26.7 to 50.1] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 29: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 52; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = 8.3, 95% CI 2-sided [-17.9 to 34.6] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 30: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Non-responders, Week 52; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = 4.2, 95% CI 2-sided [-23.6 to 31.9] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 31: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical Responders, Week 20; Test type: Superiority; p = 0.344, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = 25.0, 95% CI 2-sided [-21.9 to 71.9] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 32: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical Responders, Week 20; Test type: Superiority; p = 0.429, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = 17.9, 95% CI 2-sided [-17.8 to 53.5] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 33: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical Responders, Week 20; Test type: Superiority; p = 1.000, Chi-squared; [statistical method as in outcome 45, analysis 17]; Risk Difference (RD) = -10.7, 95% CI 2-sided [-46.4 to 25.0] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 34: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical Responders, Week 28; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = 8.3, 95% CI 2-sided [-40.4 to 57.1] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 35: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical Responders, Week 28; Test type: Superiority; p = 0.671, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = 8.3, 95% CI 2-sided [-29.9 to 46.6] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 36: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical Responders, Week 28; Test type: Superiority; p = 0.656, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = -13.1, 95% CI 2-sided [-56.7 to 30.5] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 37: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical Responders, Week 36; Test type: Superiority; p = 0.627, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = 16.7, 95% CI 2-sided [-31.4 to 64.7] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 38: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical Responders, Week 36; Test type: Superiority; p = 0.701, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = 9.5, 95% CI 2-sided [-27.7 to 46.7] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 39: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical Responders, Week 36; Test type: Superiority; p = 0.603, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = -19.0, 95% CI 2-sided [-56.2 to 18.1] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 40: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical Responders, Week 44; Test type: Superiority; p = 0.627, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = 16.7, 95% CI 2-sided [-31.4 to 64.7] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 41: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical Responders, Week 44; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = 2.4, 95% CI 2-sided [-34.2 to 39.0] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 42: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical Responders, Week 44; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = -4.8, 95% CI 2-sided [-47.6 to 38.0] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 43: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical Responders, Week 52; Test type: Superiority; p = 0.344, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = 25.0, 95% CI 2-sided [-21.9 to 71.9] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 44: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical Responders, Week 52; Test type: Superiority; p = 0.248, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = 25.0, 95% CI 2-sided [-10.9 to 60.9] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 45: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical Responders, Week 52; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = -10.7, 95% CI 2-sided [-46.4 to 25.0] — [estimate comment as in outcome 24, analysis 1]

46. Secondary Outcome: Percentage of Participants Taking Corticosteroids at Induction Baseline Who Discontinued Corticosteroid Use and Achieve Endoscopic Remission at Week 52
Description: Steroid-free endoscopic remission was defined as SES-CD <= 4 and at least 2 points reduction versus Induction Baseline and no subscore > 1 in any individual variable. Details of the SES-CD scale are provided in the description of the first primary endpoint.
Time Frame: Baseline, Week 52
Population: Participants from ITT population taking corticosteroids at Induction Baseline. Non responder imputation.
Measure: Number; unit: percentage of participants
Arm/Group | Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction | Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction | Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction | Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction | Upadacitinib 3 mg BID in Extension/ Placebo in Induction | Upadacitinib 6 mg BID in Extension/ Placebo in Induction | Upadacitinib 12 mg BID in Extension/ Placebo in Induction | Upadacitinib 24 mg QD in Extension/ Placebo in Induction
Number analyzed (Participants) | 23 | 7 | 20 | 14 | 5 | 0 | 3 | 3
percentage of participants
  Responders: number analyzed (Participants) | 8 | 2 | 8 | 5 | 0 | 0 | 0 | 0
  Responders | 25.0 | 0 | 50.0 | 0 |  |  |  |
  Non-responders: number analyzed (Participants) | 15 | 5 | 12 | 9 | 5 | 0 | 3 | 3
  Non-responders | 0 | 20.0 | 8.3 | 11.1 | 0 |  | 0 | 0
  Clinical responders: number analyzed (Participants) | 15 | 6 | 14 | 8 | 2 | 0 | 1 | 0
  Clinical responders | 13.3 | 16.7 | 35.7 | 12.5 | 0 |  | 0 |
  Clinical non-responders: number analyzed (Participants) | 8 | 1 | 6 | 6 | 3 | 0 | 2 | 3
  Clinical non-responders | 0 | 0 | 0 | 0 | 0 |  | 0 | 0
Statistical Analysis 1: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Responders; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = -25.0, 95% CI 2-sided [-55.0 to 5.0] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 2: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Responders; Test type: Superiority; p = 0.608, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = 25.0, 95% CI 2-sided [-20.8 to 70.8] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 3: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Responders; Test type: Superiority; p = 0.487, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = -25.0, 95% CI 2-sided [-55.0 to 5.0] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 4: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Non-responders; Test type: Superiority; p = 0.250, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = 20.0, 95% CI 2-sided [-15.1 to 55.1] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 5: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Non-responders; Test type: Superiority; p = 0.444, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = 8.3, 95% CI 2-sided [-7.3 to 24.0] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 6: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Non-responders; Test type: Superiority; p = 0.375, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = 11.1, 95% CI 2-sided [-9.4 to 31.6] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 7: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical responders; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = 3.3, 95% CI 2-sided [-31.1 to 37.8] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 8: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical responders; Test type: Superiority; p = 0.215, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = 22.4, 95% CI 2-sided [-8.0 to 52.8] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 9: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical responders; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = -0.8, 95% CI 2-sided [-29.5 to 27.8] — [estimate comment as in outcome 24, analysis 1]

47. Secondary Outcome: Percentage Of Participants Who Achieve CDAI < 150 Over Time During Extension Phase
Description: as for outcome 3
Time Frame: Week 20, Week 28, Week 36, Week 44, Week 52
Population: Non responder imputation.
Measure: Number; unit: percentage of participants
Arm/Group | Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction | Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction | Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction | Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction | Upadacitinib 3 mg BID in Extension/ Placebo in Induction | Upadacitinib 6 mg BID in Extension/ Placebo in Induction | Upadacitinib 12 mg BID in Extension/ Placebo in Induction | Upadacitinib 24 mg QD in Extension/ Placebo in Induction
Number analyzed (Participants) | 52 | 18 | 50 | 33 | 9 | 5 | 9 | 4
percentage of participants
  Responders, Week 20: number analyzed (Participants) | 20 | 8 | 16 | 10 | 1 | 0 | 0 | 0
  Responders, Week 20 | 65.0 | 50.0 | 75.0 | 50.0 | 0 |  |  |
  Responders, Week 28: number analyzed (Participants) | 20 | 8 | 16 | 10 | 1 | 0 | 0 | 0
  Responders, Week 28 | 75.0 | 25.0 | 62.5 | 60.0 | 0 |  |  |
  Responders, Week 36: number analyzed (Participants) | 20 | 8 | 16 | 10 | 1 | 0 | 0 | 0
  Responders, Week 36 | 70.0 | 75.0 | 62.5 | 30.0 | 0 |  |  |
  Responders, Week 44: number analyzed (Participants) | 20 | 8 | 16 | 10 | 1 | 0 | 0 | 0
  Responders, Week 44 | 45.0 | 37.5 | 62.5 | 40.0 | 0 |  |  |
  Responders, Week 52: number analyzed (Participants) | 20 | 8 | 16 | 10 | 1 | 0 | 0 | 0
  Responders, Week 52 | 55.0 | 50.0 | 68.8 | 40.0 | 0 |  |  |
  Non-responders, Week 20: number analyzed (Participants) | 32 | 10 | 34 | 23 | 8 | 5 | 9 | 4
  Non-responders, Week 20 | 28.1 | 50.0 | 17.6 | 8.7 | 75.0 | 20.0 | 11.1 | 50.0
  Non-responders, Week 28: number analyzed (Participants) | 32 | 10 | 34 | 23 | 8 | 5 | 9 | 4
  Non-responders, Week 28 | 15.6 | 40.0 | 17.6 | 13.0 | 37.5 | 20.0 | 22.2 | 50.0
  Non-responders, Week 36: number analyzed (Participants) | 32 | 10 | 34 | 23 | 8 | 5 | 9 | 4
  Non-responders, Week 36 | 15.6 | 30.0 | 14.7 | 13.0 | 37.5 | 20.0 | 33.3 | 50.0
  Non-responders, Week 44: number analyzed (Participants) | 32 | 10 | 34 | 23 | 8 | 5 | 9 | 4
  Non-responders, Week 44 | 18.8 | 30.0 | 17.6 | 8.7 | 25.0 | 20.0 | 33.3 | 25.0
  Non-responders, Week 52: number analyzed (Participants) | 32 | 10 | 34 | 23 | 8 | 5 | 9 | 4
  Non-responders, Week 52 | 9.4 | 30.0 | 20.6 | 13.0 | 25.0 | 40.0 | 33.3 | 50.0
  Clinical responders, Week 20: number analyzed (Participants) | 32 | 14 | 29 | 19 | 6 | 1 | 4 | 1
  Clinical responders, Week 20 | 59.4 | 64.3 | 51.7 | 36.8 | 83.3 | 100 | 0 | 100
  Clinical responders, Week 28: number analyzed (Participants) | 32 | 14 | 29 | 19 | 6 | 1 | 4 | 1
  Clinical responders, Week 28 | 56.3 | 42.9 | 48.3 | 47.4 | 50.0 | 100 | 25.0 | 100
  Clinical responders, Week 36: number analyzed (Participants) | 32 | 14 | 29 | 19 | 6 | 1 | 4 | 1
  Clinical responders, Week 36 | 59.4 | 64.3 | 44.8 | 31.6 | 50.0 | 100 | 25.0 | 100
  Clinical responders, Week 44: number analyzed (Participants) | 32 | 14 | 29 | 19 | 6 | 1 | 4 | 1
  Clinical responders, Week 44 | 40.6 | 42.9 | 55.2 | 31.6 | 33.3 | 100 | 25.0 | 100
  Clinical responders, Week 52: number analyzed (Participants) | 32 | 14 | 29 | 19 | 6 | 1 | 4 | 1
  Clinical responders, Week 52 | 43.8 | 50.0 | 55.2 | 36.8 | 33.3 | 100 | 25.0 | 100
  Clinical non- responders, Week 20: number analyzed (Participants) | 20 | 4 | 21 | 14 | 3 | 4 | 5 | 3
  Clinical non- responders, Week 20 | 15.0 | 0 | 14.3 | 0 | 33.3 | 0 | 20.0 | 33.3
  Clinical non- responders, Week 28: number analyzed (Participants) | 20 | 4 | 21 | 14 | 3 | 4 | 5 | 3
  Clinical non- responders, Week 28 | 10.0 | 0 | 9.5 | 0 | 0 | 0 | 20.0 | 33.3
  Clinical non- responders, Week 36: number analyzed (Participants) | 20 | 4 | 21 | 14 | 3 | 4 | 5 | 3
  Clinical non- responders, Week 36 | 0 | 0 | 9.5 | 0 | 0 | 0 | 40.0 | 33.3
  Clinical non- responders, Week 44: number analyzed (Participants) | 20 | 4 | 21 | 14 | 3 | 4 | 5 | 3
  Clinical non- responders, Week 44 | 10.0 | 0 | 0 | 0 | 0 | 0 | 40.0 | 0
  Clinical non- responders, Week 52: number analyzed (Participants) | 20 | 4 | 21 | 14 | 3 | 4 | 5 | 3
  Clinical non- responders, Week 52 | 0 | 0 | 9.5 | 0 | 0 | 25.0 | 40.0 | 33.3
Statistical Analysis 1: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 20; Test type: Superiority; p = 0.671, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = -15.0, 95% CI 2-sided [-55.5 to 25.5] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 2: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 20; Test type: Superiority; p = 0.718, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = 10.0, 95% CI 2-sided [-19.8 to 39.8] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 3: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Responders, Week 20; Test type: Superiority; p = 0.461, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = -15.0, 95% CI 2-sided [-52.4 to 22.4] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 4: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 28; Test type: Superiority; p = 0.030, Chi-squared — Statistically significant at 0.05 level. P-value was calculated based on chi-square test (or Fisher's exact test if >= 20% of the cells have expected cell count < 5); Risk Difference (RD) = -50.0, 95% CI 2-sided [-85.5 to -14.5] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 5: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 28; Test type: Superiority; p = 0.483, Chi-squared; [statistical method as in outcome 45, analysis 17]; Risk Difference (RD) = -12.5, 95% CI 2-sided [-42.9 to 17.9] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 6: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Responders, Week 28; Test type: Superiority; p = 0.431, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = -15.0, 95% CI 2-sided [-50.8 to 20.8] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 7: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 36; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = 5.0, 95% CI 2-sided [-31.1 to 41.1] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 8: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 36; Test type: Superiority; p = 0.635, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = -7.5, 95% CI 2-sided [-38.6 to 23.6] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 9: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Responders, Week 36; Test type: Superiority; p = 0.056, Chi-squared — Statistically significant at 0.1 level. P-value was calculated based on chi-square test (or Fisher's exact test if >= 20% of the cells have expected cell count < 5); Risk Difference (RD) = -40.0, 95% CI 2-sided [-74.8 to -5.2] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 10: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 44; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = -7.5, 95% CI 2-sided [-47.5 to 32.5] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 11: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 44; Test type: Superiority; p = 0.296, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = 17.5, 95% CI 2-sided [-14.7 to 49.7] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 12: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Responders, Week 44; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = -5.0, 95% CI 2-sided [-42.4 to 32.4] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 13: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 52; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = -5.0, 95% CI 2-sided [-45.9 to 35.9] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 14: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 52; Test type: Superiority; p = 0.400, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = 13.8, 95% CI 2-sided [-17.7 to 45.2] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 15: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Responders, Week 52; Test type: Superiority; p = 0.439, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = -15.0, 95% CI 2-sided [-52.4 to 22.4] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 16: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 20; Test type: Superiority; p = 0.259, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = 21.9, 95% CI 2-sided [-12.8 to 56.6] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 17: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 20; Test type: Superiority; p = 0.310, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = -10.5, 95% CI 2-sided [-30.6 to 9.7] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 18: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Non-responders, Week 20; Test type: Superiority; p = 0.097, Chi-squared — [p-value comment as in outcome 47, analysis 9]; Risk Difference (RD) = -19.4, 95% CI 2-sided [-38.8 to -0.1] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 19: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 28; Test type: Superiority; p = 0.181, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = 24.4, 95% CI 2-sided [-8.5 to 57.2] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 20: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 28; Test type: Superiority; p = 0.826, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = 2.0, 95% CI 2-sided [-15.9 to 20.0] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 21: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Non-responders, Week 28; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = -2.6, 95% CI 2-sided [-21.2 to 16.1] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 22: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 36; Test type: Superiority; p = 0.369, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = 14.4, 95% CI 2-sided [-16.7 to 45.4] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 23: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 36; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = -0.9, 95% CI 2-sided [-18.2 to 16.4] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 24: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Non-responders, Week 36; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = -2.6, 95% CI 2-sided [-21.2 to 16.1] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 25: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 44; Test type: Superiority; p = 0.660, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = 11.3, 95% CI 2-sided [-20.2 to 42.7] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 26: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 44; Test type: Superiority; p = 0.908, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = -1.1, 95% CI 2-sided [-19.7 to 17.5] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 27: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Non-responders, Week 44; Test type: Superiority; p = 0.446, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = -10.1, 95% CI 2-sided [-27.8 to 7.7] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 28: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 52; Test type: Superiority; p = 0.135, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = 20.6, 95% CI 2-sided [-9.5 to 50.8] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 29: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 52; Test type: Superiority; p = 0.306, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = 11.2, 95% CI 2-sided [-5.7 to 28.1] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 30: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Non-responders, Week 52; Test type: Superiority; p = 0.686, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = 3.7, 95% CI 2-sided [-13.4 to 20.7] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 31: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 20; Test type: Superiority; p = 0.754, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = 4.9, 95% CI 2-sided [-25.4 to 35.2] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 32: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 20; Test type: Superiority; p = 0.548, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = -7.7, 95% CI 2-sided [-32.6 to 17.3] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 33: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical responders, Week 20; Test type: Superiority; p = 0.120, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = -22.5, 95% CI 2-sided [-50.1 to 5.0] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 34: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 28; Test type: Superiority; p = 0.403, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = -13.4, 95% CI 2-sided [-44.5 to 17.7] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 35: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 28; Test type: Superiority; p = 0.533, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = -8.0, 95% CI 2-sided [-33.0 to 17.0] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 36: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical responders, Week 28; Test type: Superiority; p = 0.539, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = -8.9, 95% CI 2-sided [-37.2 to 19.4] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 37: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 36; Test type: Superiority; p = 0.754, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = 4.9, 95% CI 2-sided [-25.4 to 35.2] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 38: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 36; Test type: Superiority; p = 0.256, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = -14.5, 95% CI 2-sided [-39.4 to 10.3] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 39: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical responders, Week 36; Test type: Superiority; p = 0.055, Chi-squared — Statistically significant at 0.1 level; [statistical method as in outcome 45, analysis 17]; Risk Difference (RD) = -27.8, 95% CI 2-sided [-54.7 to -0.8] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 40: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 44; Test type: Superiority; p = 0.887, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = 2.2, 95% CI 2-sided [-28.8 to 33.2] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 41: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 44; Test type: Superiority; p = 0.256, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = 14.5, 95% CI 2-sided [-10.3 to 39.4] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 42: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical responders, Week 44; Test type: Superiority; p = 0.518, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = -9.0, 95% CI 2-sided [-36.0 to 17.9] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 43: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 52; Test type: Superiority; p = 0.695, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = 6.3, 95% CI 2-sided [-25.1 to 37.6] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 44: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 52; Test type: Superiority; p = 0.373, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = 11.4, 95% CI 2-sided [-13.5 to 36.4] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 45: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical responders, Week 52; Test type: Superiority; p = 0.628, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = -6.9, 95% CI 2-sided [-34.6 to 20.8] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 46: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 20; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = -15.0, 95% CI 2-sided [-30.6 to 0.6] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 47: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 20; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = -0.7, 95% CI 2-sided [-22.4 to 20.9] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 48: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 20; Test type: Superiority; p = 0.251, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = -15.0, 95% CI 2-sided [-30.6 to 0.6] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 49: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 28; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = -10.0, 95% CI 2-sided [-23.1 to 3.1] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 50: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 28; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = -0.5, 95% CI 2-sided [-18.7 to 17.7] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 51: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 28; Test type: Superiority; p = 0.501, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = -10.0, 95% CI 2-sided [-23.1 to 3.1] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 52: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 36; Test type: Superiority; p = 0.488, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = 9.5, 95% CI 2-sided [-3.0 to 22.1] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 53: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 44; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = -10.0, 95% CI 2-sided [-23.1 to 3.1] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 54: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 44; Test type: Superiority; p = 0.232, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = -10.0, 95% CI 2-sided [-23.1 to 3.1] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 55: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 44; Test type: Superiority; p = 0.501, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = -10.0, 95% CI 2-sided [-23.1 to 3.1] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 56: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 52; Test type: Superiority; p = 0.488, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = 9.5, 95% CI 2-sided [-3.0 to 22.1] — [estimate comment as in outcome 24, analysis 1]

48. Secondary Outcome: Percentage of Participants With Decrease in CDAI ≥ 70 Points From Induction Baseline Over Time During Extension Phase
Description: as for outcome 4
Time Frame: Week 20, Week 28, Week 36, Week 44, Week 52
Population: Non responder imputation.
Measure: Number; unit: percentage of participants
Arm/Group | Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction | Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction | Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction | Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction | Upadacitinib 3 mg BID in Extension/ Placebo in Induction | Upadacitinib 6 mg BID in Extension/ Placebo in Induction | Upadacitinib 12 mg BID in Extension/ Placebo in Induction | Upadacitinib 24 mg QD in Extension/ Placebo in Induction
Number analyzed (Participants) | 52 | 18 | 50 | 33 | 9 | 5 | 9 | 4
percentage of participants
  Responders, Week 20: number analyzed (Participants) | 20 | 8 | 16 | 10 | 1 | 0 | 0 | 0
  Responders, Week 20 | 80.0 | 100 | 93.8 | 60.0 | 100 |  |  |
  Responders, Week 28: number analyzed (Participants) | 20 | 8 | 16 | 10 | 1 | 0 | 0 | 0
  Responders, Week 28 | 85.0 | 62.5 | 68.8 | 60.0 | 0 |  |  |
  Responders, Week 36: number analyzed (Participants) | 20 | 8 | 16 | 10 | 1 | 0 | 0 | 0
  Responders, Week 36 | 75.0 | 100 | 75.0 | 50.0 | 100 |  |  |
  Responders, Week 44: number analyzed (Participants) | 20 | 8 | 16 | 10 | 1 | 0 | 0 | 0
  Responders, Week 44 | 60.0 | 87.5 | 81.3 | 40.0 | 100 |  |  |
  Responders, Week 52: number analyzed (Participants) | 20 | 8 | 16 | 10 | 1 | 0 | 0 | 0
  Responders, Week 52 | 55.0 | 75.0 | 75.0 | 40.0 | 100 |  |  |
  Non-responders, Week 20: number analyzed (Participants) | 32 | 10 | 34 | 23 | 8 | 5 | 9 | 4
  Non-responders, Week 20 | 46.9 | 70.0 | 47.1 | 34.8 | 75.0 | 20.0 | 22.2 | 50.0
  Non-responders, Week 28: number analyzed (Participants) | 32 | 10 | 34 | 23 | 8 | 5 | 9 | 4
  Non-responders, Week 28 | 34.4 | 60.0 | 29.4 | 30.4 | 50.0 | 20.0 | 33.3 | 50.0
  Non-responders, Week 36: number analyzed (Participants) | 32 | 10 | 34 | 23 | 8 | 5 | 9 | 4
  Non-responders, Week 36 | 28.1 | 50.0 | 26.5 | 17.4 | 50.0 | 20.0 | 33.3 | 50.0
  Non-responders, Week 44: number analyzed (Participants) | 32 | 10 | 34 | 23 | 8 | 5 | 9 | 4
  Non-responders, Week 44 | 25.0 | 30.0 | 29.4 | 26.1 | 37.5 | 40.0 | 33.3 | 25.0
  Non-responders, Week 52: number analyzed (Participants) | 32 | 10 | 34 | 23 | 8 | 5 | 9 | 4
  Non-responders, Week 52 | 12.5 | 40.0 | 26.5 | 17.4 | 37.5 | 40.0 | 33.3 | 50.0
  Clinical responders, Week 20: number analyzed (Participants) | 32 | 14 | 29 | 19 | 6 | 1 | 4 | 1
  Clinical responders, Week 20 | 75.0 | 100 | 89.7 | 63.2 | 100 | 100 | 0 | 100
  Clinical responders, Week 28: number analyzed (Participants) | 32 | 14 | 29 | 19 | 6 | 1 | 4 | 1
  Clinical responders, Week 28 | 75.0 | 71.4 | 58.6 | 57.9 | 66.7 | 100 | 25.0 | 100
  Clinical responders, Week 36: number analyzed (Participants) | 32 | 14 | 29 | 19 | 6 | 1 | 4 | 1
  Clinical responders, Week 36 | 65.6 | 85.7 | 62.1 | 42.1 | 83.3 | 100 | 25.0 | 100
  Clinical responders, Week 44: number analyzed (Participants) | 32 | 14 | 29 | 19 | 6 | 1 | 4 | 1
  Clinical responders, Week 44 | 56.3 | 71.4 | 72.4 | 42.1 | 66.7 | 100 | 25.0 | 100
  Clinical responders, Week 52: number analyzed (Participants) | 32 | 14 | 29 | 19 | 6 | 1 | 4 | 1
  Clinical responders, Week 52 | 46.9 | 71.4 | 62.1 | 36.8 | 66.7 | 100 | 25.0 | 100
  Clinical non-responders, Week 20: number analyzed (Participants) | 20 | 4 | 21 | 14 | 3 | 4 | 5 | 3
  Clinical non-responders, Week 20 | 35.0 | 25.0 | 23.8 | 14.3 | 33.3 | 0 | 40.0 | 33.3
  Clinical non-responders, Week 28: number analyzed (Participants) | 20 | 4 | 21 | 14 | 3 | 4 | 5 | 3
  Clinical non-responders, Week 28 | 20.0 | 25.0 | 19.0 | 14.3 | 0 | 0 | 40.0 | 33.3
  Clinical non-responders, Week 36: number analyzed (Participants) | 20 | 4 | 21 | 14 | 3 | 4 | 5 | 3
  Clinical non-responders, Week 36 | 15.0 | 25.0 | 14.3 | 7.1 | 0 | 0 | 40.0 | 33.3
  Clinical non-responders, Week 44: number analyzed (Participants) | 20 | 4 | 21 | 14 | 3 | 4 | 5 | 3
  Clinical non-responders, Week 44 | 10.0 | 0 | 9.5 | 14.3 | 0 | 25.0 | 40.0 | 0
  Clinical non-responders, Week 52: number analyzed (Participants) | 20 | 4 | 21 | 14 | 3 | 4 | 5 | 3
  Clinical non-responders, Week 52 | 0 | 0 | 14.3 | 7.1 | 0 | 25.0 | 40.0 | 33.3
Statistical Analysis 1: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 20; Test type: Superiority; p = 0.295, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = 20.0, 95% CI 2-sided [2.5 to 37.5] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 2: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 20; Test type: Superiority; p = 0.355, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = 13.8, 95% CI 2-sided [-7.4 to 34.9] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 3: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Responders, Week 20; Test type: Superiority; p = 0.384, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = -20.0, 95% CI 2-sided [-55.1 to 15.1] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 4: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 28; Test type: Superiority; p = 0.311, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = -22.5, 95% CI 2-sided [-59.5 to 14.5] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 5: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 28; Test type: Superiority; p = 0.422, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = -16.3, 95% CI 2-sided [-43.8 to 11.3] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 6: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Responders, Week 28; Test type: Superiority; p = 0.181, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = -25.0, 95% CI 2-sided [-59.2 to 9.2] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 7: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 36; Test type: Superiority; p = 0.281, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = 25.0, 95% CI 2-sided [6.0 to 44.0] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 8: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 36; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = 0.0, 95% CI 2-sided [-28.5 to 28.5] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 9: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Responders, Week 36; Test type: Superiority; p = 0.231, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = -25.0, 95% CI 2-sided [-61.3 to 11.3] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 10: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 44; Test type: Superiority; p = 0.214, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = 27.5, 95% CI 2-sided [-3.9 to 58.9] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 11: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 44; Test type: Superiority; p = 0.277, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = 21.3, 95% CI 2-sided [-7.5 to 50.0] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 12: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Responders, Week 44; Test type: Superiority; p = 0.442, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = -20.0, 95% CI 2-sided [-57.2 to 17.2] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 13: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 52; Test type: Superiority; p = 0.419, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = 20.0, 95% CI 2-sided [-17.1 to 57.1] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 14: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 52; Test type: Superiority; p = 0.214, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = 20.0, 95% CI 2-sided [-10.4 to 50.4] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 15: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Responders, Week 52; Test type: Superiority; p = 0.439, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = -15.0, 95% CI 2-sided [-52.4 to 22.4] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 16: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 20; Test type: Superiority; p = 0.284, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = 23.1, 95% CI 2-sided [-10.1 to 56.4] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 17: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 20; Test type: Superiority; p = 0.988, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = 0.2, 95% CI 2-sided [-23.9 to 24.3] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 18: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Non-responders, Week 20; Test type: Superiority; p = 0.370, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = -12.1, 95% CI 2-sided [-38.1 to 13.9] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 19: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 28; Test type: Superiority; p = 0.268, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = 25.6, 95% CI 2-sided [-8.9 to 60.2] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 20: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 28; Test type: Superiority; p = 0.665, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = -5.0, 95% CI 2-sided [-27.4 to 17.5] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 21: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Non-responders, Week 28; Test type: Superiority; p = 0.759, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = -3.9, 95% CI 2-sided [-28.9 to 21.0] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 22: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 36; Test type: Superiority; p = 0.259, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = 21.9, 95% CI 2-sided [-12.8 to 56.6] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 23: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 36; Test type: Superiority; p = 0.880, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = -1.7, 95% CI 2-sided [-23.2 to 19.9] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 24: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Non-responders, Week 36; Test type: Superiority; p = 0.355, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = -10.7, 95% CI 2-sided [-32.7 to 11.2] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 25: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 44; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = 5.0, 95% CI 2-sided [-27.1 to 37.1] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 26: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 44; Test type: Superiority; p = 0.688, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = 4.4, 95% CI 2-sided [-17.0 to 25.9] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 27: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Non-responders, Week 44; Test type: Superiority; p = 0.927, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = 1.1, 95% CI 2-sided [-22.3 to 24.5] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 28: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 52; Test type: Superiority; p = 0.075, Chi-squared — [p-value comment as in outcome 47, analysis 9]; Risk Difference (RD) = 27.5, 95% CI 2-sided [-5.0 to 60.0] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 29: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 52; Test type: Superiority; p = 0.154, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = 14.0, 95% CI 2-sided [-4.8 to 32.7] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 30: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Non-responders, Week 52; Test type: Superiority; p = 0.707, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = 4.9, 95% CI 2-sided [-14.4 to 24.2] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 31: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 20; Test type: Superiority; p = 0.085, Chi-squared — [p-value comment as in outcome 47, analysis 9]; Risk Difference (RD) = 25.0, 95% CI 2-sided [10.0 to 40.0] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 32: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 20; Test type: Superiority; p = 0.137, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = 14.7, 95% CI 2-sided [-4.0 to 33.3] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 33: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical responders, Week 20; Test type: Superiority; p = 0.370, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = -11.8, 95% CI 2-sided [-38.2 to 14.5] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 34: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 28; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = -3.6, 95% CI 2-sided [-31.6 to 24.4] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 35: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 28; Test type: Superiority; p = 0.174, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = -16.4, 95% CI 2-sided [-39.8 to 7.0] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 36: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical responders, Week 28; Test type: Superiority; p = 0.203, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = -17.1, 95% CI 2-sided [-43.9 to 9.7] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 37: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 36; Test type: Superiority; p = 0.286, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = 20.1, 95% CI 2-sided [-4.5 to 44.7] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 38: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 36; Test type: Superiority; p = 0.773, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = -3.6, 95% CI 2-sided [-27.7 to 20.6] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 39: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical responders, Week 36; Test type: Superiority; p = 0.101, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = -23.5, 95% CI 2-sided [-51.2 to 4.1] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 40: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 44; Test type: Superiority; p = 0.332, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = 15.2, 95% CI 2-sided [-14.1 to 44.4] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 41: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 44; Test type: Superiority; p = 0.189, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = 16.2, 95% CI 2-sided [-7.5 to 39.8] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 42: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical responders, Week 44; Test type: Superiority; p = 0.329, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = -14.1, 95% CI 2-sided [-42.2 to 13.9] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 43: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 52; Test type: Superiority; p = 0.124, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = 24.6, 95% CI 2-sided [-4.8 to 53.9] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 44: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 52; Test type: Superiority; p = 0.234, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = 15.2, 95% CI 2-sided [-9.5 to 39.9] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 45: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical responders, Week 52; Test type: Superiority; p = 0.484, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = -10.0, 95% CI 2-sided [-37.8 to 17.7] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 46: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 20; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = -10.0, 95% CI 2-sided [-57.3 to 37.3] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 47: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 20; Test type: Superiority; p = 0.431, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = -11.2, 95% CI 2-sided [-38.9 to 16.5] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 48: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 20; Test type: Superiority; p = 0.250, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = -20.7, 95% CI 2-sided [-48.5 to 7.1] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 49: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 28; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = 5.0, 95% CI 2-sided [-40.9 to 50.9] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 50: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 28; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = -1.0, 95% CI 2-sided [-25.2 to 23.3] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 51: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 28; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = -5.7, 95% CI 2-sided [-31.1 to 19.6] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 52: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 36; Test type: Superiority; p = 0.544, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = 10.0, 95% CI 2-sided [-35.2 to 55.2] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 53: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 36; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = -0.7, 95% CI 2-sided [-22.4 to 20.9] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 54: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 36; Test type: Superiority; p = 0.627, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = -7.9, 95% CI 2-sided [-28.5 to 12.8] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 55: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 44; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = -10.0, 95% CI 2-sided [-23.1 to 3.1] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 56: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 44; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = -0.5, 95% CI 2-sided [-18.7 to 17.7] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 57: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 44; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = 4.3, 95% CI 2-sided [-18.3 to 26.8] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 58: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 52; Test type: Superiority; p = 0.232, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = 14.3, 95% CI 2-sided [-0.7 to 29.3] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 59: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 52; Test type: Superiority; p = 0.412, Chi-squared — [p-value comment as in outcome 45, analysis 2]; Risk Difference (RD) = 7.1, 95% CI 2-sided [-6.3 to 20.6] — [estimate comment as in outcome 24, analysis 1]

49. Secondary Outcome: Change From Induction Baseline in Fecal Calprotectin Level Over Time During Extension Phase
Time Frame: Baseline, Week 28, Week 52
Population: Participants from ITT population with an assessment at given time point. Last observation carried forward.
Measure: Mean (Standard Deviation); unit: mcg/g
Arm/Group | Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction | Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction | Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction | Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction | Upadacitinib 3 mg BID in Extension/ Placebo in Induction | Upadacitinib 6 mg BID in Extension/ Placebo in Induction | Upadacitinib 12 mg BID in Extension/ Placebo in Induction | Upadacitinib 24 mg QD in Extension/ Placebo in Induction
Number analyzed (Participants) | 39 | 15 | 30 | 13 | 5 | 4 | 4 | 2
mcg/g
  Responders, Week 28: number analyzed (Participants) | 16 | 7 | 9 | 3 | 1 | 0 | 0 | 0
  Responders, Week 28 | -153.4 (2722.96) | -532.0 (519.42) | -2878.6 (2584.43) | -3563.7 (4747.26) | -194.0 (NA) — not applicable (1 participant in arm) |  |  |
  Responders, Week 52: number analyzed (Participants) | 16 | 7 | 10 | 4 | 1 | 0 | 0 | 0
  Responders, Week 52 | -51.9 (2650.98) | -524.1 (521.31) | -3047.5 (2509.27) | -2371.8 (2786.97) | -44.0 (NA) — not applicable (1 participant in arm) |  |  |
  Non-responders, Week 28: number analyzed (Participants) | 21 | 7 | 16 | 9 | 4 | 4 | 4 | 2
  Non-responders, Week 28 | -150.3 (958.76) | -148.3 (1315.46) | -834.5 (3011.51) | -850.2 (1821.34) | -16.5 (304.33) | -121.0 (395.16) | -326.8 (817.71) | 760.5 (1075.51)
  Non-responders, Week 52: number analyzed (Participants) | 23 | 8 | 20 | 9 | 4 | 4 | 4 | 2
  Non-responders, Week 52 | -87.2 (1494.35) | 88.3 (1689.67) | -704.0 (2801.08) | -562.8 (1738.58) | -8.3 (344.29) | -121.0 (395.16) | -434.0 (1030.64) | 760.5 (1075.51)
  Clinical responders, Week 28: number analyzed (Participants) | 25 | 11 | 16 | 9 | 4 | 1 | 2 | 0
  Clinical responders, Week 28 | -226.2 (2261.16) | -424.5 (1102.22) | -2794.6 (3018.26) | -2099.3 (3083.34) | -65.0 (316.06) | -694.0 (NA) — not applicable (1 participant in arm) | 117.5 (166.17) |
  Clinical responders, Week 52: number analyzed (Participants) | 26 | 12 | 18 | 10 | 4 | 1 | 2 | 0
  Clinical responders, Week 52 | 1.0 (2457.22) | -239.3 (1443.14) | -2617.4 (3232.04) | -1510.3 (2773.90) | -44.3 (350.61) | -694.0 (NA) — not applicable (1 participant in arm) | 117.5 (166.17) |
  Clinical non-responders, Week 28: number analyzed (Participants) | 12 | 3 | 9 | 3 | 1 | 3 | 2 | 2
  Clinical non-responders, Week 28 | 3.7 (766.69) | -30.7 (32.65) | 606.0 (1133.70) | 183.7 (443.97) | 0.0 (NA) — not applicable (1 participant in arm) | 70.0 (123.85) | -771.0 (1090.36) | 760.5 (1075.51)
  Clinical non-responders, Week 52: number analyzed (Participants) | 13 | 3 | 12 | 3 | 1 | 3 | 2 | 2
  Clinical non-responders, Week 52 | -220.2 (514.97) | -30.7 (32.65) | 213.3 (802.34) | 183.7 (443.97) | 0.0 (NA) — not applicable (1 participant in arm) | 70.0 (123.85) | -985.5 (1393.71) | 760.5 (1075.51)
Statistical Analysis 1: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 28; Test type: Superiority; p = 0.356, ANCOVA — P-value for test of difference between each upadacitinib higher dose and upadacitinib lower dose for mean change from induction baseline using analysis of covariance with treatment as factor and induction baseline value as covariate; LS Mean of Difference = -745.7, 95% CI 2-sided [-2369.73 to 878.37]
Statistical Analysis 2: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 28; Test type: Superiority; p = 0.158, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = -1119.5, 95% CI 2-sided [-2698.52 to 459.50]
Statistical Analysis 3: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Responders, Week 28; Test type: Superiority; p = 0.322, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = -1166.0, 95% CI 2-sided [-3531.30 to 1199.32]
Statistical Analysis 4: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 52; Test type: Superiority; p = 0.287, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = -828.2, 95% CI 2-sided [-2387.16 to 730.75]
Statistical Analysis 5: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 52; Test type: Superiority; p = 0.088, ANCOVA — [p-value comment as in outcome 49, analysis 1]; Prespecified statistically significant at 0.1 level; LS Mean of Difference = -1286.1, 95% CI 2-sided [-2772.59 to 200.43]
Statistical Analysis 6: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Responders, Week 52; Test type: Superiority; p = 0.613, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = -502.2, 95% CI 2-sided [-2505.74 to 1501.38]
Statistical Analysis 7: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 28; Test type: Superiority; p = 0.609, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = 283.4, 95% CI 2-sided [-823.64 to 1390.49]
Statistical Analysis 8: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 28; Test type: Superiority; p = 0.855, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = -78.2, 95% CI 2-sided [-930.47 to 774.16]
Statistical Analysis 9: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Non-responders, Week 28; Test type: Superiority; p = 0.584, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = 283.5, 95% CI 2-sided [-751.66 to 1318.57]
Statistical Analysis 10: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 52; Test type: Superiority; p = 0.624, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = 356.6, 95% CI 2-sided [-1095.03 to 1808.19]
Statistical Analysis 11: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 52; Test type: Superiority; p = 0.806, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = -135.1, 95% CI 2-sided [-1233.48 to 963.25]
Statistical Analysis 12: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Non-responders, Week 52; Test type: Superiority; p = 0.793, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = 186.2, 95% CI 2-sided [-1229.59 to 1602.06]
Statistical Analysis 13: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 28; Test type: Superiority; p = 0.561, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = -304.8, 95% CI 2-sided [-1350.04 to 740.44]
Statistical Analysis 14: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 28; Test type: Superiority; p = 0.024, ANCOVA — [p-value comment as in outcome 49, analysis 1]; Prespecified statistically significant at 0.05 level; LS Mean of Difference = -1119.0, 95% CI 2-sided [-2083.81 to -154.11]
Statistical Analysis 15: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical responders, Week 28; Test type: Superiority; p = 0.156, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = -819.3, 95% CI 2-sided [-1959.79 to 321.21]
Statistical Analysis 16: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 52; Test type: Superiority; p = 0.580, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = -346.6, 95% CI 2-sided [-1592.66 to 899.45]
Statistical Analysis 17: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 52; Test type: Superiority; p = 0.029, ANCOVA — [p-value comment as in outcome 49, analysis 1]; Prespecified statistically significant at 0.05 level; LS Mean of Difference = -1275.9, 95% CI 2-sided [-2415.88 to -135.92]
Statistical Analysis 18: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical responders, Week 52; Test type: Superiority; p = 0.431, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = -534.9, 95% CI 2-sided [-1883.23 to 813.50]
Statistical Analysis 19: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 28; Test type: Superiority; p = 0.965, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = -25.4, 95% CI 2-sided [-1200.67 to 1149.95]
Statistical Analysis 20: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 28; Test type: Superiority; p = 0.123, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = 623.6, 95% CI 2-sided [-183.52 to 1430.64]
Statistical Analysis 21: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 28; Test type: Superiority; p = 0.591, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = 368.2, 95% CI 2-sided [-1031.23 to 1767.60]
Statistical Analysis 22: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 52; Test type: Superiority; p = 0.642, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = 192.2, 95% CI 2-sided [-648.22 to 1032.68]
Statistical Analysis 23: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 52; Test type: Superiority; p = 0.093, ANCOVA — [p-value comment as in outcome 49, analysis 1]; Prespecified statistically significant at 0.1 level; LS Mean of Difference = 455.8, 95% CI 2-sided [-81.37 to 992.95]
Statistical Analysis 24: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 52; Test type: Superiority; p = 0.296, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = 463.6, 95% CI 2-sided [-428.99 to 1356.20]

50. Secondary Outcome: Change From Induction Baseline in Hs-CRP Over Time During Extension Phase
Time Frame: Baseline, Week 20, Week 28, Week 36, Week 44, Week 52
Population: Participants from ITT population with an assessment at given time point. Last observation carried forward.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction | Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction | Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction | Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction | Upadacitinib 3 mg BID in Extension/ Placebo in Induction | Upadacitinib 6 mg BID in Extension/ Placebo in Induction | Upadacitinib 12 mg BID in Extension/ Placebo in Induction | Upadacitinib 24 mg QD in Extension/ Placebo in Induction
Number analyzed (Participants) | 49 | 18 | 47 | 31 | 9 | 4 | 7 | 4
mg/L
  Responders, Week 20: number analyzed (Participants) | 19 | 8 | 16 | 9 | 1 | 0 | 0 | 0
  Responders, Week 20 | -9.5 (21.77) | -9.4 (11.14) | -20.8 (19.78) | 4.1 (36.50) | -3.1 (NA) — not applicable (1 participants analyzed) |  |  |
  Responders, Week 28: number analyzed (Participants) | 19 | 8 | 16 | 9 | 1 | 0 | 0 | 0
  Responders, Week 28 | -6.0 (22.53) | -3.6 (16.12) | -21.8 (17.93) | 7.0 (35.65) | -4.2 (NA) — not applicable (1 participants analyzed) |  |  |
  Responders, Week 36: number analyzed (Participants) | 19 | 8 | 16 | 9 | 1 | 0 | 0 | 0
  Responders, Week 36 | -1.8 (25.57) | -7.2 (10.86) | -22.5 (18.01) | 5.6 (35.87) | -4.0 (NA) — not applicable (1 participants analyzed) |  |  |
  Responders, Week 44: number analyzed (Participants) | 19 | 8 | 16 | 9 | 1 | 0 | 0 | 0
  Responders, Week 44 | -5.4 (22.95) | -8.5 (12.18) | -21.5 (19.78) | 5.8 (35.77) | 10.6 (NA) — not applicable (1 participants analyzed) |  |  |
  Responders, Week 52: number analyzed (Participants) | 19 | 8 | 16 | 9 | 1 | 0 | 0 | 0
  Responders, Week 52 | -4.3 (22.68) | -7.0 (12.66) | -20.4 (18.76) | 6.2 (35.82) | 0.4 (NA) — not applicable (1 participants analyzed) |  |  |
  Non-responders, Week 20: number analyzed (Participants) | 30 | 10 | 31 | 21 | 7 | 4 | 7 | 4
  Non-responders, Week 20 | -2.2 (9.72) | -1.6 (8.24) | -8.5 (25.00) | -8.0 (18.77) | 0.3 (10.89) | -1.0 (0.97) | -6.8 (8.82) | -1.5 (2.39)
  Non-responders, Week 28: number analyzed (Participants) | 30 | 10 | 31 | 22 | 8 | 4 | 7 | 4
  Non-responders, Week 28 | -3.0 (9.61) | -0.2 (5.92) | -6.4 (27.03) | -6.5 (20.14) | 0.3 (9.78) | -1.1 (1.06) | -5.9 (6.58) | 3.8 (9.55)
  Non-responders, Week 36: number analyzed (Participants) | 30 | 10 | 31 | 22 | 8 | 4 | 7 | 4
  Non-responders, Week 36 | -0.7 (8.86) | 5.2 (15.34) | -7.3 (24.87) | 0.8 (45.98) | 3.3 (8.88) | 0.5 (0.41) | -3.7 (7.80) | 8.3 (12.71)
  Non-responders, Week 44: number analyzed (Participants) | 30 | 10 | 31 | 22 | 8 | 4 | 7 | 4
  Non-responders, Week 44 | -1.3 (7.82) | 11.1 (33.68) | -4.1 (27.93) | 0.9 (45.88) | 3.0 (9.51) | -0.9 (0.87) | -4.1 (7.12) | 5.5 (9.39)
  Non-responders, Week 52: number analyzed (Participants) | 30 | 10 | 31 | 22 | 8 | 4 | 7 | 4
  Non-responders, Week 52 | -1.2 (8.67) | 2.8 (17.81) | -3.4 (32.58) | 1.3 (45.26) | 4.7 (11.50) | -0.2 (0.42) | -5.1 (8.52) | 2.5 (9.89)
  Clinical responders, Week 20: number analyzed (Participants) | 30 | 14 | 28 | 17 | 6 | 1 | 3 | 1
  Clinical responders, Week 20 | -7.1 (18.6) | -6.9 (10.80) | -18.0 (29.20) | -3.0 (31.35) | -3.8 (5.59) | -2.2 (NA) — not applicable (1 participants analyzed) | -9.5 (12.15) | -4.4 (NA) — not applicable (1 participants analyzed)
  Clinical responders, Week 28: number analyzed (Participants) | 30 | 14 | 28 | 17 | 6 | 1 | 3 | 1
  Clinical responders, Week 28 | -5.4 (19.26) | -2.0 (12.93) | -19.2 (30.13) | 0.0 (32.17) | -4.0 (4.77) | -2.3 (NA) — not applicable (1 participants analyzed) | -6.1 (6.32) | -5.3 (NA) — not applicable (1 participants analyzed)
  Clinical responders, Week 36: number analyzed (Participants) | 30 | 14 | 28 | 17 | 6 | 1 | 3 | 1
  Clinical responders, Week 36 | -0.8 (20.85) | -0.5 (16.69) | -18.6 (28.62) | 9.1 (56.33) | 0.1 (5.93) | 0.4 (NA) — not applicable (1 participants analyzed) | -3.2 (9.54) | -4.9 (NA) — not applicable (1 participants analyzed)
  Clinical responders, Week 44: number analyzed (Participants) | 30 | 14 | 28 | 17 | 6 | 1 | 3 | 1
  Clinical responders, Week 44 | -3.5 (18.87) | 3.0 (31.54) | -15.3 (32.75) | 9.3 (56.18) | 2.2 (7.92) | -1.5 (NA) — not applicable (1 participants analyzed) | -1.8 (7.26) | -3.9 (NA) — not applicable (1 participants analyzed)
  Clinical responders, Week 52: number analyzed (Participants) | 30 | 14 | 28 | 17 | 6 | 1 | 3 | 1
  Clinical responders, Week 52 | -2.8 (18.91) | -2.1 (18.36) | -13.9 (37.06) | 10.2 (55.66) | 2.7 (10.77) | -0.7 (NA) — not applicable (1 participants analyzed) | -4.2 (11.29) | -4.6 (NA) — not applicable (1 participants analyzed)
  Clinical non-responders, Week 20: number analyzed (Participants) | 19 | 4 | 19 | 13 | 2 | 3 | 4 | 3
  Clinical non-responders, Week 20 | -1.7 (10.51) | 1.4 (2.83) | -4.9 (8.36) | -6.2 (15.35) | 10.9 (15.47) | -0.6 (0.71) | -4.8 (6.69) | -0.5 (1.68)
  Clinical non-responders, Week 28: number analyzed (Participants) | 19 | 4 | 19 | 14 | 3 | 3 | 4 | 3
  Clinical non-responders, Week 28 | -2.2 (7.71) | -0.6 (1.43) | -0.6 (6.82) | -5.7 (15.26) | 7.3 (12.63) | -0.7 (0.81) | -5.8 (7.73) | 6.8 (9.10)
  Clinical non-responders, Week 36: number analyzed (Participants) | 19 | 4 | 19 | 14 | 3 | 3 | 4 | 3
  Clinical non-responders, Week 36 | -1.7 (8.94) | 0.4 (0.51) | -3.4 (8.04) | -6.1 (13.28) | 7.3 (12.63) | 0.6 (0.50) | -4.1 (7.77) | 12.7 (11.20)
  Clinical non-responders, Week 44: number analyzed (Participants) | 19 | 4 | 19 | 14 | 3 | 3 | 4 | 3
  Clinical non-responders, Week 44 | -1.9 (7.83) | 0.4 (0.51) | -2.3 (9.37) | -6.2 (13.15) | 7.3 (12.63) | -0.7 (0.95) | -5.8 (7.55) | 8.6 (8.55)
  Clinical non-responders, Week 52: number analyzed (Participants) | 19 | 4 | 19 | 14 | 3 | 3 | 4 | 3
  Clinical non-responders, Week 52 | -1.9 (8.11) | 0.4 (0.51) | -2.2 (9.28) | -6.3 (11.71) | 7.3 (12.63) | 0.0 (0.33) | -5.8 (7.66) | 4.9 (10.60)
Statistical Analysis 1: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 20; Test type: Superiority; p = 0.822, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = -2.0, 95% CI 2-sided [-19.83 to 15.83]
Statistical Analysis 2: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 20; Test type: Superiority; p = 0.386, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = -6.4, 95% CI 2-sided [-20.97 to 8.25]
Statistical Analysis 3: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Responders, Week 20; Test type: Superiority; p = 0.136, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = 12.9, 95% CI 2-sided [-4.22 to 29.95]
Statistical Analysis 4: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 28; Test type: Superiority; p = 0.912, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = 1.0, 95% CI 2-sided [-17.87 to 19.97]
Statistical Analysis 5: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 28; Test type: Superiority; p = 0.118, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = -12.3, 95% CI 2-sided [-27.77 to 3.25]
Statistical Analysis 6: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Responders, Week 28; Test type: Superiority; p = 0.171, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = 12.5, 95% CI 2-sided [-5.61 to 30.65]
Statistical Analysis 7: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 36; Test type: Superiority; p = 0.479, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = -6.9, 95% CI 2-sided [-26.50 to 12.63]
Statistical Analysis 8: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 36; Test type: Superiority; p = 0.037, ANCOVA — [p-value comment as in outcome 49, analysis 1]; Prespecified statistically significant at 0.05 level; LS Mean of Difference = -17.1, 95% CI 2-sided [-33.12 to -1.04]
Statistical Analysis 9: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Responders, Week 36; Test type: Superiority; p = 0.463, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = 6.9, 95% CI 2-sided [-11.86 to 25.65]
Statistical Analysis 10: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 44; Test type: Superiority; p = 0.627, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = -4.6, 95% CI 2-sided [-23.59 to 14.37]
Statistical Analysis 11: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 44; Test type: Superiority; p = 0.122, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = -12.2, 95% CI 2-sided [-27.75 to 3.37]
Statistical Analysis 12: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Responders, Week 44; Test type: Superiority; p = 0.243, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = 10.7, 95% CI 2-sided [-7.49 to 28.89]
Statistical Analysis 13: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 52; Test type: Superiority; p = 0.658, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = -4.2, 95% CI 2-sided [-22.95 to 14.63]
Statistical Analysis 14: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Responders, Week 52; Test type: Superiority; p = 0.115, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = -12.3, 95% CI 2-sided [-27.69 to 3.12]
Statistical Analysis 15: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Responders, Week 52; Test type: Superiority; p = 0.267, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = 10.0, 95% CI 2-sided [-7.96 to 28.06]
Statistical Analysis 16: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 20; Test type: Superiority; p = 0.974, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = 0.2, 95% CI 2-sided [-9.74 to 10.06]
Statistical Analysis 17: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 20; Test type: Superiority; p = 0.882, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = -0.5, 95% CI 2-sided [-7.61 to 6.55]
Statistical Analysis 18: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Non-responders, Week 20; Test type: Superiority; p = 0.982, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = -0.1, 95% CI 2-sided [-7.92 to 7.75]
Statistical Analysis 19: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 28; Test type: Superiority; p = 0.673, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = 2.2, 95% CI 2-sided [-8.11 to 12.51]
Statistical Analysis 20: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 28; Test type: Superiority; p = 0.467, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = 2.7, 95% CI 2-sided [-4.64 to 10.04]
Statistical Analysis 21: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Non-responders, Week 28; Test type: Superiority; p = 0.583, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = 2.2, 95% CI 2-sided [-5.79 to 10.23]
Statistical Analysis 22: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 36; Test type: Superiority; p = 0.564, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = 5.5, 95% CI 2-sided [-13.33 to 24.31]
Statistical Analysis 23: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 36; Test type: Superiority; p = 0.728, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = -2.4, 95% CI 2-sided [-15.74 to 11.04]
Statistical Analysis 24: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Non-responders, Week 36; Test type: Superiority; p = 0.460, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = 5.5, 95% CI 2-sided [-9.16 to 20.08]
Statistical Analysis 25: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 44; Test type: Superiority; p = 0.253, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = 12.0, 95% CI 2-sided [-8.72 to 32.75]
Statistical Analysis 26: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 44; Test type: Superiority; p = 0.884, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = 1.1, 95% CI 2-sided [-13.67 to 15.84]
Statistical Analysis 27: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Non-responders, Week 44; Test type: Superiority; p = 0.474, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = 5.8, 95% CI 2-sided [-10.28 to 21.95]
Statistical Analysis 28: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 52; Test type: Superiority; p = 0.727, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = 3.6, 95% CI 2-sided [-17.03 to 24.30]
Statistical Analysis 29: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Non-responders, Week 52; Test type: Superiority; p = 0.780, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = 2.1, 95% CI 2-sided [-12.63 to 16.78]
Statistical Analysis 30: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Non-responders, Week 52; Test type: Superiority; p = 0.424, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = 6.5, 95% CI 2-sided [-9.57 to 22.54]
Statistical Analysis 31: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 20; Test type: Superiority; p = 0.841, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = -1.3, 95% CI 2-sided [-14.23 to 11.62]
Statistical Analysis 32: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 20; Test type: Superiority; p = 0.702, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = -2.1, 95% CI 2-sided [-12.94 to 8.75]
Statistical Analysis 33: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical responders, Week 20; Test type: Superiority; p = 0.353, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = 5.7, 95% CI 2-sided [-6.43 to 17.83]
Statistical Analysis 34: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 28; Test type: Superiority; p = 0.770, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = 2.1, 95% CI 2-sided [-11.89 to 16.00]
Statistical Analysis 35: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 28; Test type: Superiority; p = 0.367, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = -5.3, 95% CI 2-sided [-17.04 to 6.37]
Statistical Analysis 36: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical responders, Week 28; Test type: Superiority; p = 0.291, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = 7.0, 95% CI 2-sided [-6.09 to 20.07]
Statistical Analysis 37: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 36; Test type: Superiority; p = 0.942, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = -0.7, 95% CI 2-sided [-20.87 to 19.40]
Statistical Analysis 38: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 36; Test type: Superiority; p = 0.162, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = -12.0, 95% CI 2-sided [-28.89 to 4.91]
Statistical Analysis 39: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical responders, Week 36; Test type: Superiority; p = 0.253, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = 10.9, 95% CI 2-sided [-7.96 to 29.82]
Statistical Analysis 40: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 44; Test type: Superiority; p = 0.617, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = 5.5, 95% CI 2-sided [-16.25 to 27.21]
Statistical Analysis 41: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 44; Test type: Superiority; p = 0.515, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = -6.0, 95% CI 2-sided [-24.22 to 12.24]
Statistical Analysis 42: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical responders, Week 44; Test type: Superiority; p = 0.180, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = 13.8, 95% CI 2-sided [-6.53 to 34.23]
Statistical Analysis 43: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 52; Test type: Superiority; p = 0.972, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = -0.4, 95% CI 2-sided [-21.86 to 21.09]
Statistical Analysis 44: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical responders, Week 52; Test type: Superiority; p = 0.589, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = -4.9, 95% CI 2-sided [-22.94 to 13.10]
Statistical Analysis 45: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical responders, Week 52; Test type: Superiority; p = 0.168, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = 14.1, 95% CI 2-sided [-6.07 to 34.22]
Statistical Analysis 46: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 20; Test type: Superiority; p = 0.712, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = 1.9, 95% CI 2-sided [-8.50 to 12.36]
Statistical Analysis 47: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 20; Test type: Superiority; p = 0.465, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = -2.3, 95% CI 2-sided [-8.41 to 3.90]
Statistical Analysis 48: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 20; Test type: Superiority; p = 0.924, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = 0.3, 95% CI 2-sided [-6.83 to 7.52]
Statistical Analysis 49: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 28; Test type: Superiority; p = 0.938, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = 0.4, 95% CI 2-sided [-8.88 to 9.60]
Statistical Analysis 50: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 28; Test type: Superiority; p = 0.410, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = 2.2, 95% CI 2-sided [-3.17 to 7.64]
Statistical Analysis 51: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 28; Test type: Superiority; p = 0.941, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = 0.2, 95% CI 2-sided [-5.89 to 6.35]
Statistical Analysis 52: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 36; Test type: Superiority; p = 0.872, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = 0.7, 95% CI 2-sided [-8.23 to 9.67]
Statistical Analysis 53: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 36; Test type: Superiority; p = 0.692, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = -1.0, 95% CI 2-sided [-6.27 to 4.20]
Statistical Analysis 54: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 36; Test type: Superiority; p = 0.896, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = -0.4, 95% CI 2-sided [-6.32 to 5.54]
Statistical Analysis 55: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 44; Test type: Superiority; p = 0.826, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = 1.0, 95% CI 2-sided [-7.92 to 9.87]
Statistical Analysis 56: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 44; Test type: Superiority; p = 0.885, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = 0.4, 95% CI 2-sided [-4.82 to 5.58]
Statistical Analysis 57: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 44; Test type: Superiority; p = 0.964, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = -0.1, 95% CI 2-sided [-6.03 to 5.76]
Statistical Analysis 58: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 52; Test type: Superiority; p = 0.806, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = 1.1, 95% CI 2-sided [-7.59 to 9.72]
Statistical Analysis 59: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 52; Test type: Superiority; p = 0.871, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = 0.4, 95% CI 2-sided [-4.65 to 5.47]
Statistical Analysis 60: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical non-responders, Week 52; Test type: Superiority; p = 0.850, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = -0.5, 95% CI 2-sided [-6.28 to 5.19]

51. Secondary Outcome: Change From Induction Baseline in IBDQ at Week 52
Description: The IBDQ is a disease-specific instrument composed of 32 Likert-scaled items. The total score ranges from 32 to 224 using the 7-point response options, with higher scores indicating better health-related quality of life. The IBDQ scale contains 4 component subscales: bowel symptoms, systemic symptoms, emotional function, and social function. Each subscale can be computed with total scores ranging from 10 to 70, 5 to 35, 12 to 84, and 5 to 35, respectively.
Time Frame: Baseline, Week 52
Population: Participants from ITT population with an assessment at given time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction | Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction | Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction | Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction | Upadacitinib 3 mg BID in Extension/ Placebo in Induction | Upadacitinib 6 mg BID in Extension/ Placebo in Induction | Upadacitinib 12 mg BID in Extension/ Placebo in Induction | Upadacitinib 24 mg QD in Extension/ Placebo in Induction
Number analyzed (Participants) | 36 | 15 | 38 | 22 | 7 | 4 | 5 | 2
units on a scale
  Responders: number analyzed (Participants) | 14 | 8 | 14 | 7 | 1 | 0 | 0 | 0
  Responders | 43.9 (38.06) | 56.4 (14.52) | 82.3 (35.59) | 45.3 (49.89) | -5.0 (NA) — not applicable (1 participant analyzed) |  |  |
  Non-responders: number analyzed (Participants) | 22 | 7 | 24 | 15 | 6 | 4 | 5 | 2
  Non-responders | 20.8 (43.58) | 26.0 (33.14) | 25.9 (47.05) | 2.9 (35.25) | 4.8 (16.42) | 35.5 (28.78) | 45.4 (36.16) | 41.5 (24.75)
  Clinical responders: number analyzed (Participants) | 22 | 13 | 23 | 14 | 5 | 1 | 2 | 1
  Clinical responders | 42.8 (44.13) | 46.6 (27.76) | 70.7 (46.99) | 26.6 (53.11) | 4.8 (18.70) | 68.0 (NA) — not applicable (1 participant analyzed) | 34.5 (4.95) | 24.0 (NA) — not applicable (1 participant analyzed)
  Clinical non-responders: number analyzed (Participants) | 14 | 2 | 15 | 8 | 2 | 3 | 3 | 1
  Clinical non-responders | 9.4 (31.46) | 13.5 (19.09) | 9.8 (30.81) | -1.5 (5.81) | 0.0 (0.00) | 24.6 (23.17) | 52.7 (49.03) | 59.0 (NA) — not applicable (1 participant analyzed)
Statistical Analysis 1: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Responders; Test type: Superiority; p = 0.792, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = -3.9, 95% CI 2-sided [-33.73 to 25.90]
Statistical Analysis 2: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Responders; Test type: Superiority; p = 0.179, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = 18.1, 95% CI 2-sided [-8.62 to 44.75]
Statistical Analysis 3: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Responders; Test type: Superiority; p = 0.230, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = -19.1, 95% CI 2-sided [-50.87 to 12.63]
Statistical Analysis 4: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Non-responders; Test type: Superiority; p = 0.337, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = 16.4, 95% CI 2-sided [-17.54 to 50.40]
Statistical Analysis 5: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Non-responders; Test type: Superiority; p = 0.924, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = 1.1, 95% CI 2-sided [-21.75 to 23.93]
Statistical Analysis 6: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Non-responders; Test type: Superiority; p = 0.373, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = -11.7, 95% CI 2-sided [-37.69 to 14.35]
Statistical Analysis 7: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical responders; Test type: Superiority; p = 0.813, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = -3.1, 95% CI 2-sided [-28.94 to 22.79]
Statistical Analysis 8: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical responders; Test type: Superiority; p = 0.651, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = 5.3, 95% CI 2-sided [-18.02 to 28.65]
Statistical Analysis 9: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical responders; Test type: Superiority; p = 0.065, ANCOVA — [p-value comment as in outcome 49, analysis 1]; Prespecified statistically significant at 0.1 level; LS Mean of Difference = -23.8, 95% CI 2-sided [-49.12 to 1.49]
Statistical Analysis 10: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical non-responders; Test type: Superiority; p = 0.802, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = 5.3, 95% CI 2-sided [-37.61 to 48.28]
Statistical Analysis 11: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical non-responders; Test type: Superiority; p = 0.955, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = 0.6, 95% CI 2-sided [-20.46 to 21.63]
Statistical Analysis 12: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical non-responders; Test type: Superiority; p = 0.395, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = -10.6, 95% CI 2-sided [-35.73 to 14.47]

52. Secondary Outcome: Change From Induction Baseline in European Quality of Life (EuroQol) 5 Dimensions Questionnaire (EQ-5D) Index Score at Week 52
Description: The EQ-5D is a standardized instrument for use as a measure of health-related quality of life. The EQ-5D Index Score has five dimensions of health (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). Health states are converted into a weighted health state index. These weights lie on a scale on which full health has a value of 1 and dead has a value of 0. A positive change represents an improvement in health-related quality of life.
Time Frame: Baseline, Week 52
Population: Participants from ITT population with an assessment at given time point. Observed cases.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction | Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction | Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction | Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction | Upadacitinib 3 mg BID in Extension/ Placebo in Induction | Upadacitinib 6 mg BID in Extension/ Placebo in Induction | Upadacitinib 12 mg BID in Extension/ Placebo in Induction | Upadacitinib 24 mg QD in Extension/ Placebo in Induction
Number analyzed (Participants) | 36 | 15 | 38 | 22 | 7 | 4 | 6 | 3
units on a scale
  Responders: number analyzed (Participants) | 14 | 8 | 14 | 7 | 1 | 0 | 0 | 0
  Responders | 0.1350 (0.1473) | 0.1673 (0.1090) | 0.2274 (0.1524) | 0.0122 (0.1276) | 0.3260 (NA) — not applicable (1 participant was analyzed) |  |  |
  Non-responders: number analyzed (Participants) | 22 | 7 | 24 | 15 | 6 | 4 | 6 | 3
  Non-responders | 0.0208 (0.2231) | 0.0697 (0.2091) | 0.1090 (0.1791) | 0.0449 (0.1008) | 0.1288 (0.1674) | 0.1125 (0.2210) | 0.1542 (0.2377) | 0.1187 (0.1128)
  Clinical responders: number analyzed (Participants) | 22 | 13 | 23 | 14 | 5 | 1 | 3 | 1
  Clinical responders | 0.1435 (0.1461) | 0.1334 (0.1740) | 0.2306 (0.1840) | 0.0587 (0.1298) | 0.2198 (0.1615) | 0.4325 (NA) — not applicable (1 participant was analyzed) | 0.1758 (0.3559) | 0.1316 (NA) — not applicable (1 participant was analyzed)
  Clinical non-responders: number analyzed (Participants) | 14 | 2 | 15 | 8 | 2 | 3 | 3 | 2
  Clinical non-responders | -0.0577 (0.2225) | 0.0455 (0.0643) | 0.0330 (0.0677) | -0.0079 (0.0228) | 0.0000 (0.0000) | 0.0058 (0.0708) | 0.1325 (0.1148) | 0.1122 (0.1587)
Statistical Analysis 1: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Responders; Test type: Superiority; p = 0.893, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = -0.0082, 95% CI 2-sided [-0.1299 to 0.1136]
Statistical Analysis 2: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Responders; Test type: Superiority; p = 0.182, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = 0.0685, 95% CI 2-sided [-0.0334 to 0.1705]
Statistical Analysis 3: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Responders; Test type: Superiority; p = 0.036, ANCOVA — [p-value comment as in outcome 49, analysis 1]; Prespecified statistically significant at 0.05 level; LS Mean of Difference = -0.1323, 95% CI 2-sided [-0.2552 to -0.0093]
Statistical Analysis 4: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Non-responders; Test type: Superiority; p = 0.316, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = 0.0768, 95% CI 2-sided [-0.0749 to 0.2286]
Statistical Analysis 5: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Non-responders; Test type: Superiority; p = 0.277, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = 0.0573, 95% CI 2-sided [-0.0471 to 0.1617]
Statistical Analysis 6: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Non-responders; Test type: Superiority; p = 0.467, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = 0.0428, 95% CI 2-sided [-0.0741 to 0.1597]
Statistical Analysis 7: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical responders; Test type: Superiority; p = 0.464, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = -0.0360, 95% CI 2-sided [-0.1336 to 0.0616]
Statistical Analysis 8: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical responders; Test type: Superiority; p = 0.345, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = 0.0404, 95% CI 2-sided [-0.0444 to 0.1252]
Statistical Analysis 9: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical responders; Test type: Superiority; p = 0.071, ANCOVA — [p-value comment as in outcome 49, analysis 1]; Prespecified statistically significant at 0.1 level; LS Mean of Difference = -0.0873, 95% CI 2-sided [-0.1822 to 0.0076]
Statistical Analysis 10: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical non-responders; Test type: Superiority; p = 0.317, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = 0.1109, 95% CI 2-sided [-0.1109 to 0.3326]
Statistical Analysis 11: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical non-responders; Test type: Superiority; p = 0.125, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = 0.0848, 95% CI 2-sided [-0.0248 to 0.1945]
Statistical Analysis 12: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical non-responders; Test type: Superiority; p = 0.390, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = 0.0559, 95% CI 2-sided [-0.0745 to 0.1864]

53. Secondary Outcome: Change From Induction Baseline in EQ-5D VAS at Week 52
Description: The EQ-5D is a standardized instrument for use as a measure of health-related quality of life. The EQ-5D VAS is a 20-cm scale with endpoints labeled "best imaginable health" and "worst imaginable health" anchored at 100 and 0, respectively. A positive change represents an improvement in health-related quality of life.
Time Frame: Baseline, Week 52
Population: Participants from ITT population with an assessment at given time point. Observed cases.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction | Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction | Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction | Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction | Upadacitinib 3 mg BID in Extension/ Placebo in Induction | Upadacitinib 6 mg BID in Extension/ Placebo in Induction | Upadacitinib 12 mg BID in Extension/ Placebo in Induction | Upadacitinib 24 mg QD in Extension/ Placebo in Induction
Number analyzed (Participants) | 36 | 15 | 37 | 22 | 7 | 4 | 6 | 3
units on a scale
  Responders: number analyzed (Participants) | 14 | 8 | 14 | 7 | 1 | 0 | 0 | 0
  Responders | 12.9 (14.65) | 26.9 (12.80) | 34.8 (22.55) | 5.0 (17.80) | 5.0 (NA) — not applicable (1 participant was analyzed) |  |  |
  Non-responders: number analyzed (Participants) | 22 | 7 | 23 | 15 | 6 | 4 | 6 | 3
  Non-responders | 12.3 (24.79) | 11.9 (18.73) | 13.9 (27.81) | 4.7 (14.22) | 12.2 (16.01) | 17.5 (16.58) | 20.3 (21.23) | 0.0 (15.00)
  Clinical responders: number analyzed (Participants) | 22 | 13 | 22 | 14 | 5 | 1 | 3 | 1
  Clinical responders | 18.2 (19.19) | 22.2 (17.16) | 36.1 (26.19) | 8.1 (17.95) | 15.6 (15.63) | 40.0 (NA) — not applicable (1 participant was analyzed) | 11.7 (16.07) | -15.0 (NA) — not applicable (1 participant was analyzed)
  Clinical non-responders: number analyzed (Participants) | 14 | 2 | 15 | 8 | 2 | 3 | 3 | 2
  Clinical non-responders | 3.7 (21.79) | 5.0 (7.07) | 0.8 (11.72) | -1.0 (4.24) | 0.0 (0.00) | 10.0 (8.66) | 29.0 (25.36) | 7.5 (10.61)
Statistical Analysis 1: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Responders; Test type: Superiority; p = 0.263, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = 8.7, 95% CI 2-sided [-6.79 to 24.16]
Statistical Analysis 2: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Responders; Test type: Superiority; p = 0.031, ANCOVA — [p-value comment as in outcome 49, analysis 1]; Prespecified statistically significant at 0.05 level; LS Mean of Difference = 15.2, 95% CI 2-sided [1.47 to 28.93]
Statistical Analysis 3: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Responders; Test type: Superiority; p = 0.135, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = -12.0, 95% CI 2-sided [-27.93 to 3.90]
Statistical Analysis 4: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Non-responders; Test type: Superiority; p = 0.458, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = 6.3, 95% CI 2-sided [-10.61 to 23.27]
Statistical Analysis 5: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Non-responders; Test type: Superiority; p = 0.738, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = 1.9, 95% CI 2-sided [-9.59 to 13.45]
Statistical Analysis 6: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Non-responders; Test type: Superiority; p = 0.412, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = -5.4, 95% CI 2-sided [-18.32 to 7.60]
Statistical Analysis 7: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical responders; Test type: Superiority; p = 0.534, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = 3.9, 95% CI 2-sided [-8.56 to 16.36]
Statistical Analysis 8: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical responders; Test type: Superiority; p = 0.052, ANCOVA — [p-value comment as in outcome 49, analysis 1]; Prespecified statistically significant at 0.1 level; LS Mean of Difference = 11.0, 95% CI 2-sided [-0.10 to 22.01]
Statistical Analysis 9: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical responders; Test type: Superiority; p = 0.027, ANCOVA — [p-value comment as in outcome 49, analysis 1]; Prespecified statistically significant at 0.05 level; LS Mean of Difference = -13.9, 95% CI 2-sided [-26.15 to -1.63]
Statistical Analysis 10: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical non-responders; Test type: Superiority; p = 0.928, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = -1.0, 95% CI 2-sided [-24.02 to 21.97]
Statistical Analysis 11: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical non-responders; Test type: Superiority; p = 0.658, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = -2.5, 95% CI 2-sided [-13.72 to 8.77]
Statistical Analysis 12: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical non-responders; Test type: Superiority; p = 0.601, ANCOVA — [p-value comment as in outcome 49, analysis 1]; LS Mean of Difference = -3.5, 95% CI 2-sided [-16.96 to 9.96]

54. Secondary Outcome: Cross Tabulation of Induction Baseline and Week 52 in Total Number of Extra-Intestinal Manifestations (EIMs) of Crohn's Disease
Description: Presented as percentage of participants with given number of EIMs at Baseline (BL) and Week (Wk) 52. EIMs of Crohn's disease included anemia, autoimmune hepatitis, axial arthropathy, bronchiectasis, chronic obstructive pulmonary disease, episcleritis, erythema nodosum, iritis, nephrolithiasis, oral aphthous ulcers, peripheral arthropathy, primary sclerosing cholangitis, pyoderma gangrenosum, Sweet's syndrome, uveitis, and venous thromboembolism.
Time Frame: Baseline, Week 52
Population: Participants from modified ITT population (all randomized participants who took at least 1 dose of study drug in the Induction Period).
Measure: Number; unit: percentage of participants
Groups:
- Double Blind Induction Phase: 12 mg BID: Upadacitinib 12 mg BID during the 16-week double-blind Induction Phase.
- Double Blind Induction Phase: 24 mg BID: Upadacitinib 24 mg BID during the 16-week double-blind Induction Phase.
- Double Blind Induction Phase: 24 mg QD: Upadacitinib 24 mg QD during the 16-week double-blind Induction Phase.
Arm/Group | Double-Blind Induction Phase: Placebo BID | Double-Blind Induction Phase: Upadacitinib 3 mg BID | Double-Blind Induction Phase: Upadacitinib 6 mg BID | Double Blind Induction Phase: 12 mg BID | Double Blind Induction Phase: 24 mg BID | Double Blind Induction Phase: 24 mg QD
Number analyzed (Participants) | 37 | 39 | 37 | 36 | 36 | 35
percentage of participants
  0 at BL/0 at Wk 52: number analyzed (Participants) | 14 | 13 | 22 | 25 | 15 | 20
  0 at BL/0 at Wk 52 | 85.7 | 100 | 86.4 | 76.0 | 73.3 | 85.0
  0 at BL/1 at Wk 52: number analyzed (Participants) | 14 | 13 | 22 | 25 | 15 | 20
  0 at BL/1 at Wk 52 | 7.1 | 0 | 9.1 | 16.0 | 13.3 | 10.0
  0 at BL/2 at Wk 52: number analyzed (Participants) | 14 | 13 | 22 | 25 | 15 | 20
  0 at BL/2 at Wk 52 | 0 | 0 | 0 | 0 | 0 | 0
  0 at BL/3 at Wk 52: number analyzed (Participants) | 14 | 13 | 22 | 25 | 15 | 20
  0 at BL/3 at Wk 52 | 0 | 0 | 0 | 0 | 0 | 0
  0 at BL/4 at Wk 52: number analyzed (Participants) | 14 | 13 | 22 | 25 | 15 | 20
  0 at BL/4 at Wk 52 | 0 | 0 | 0 | 0 | 0 | 0
  0 at BL/5 at Wk 52: number analyzed (Participants) | 14 | 13 | 22 | 25 | 15 | 20
  0 at BL/5 at Wk 52 | 0 | 0 | 0 | 0 | 0 | 0
  0 at BL/missing at Wk 52: number analyzed (Participants) | 14 | 13 | 22 | 25 | 15 | 20
  0 at BL/missing at Wk 52 | 7.1 | 0 | 4.5 | 8.0 | 13.3 | 5.0
  1 at BL/0 at Wk 52: number analyzed (Participants) | 14 | 19 | 10 | 8 | 18 | 11
  1 at BL/0 at Wk 52 | 42.9 | 31.6 | 40.0 | 62.5 | 50.0 | 54.5
  1 at BL/1 at Wk 52: number analyzed (Participants) | 14 | 19 | 10 | 8 | 18 | 11
  1 at BL/1 at Wk 52 | 50.0 | 57.9 | 60.0 | 12.5 | 33.3 | 36.4
  1 at BL/2 at Wk 52: number analyzed (Participants) | 14 | 19 | 10 | 8 | 18 | 11
  1 at BL/2 at Wk 52 | 7.1 | 5.3 | 0 | 25.0 | 11.1 | 9.1
  1 at BL/3 at Wk 52: number analyzed (Participants) | 14 | 19 | 10 | 8 | 18 | 11
  1 at BL/3 at Wk 52 | 0 | 0 | 0 | 0 | 0 | 0
  1 at BL/4 at Wk 52: number analyzed (Participants) | 14 | 19 | 10 | 8 | 18 | 11
  1 at BL/4 at Wk 52 | 0 | 0 | 0 | 0 | 0 | 0
  1 at BL/5 at Wk 52: number analyzed (Participants) | 14 | 19 | 10 | 8 | 18 | 11
  1 at BL/5 at Wk 52 | 0 | 0 | 0 | 0 | 0 | 0
  1 at BL/missing at Wk 52: number analyzed (Participants) | 14 | 19 | 10 | 8 | 18 | 11
  1 at BL/missing at Wk 52 | 0 | 5.3 | 0 | 0 | 5.6 | 0
  2 at BL/0 at Wk 52: number analyzed (Participants) | 5 | 4 | 3 | 3 | 0 | 4
  2 at BL/0 at Wk 52 | 20.0 | 50.0 | 0 | 33.3 |  | 25.0
  2 at BL/1 at Wk 52: number analyzed (Participants) | 5 | 4 | 3 | 3 | 0 | 4
  2 at BL/1 at Wk 52 | 0 | 25.0 | 66.7 | 33.3 |  | 25.0
  2 at BL/2 at Wk 52: number analyzed (Participants) | 5 | 4 | 3 | 3 | 0 | 4
  2 at BL/2 at Wk 52 | 60.0 | 25.0 | 33.3 | 33.3 |  | 50.0
  2 at BL/3 at Wk 52: number analyzed (Participants) | 5 | 4 | 3 | 3 | 0 | 4
  2 at BL/3 at Wk 52 | 0 | 0 | 0 | 0 |  | 0
  2 at BL/4 at Wk 52: number analyzed (Participants) | 5 | 4 | 3 | 3 | 0 | 4
  2 at BL/4 at Wk 52 | 0 | 0 | 0 | 0 |  | 0
  2 at BL/5 at Wk 52: number analyzed (Participants) | 5 | 4 | 3 | 3 | 0 | 4
  2 at BL/5 at Wk 52 | 0 | 0 | 0 | 0 |  | 0
  2 at BL/missing at Wk 52: number analyzed (Participants) | 5 | 4 | 3 | 3 | 0 | 4
  2 at BL/missing at Wk 52 | 20.0 | 0 | 0 | 0 |  | 0
  3 at BL/0 at Wk 52: number analyzed (Participants) | 2 | 2 | 1 | 0 | 3 | 0
  3 at BL/0 at Wk 52 | 0 | 50.0 | 0 |  | 66.7 |
  3 at BL/1 at Wk 52: number analyzed (Participants) | 2 | 2 | 1 | 0 | 3 | 0
  3 at BL/1 at Wk 52 | 50.0 | 50.0 | 0 |  | 0 |
  3 at BL/2 at Wk 52: number analyzed (Participants) | 2 | 2 | 1 | 0 | 3 | 0
  3 at BL/2 at Wk 52 | 0 | 0 | 100 |  | 33.3 |
  3 at BL/3 at Wk 52: number analyzed (Participants) | 2 | 2 | 1 | 0 | 3 | 0
  3 at BL/3 at Wk 52 | 0 | 0 | 0 |  | 0 |
  3 at BL/4 at Wk 52: number analyzed (Participants) | 2 | 2 | 1 | 0 | 3 | 0
  3 at BL/4 at Wk 52 | 50.0 | 0 | 0 |  | 0 |
  3 at BL/5 at Wk 52: number analyzed (Participants) | 2 | 2 | 1 | 0 | 3 | 0
  3 at BL/5 at Wk 52 | 0 | 0 | 0 |  | 0 |
  3 at BL/missing at Wk 52: number analyzed (Participants) | 2 | 2 | 1 | 0 | 3 | 0
  3 at BL/missing at Wk 52 | 0 | 0 | 0 |  | 0 |
  4 at BL/0 at Wk 52: number analyzed (Participants) | 1 | 1 | 1 | 0 | 0 | 0
  4 at BL/0 at Wk 52 | 0 | 100 | 0 |  |  |
  4 at BL/1 at Wk 52: number analyzed (Participants) | 1 | 1 | 1 | 0 | 0 | 0
  4 at BL/1 at Wk 52 | 0 | 0 | 0 |  |  |
  4 at BL/2 at Wk 52: number analyzed (Participants) | 1 | 1 | 1 | 0 | 0 | 0
  4 at BL/2 at Wk 52 | 0 | 0 | 0 |  |  |
  4 at BL/3 at Wk 52: number analyzed (Participants) | 1 | 1 | 1 | 0 | 0 | 0
  4 at BL/3 at Wk 52 | 0 | 0 | 0 |  |  |
  4 at BL/4 at Wk 52: number analyzed (Participants) | 1 | 1 | 1 | 0 | 0 | 0
  4 at BL/4 at Wk 52 | 100 | 0 | 0 |  |  |
  4 at BL/5 at Wk 52: number analyzed (Participants) | 1 | 1 | 1 | 0 | 0 | 0
  4 at BL/5 at Wk 52 | 0 | 0 | 0 |  |  |
  4 at BL/missing at Wk 52: number analyzed (Participants) | 1 | 1 | 1 | 0 | 0 | 0
  4 at BL/missing at Wk 52 | 0 | 0 | 100 |  |  |
  5 at BL/0 at Wk 52: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0
  5 at BL/0 at Wk 52 | 0 |  |  |  |  |
  5 at BL/1 at Wk 52: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0
  5 at BL/1 at Wk 52 | 0 |  |  |  |  |
  5 at BL/2 at Wk 52: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0
  5 at BL/2 at Wk 52 | 0 |  |  |  |  |
  5 at BL/3 at Wk 52: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0
  5 at BL/3 at Wk 52 | 0 |  |  |  |  |
  5 at BL/4 at Wk 52: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0
  5 at BL/4 at Wk 52 | 0 |  |  |  |  |
  5 at BL/5 at Wk 52: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0
  5 at BL/5 at Wk 52 | 100 |  |  |  |  |
  5 at BL/missing at Wk 52: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0
  5 at BL/missing at Wk 52 | 0 |  |  |  |  |

55. Secondary Outcome: Percentage of Participants Who Achieve Remission at Week 52 Among Participants With Isolated Ileal Crohn's Disease at Baseline
Description: Remission at Week 52 is defined as endoscopic remission at Week 52 AND clinical remission at Week 52. Endoscopic remission: SES-CD ≤ 4 and at least 2-point reduction versus Baseline and no subscore > 1 in any individual variable. Clinical remission: average daily stool frequency ≤ 1.5 and not worse than Baseline AND average daily abdominal pain ≤ 1.0 and not worse than Baseline. The very soft/liquid stool frequency and abdominal pain scores at a visit were the average of the daily values reported during the 7 usable days preceding the scheduled assessment visit. Abdominal Pain was rated on a 4-point scale from 0 (none) to 3 (severe). Details of the SES-CD scale are provided in the description of the first primary endpoint.
Time Frame: Baseline, Week 52
Population: Participants from ITT population with isolated ileal Crohn's disease at Induction Baseline. Non responder imputation.
Measure: Number; unit: percentage of participants
Arm/Group | Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction | Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction | Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction | Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction | Upadacitinib 3 mg BID in Extension/ Placebo in Induction | Upadacitinib 6 mg BID in Extension/ Placebo in Induction | Upadacitinib 12 mg BID in Extension/ Placebo in Induction | Upadacitinib 24 mg QD in Extension/ Placebo in Induction
Number analyzed (Participants) | 15 | 4 | 7 | 3 | 2 | 2 | 2 | 0
percentage of participants
  Responders: number analyzed (Participants) | 4 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Responders | 50.0 |  | 0 |  |  |  |  |
  Non-responders: number analyzed (Participants) | 11 | 4 | 6 | 3 | 2 | 2 | 2 | 0
  Non-responders | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
  Clinical responders: number analyzed (Participants) | 8 | 2 | 3 | 2 | 2 | 1 | 1 | 0
  Clinical responders | 25.0 | 0 | 0 | 0 | 0 | 0 | 0 |
  Clinical non-responders: number analyzed (Participants) | 7 | 2 | 4 | 1 | 0 | 1 | 1 | 0
  Clinical non-responders | 0 | 0 | 0 | 0 |  | 0 | 0 |
Statistical Analysis 1: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Responders; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -50.0, 95% CI 2-sided [-99.0 to -1.0] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 2: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical Responders; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -25.0, 95% CI 2-sided [-55.0 to 5.0] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 3: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical Responders; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -25.0, 95% CI 2-sided [-55.0 to 5.0] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 4: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical Responders; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -25.0, 95% CI 2-sided [-55.0 to 5.0] — [estimate comment as in outcome 25, analysis 1]

56. Secondary Outcome: Percentage of Participants Who Achieve Modified Clinical Remission at Week 52 Among Participants With Isolated Ileal Crohn's Disease at Baseline And Daily Stool Frequency ≥ 4.0 or Daily Abdominal Pain ≥ 2.0 at Induction Baseline
Description: as for outcome 29
Time Frame: Week 52
Population: Participants from ITT population with isolated ileal Crohn's disease at Induction Baseline and daily stool frequency >= 4.0 or daily abdominal pain >=2.0 at Induction Baseline. Non responder imputation.
Measure: Number; unit: percentage of participants
Arm/Group | Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction | Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction | Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction | Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction | Upadacitinib 3 mg BID in Extension/ Placebo in Induction | Upadacitinib 6 mg BID in Extension/ Placebo in Induction | Upadacitinib 12 mg BID in Extension/ Placebo in Induction | Upadacitinib 24 mg QD in Extension/ Placebo in Induction
Number analyzed (Participants) | 12 | 3 | 7 | 2 | 2 | 2 | 2 | 0
percentage of participants
  Responders: number analyzed (Participants) | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Responders | 66.7 |  | 0 |  |  |  |  |
  Non-responders: number analyzed (Participants) | 9 | 3 | 6 | 2 | 2 | 2 | 2 | 0
  Non-responders | 0 | 33.3 | 0 | 0 | 50.0 | 0 | 0 |
  Clinical responders: number analyzed (Participants) | 6 | 2 | 3 | 1 | 2 | 1 | 1 | 0
  Clinical responders | 33.3 | 50.0 | 0 | 0 | 50.0 | 0 | 0 |
  Clinical non-responders: number analyzed (Participants) | 6 | 1 | 4 | 1 | 0 | 1 | 1 | 0
  Clinical non-responders | 0 | 0 | 0 | 0 |  | 0 | 0 |
Statistical Analysis 1: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Responders; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -66.7, 95% CI 2-sided [-100.0 to -13.3] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 2: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Non-responders; Test type: Superiority; p = 0.250, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 33.3, 95% CI 2-sided [-20.0 to 86.7] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 3: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 6 mg BID in Extension/ Upadacitinib in Induction; Clinical responders; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = 16.7, 95% CI 2-sided [-62.2 to 95.6] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 4: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 12 mg BID in Extension/ Upadacitinib in Induction; Clinical responders; Test type: Superiority; p = 0.500, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -33.3, 95% CI 2-sided [-71.1 to 4.4] — [estimate comment as in outcome 25, analysis 1]
Statistical Analysis 5: Comparison: Upadacitinib 3 mg BID in Extension/Upadacitinib in Induction vs Upadacitinib 24 mg QD in Extension/ Upadacitinib in Induction; Clinical responders; Test type: Superiority; p = 1.000, Chi-squared — [p-value comment as in outcome 25, analysis 1]; Risk Difference (RD) = -33.3, 95% CI 2-sided [-71.1 to 4.4] — [estimate comment as in outcome 25, analysis 1]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events AEs (TEAEs): collected from the first dose of study drug through Week 52 plus 30 days.
Description: For the Extension Phase, a TEAE was defined as any AE with an onset date on or after the first dose of double-blind Extension dose and prior to the open-label dose or up to 30 days after the last dose of double-blind Extension dose if subject discontinued prematurely in the double-blind Extension Phase.
Groups:
- Double Blind Extension Phase: 3 mg BID: Upadacitinib 3 mg BID during the 36-week double-blind Extension Phase.
- Double Blind Extension Phase: 6 mg BID: Upadacitinib 6 mg BID during the 36-week double-blind Extension Phase.
- Double Blind Extension 12 mg BID: Upadacitinib 12 mg BID during the 36-week double-blind Extension Phase.
  (Participants in this arm who met inadequate response criteria at or after Week 20 and switched to OL 12 mg BID are included.)
- Double Blind Extension 24 mg QD: Upadacitinib 24 mg BID during the 36-week double-blind Extension Phase.
- Open Label Extension Subjects Never Received OL 24 mg BID: Participants from the Double Blind Extension 3 mg, 6 mg, and 24 mg arms who met inadequate response criteria at or after Week 20 and switched to OL 12 mg BID.
- Open Label Extension Subjects Received OL 24 mg BID: Participants from the Double Blind Extension 3 mg, 6 mg, 12 mg, and 24 mg arms who met inadequate response criteria at or after Week 20 and switched to OL 12 mg BID and then further dose escalated to OL 24 mg BID.
Arm/Group | Double-Blind Induction Phase: Placebo BID | Double-Blind Induction Phase: Upadacitinib 3 mg BID | Double-Blind Induction Phase: Upadacitinib 6 mg BID | Double Blind Induction Phase: 12 mg BID | Double Blind Induction Phase: 24 mg BID | Double Blind Induction Phase: 24 mg QD | Double Blind Extension Phase: 3 mg BID | Double Blind Extension Phase: 6 mg BID | Double Blind Extension 12 mg BID | Double Blind Extension 24 mg QD | Open Label Extension Subjects Never Received OL 24 mg BID | Open Label Extension Subjects Received OL 24 mg BID
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/39 | 0/37 | 0/36 | 0/36 | 0/35 | 0/60 | 0/23 | 0/59 | 0/36 | 0/33 | 0/27
Serious Adverse Events (participants affected / at risk) | 2/37 | 5/39 | 2/37 | 10/36 | 3/36 | 7/35 | 18/60 | 2/23 | 5/59 | 5/36 | 11/33 | 4/27
Other Adverse Events (participants affected / at risk) | 25/37 | 32/39 | 27/37 | 23/36 | 28/36 | 25/35 | 31/60 | 9/23 | 35/59 | 14/36 | 8/33 | 17/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double-Blind Induction Phase: Placebo BID (N=37) | Double-Blind Induction Phase: Upadacitinib 3 mg BID (N=39) | Double-Blind Induction Phase: Upadacitinib 6 mg BID (N=37) | Double Blind Induction Phase: 12 mg BID (N=36) | Double Blind Induction Phase: 24 mg BID (N=36) | Double Blind Induction Phase: 24 mg QD (N=35) | Double Blind Extension Phase: 3 mg BID (N=60) | Double Blind Extension Phase: 6 mg BID (N=23) | Double Blind Extension 12 mg BID (N=59) | Double Blind Extension 24 mg QD (N=36) | Open Label Extension Subjects Never Received OL 24 mg BID (N=33) | Open Label Extension Subjects Received OL 24 mg BID (N=27)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PULSELESS ELECTRICAL ACTIVITY (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SINUS BRADYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SINUS TACHYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
ANAL FISTULA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ANAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CROHN'S DISEASE (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (3) | 1 (1) | 2 (3) | 0 (0) | 7 (8) | 0 (0) | 2 (2) | 4 (4) | 7 (9) | 3 (3)
FISTULA OF SMALL INTESTINE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
GASTROINTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ILEAL PERFORATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ILEUS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INTESTINAL FISTULA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INTESTINAL STENOSIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
IRRITABLE BOWEL SYNDROME (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MESENTERIC VEIN THROMBOSIS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PERITONEAL ADHESIONS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (4) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
SMALL INTESTINAL PERFORATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CHEST PAIN (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ABSCESS INTESTINAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ANAL ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CELLULITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ESCHERICHIA BACTERAEMIA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INFLUENZA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PERITONITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RECTAL ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SEPSIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SUBCUTANEOUS ABSCESS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HODGKIN'S DISEASE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MALIGNANT NEOPLASM OF THYMUS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SYNCOPE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BIPOLAR DISORDER (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DEPRESSION (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SUICIDE ATTEMPT (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NEPHROLITHIASIS (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double-Blind Induction Phase: Placebo BID (N=37) | Double-Blind Induction Phase: Upadacitinib 3 mg BID (N=39) | Double-Blind Induction Phase: Upadacitinib 6 mg BID (N=37) | Double Blind Induction Phase: 12 mg BID (N=36) | Double Blind Induction Phase: 24 mg BID (N=36) | Double Blind Induction Phase: 24 mg QD (N=35) | Double Blind Extension Phase: 3 mg BID (N=60) | Double Blind Extension Phase: 6 mg BID (N=23) | Double Blind Extension 12 mg BID (N=59) | Double Blind Extension 24 mg QD (N=36) | Open Label Extension Subjects Never Received OL 24 mg BID (N=33) | Open Label Extension Subjects Received OL 24 mg BID (N=27)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 1 (1) | 3 (3) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
EYE PAIN (Eye disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 5 (6) | 2 (2) | 6 (8) | 2 (2) | 5 (5) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
ANORECTAL DISCOMFORT (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CROHN'S DISEASE (Gastrointestinal disorders) | 6 (6) | 6 (6) | 4 (4) | 7 (8) | 3 (3) | 2 (2) | 6 (6) | 2 (2) | 6 (7) | 2 (2) | 2 (3) | 3 (4)
DIARRHOEA (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
DYSPEPSIA (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FLATULENCE (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
HAEMATOCHEZIA (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 3 (3) | 2 (2) | 3 (4) | 3 (3) | 3 (4) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 2 (2) | 1 (1)
PROCTALGIA (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VOMITING (Gastrointestinal disorders) | 1 (1) | 4 (4) | 1 (1) | 3 (3) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 3 (3)
CHILLS (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FATIGUE (General disorders) | 3 (3) | 8 (9) | 2 (2) | 2 (2) | 4 (4) | 2 (2) | 2 (2) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
INFLUENZA LIKE ILLNESS (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OEDEMA PERIPHERAL (General disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PYREXIA (General disorders) | 3 (3) | 5 (6) | 0 (0) | 2 (2) | 1 (2) | 1 (2) | 1 (2) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
BRONCHITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
GASTROENTERITIS (Infections and infestations) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INFLUENZA (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ORAL HERPES (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
SINUSITIS (Infections and infestations) | 1 (2) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 (2) | 2 (3) | 2 (2) | 4 (4) | 4 (4) | 1 (2) | 3 (5) | 1 (1) | 4 (4) | 2 (2) | 0 (0) | 2 (2)
URINARY TRACT INFECTION (Infections and infestations) | 2 (2) | 1 (1) | 4 (4) | 0 (0) | 5 (5) | 2 (2) | 4 (5) | 1 (1) | 5 (6) | 0 (0) | 0 (0) | 0 (0)
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (2) | 4 (5) | 4 (5) | 4 (4) | 3 (5) | 2 (2) | 5 (5) | 1 (1) | 7 (8) | 2 (3) | 2 (2) | 3 (3)
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 4 (5) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
C-REACTIVE PROTEIN INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HAEMOGLOBIN DECREASED (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MALNUTRITION (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 3 (3) | 5 (5) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (4) | 2 (2) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LIPOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HEADACHE (Nervous system disorders) | 3 (3) | 7 (8) | 7 (11) | 3 (3) | 8 (9) | 5 (5) | 0 (0) | 1 (1) | 5 (6) | 1 (1) | 0 (0) | 0 (0)
ANXIETY (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INSOMNIA (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ACNE (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 3 (3) | 3 (3) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
ALOPECIA (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RASH (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 0 (0) | 1 (1) | 3 (3) | 2 (2) | 2 (2) | 3 (3)
RASH ERYTHEMATOUS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ROSACEA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
URTICARIA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HOT FLUSH (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERTENSION (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2016-11-07): https://cdn.clinicaltrials.gov/large-docs/49/NCT02365649/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-14): https://cdn.clinicaltrials.gov/large-docs/49/NCT02365649/SAP_001.pdf